| | Statistical Analysis Flatt Fillal | |
|---|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan | |
| Detailed Title: | A phase IIIA, randomised, observer-blind, multi-centre study to evaluate the clinical consistency of three production lots of the Porcine circovirus (PCV)-free liquid formulation of GlaxoSmithKline (GSK) Biologicals' oral live attenuated human rotavirus (HRV) vaccine and to evaluate the PCV-free liquid formulation of GSK Biologicals' HRV vaccine as compared to the currently licensed lyophilised formulation of the HRV vaccine in terms of immunogenicity, reactogenicity and safety when administered as a two-dose vaccination in healthy infants starting at age 6-12 weeks. | |
| eTrack study number and<br>Abbreviated Title | 115461 (F | ROTA-081) |
| Scope: | All data pertaining to the above study. Note that this analysis plan does not cover analyses devoted to iDMC. A separate SAP is available for the iDMC analyses. | |
| Date of Statistical Analysis<br>Plan | | May-2017 |
| Co-ordinating authors: | manager) | (study statistician); PPD (Stat |
| Reviewed by: | PPD<br>PPD | (Clinical and Epidemiology Project Lead) (Clinical Research and Development |
| | Lead) PPD PPD PPD PPD PPD PPD | (Lead statistician) (peer reviewer statistician), (Lead statistical analyst) (Lead Scientific writer) (Regulatory Affair) (Clinical Safety representative) (Public Disclosure) |
| Approved by: | PPD PPD Lead) PPD PPD PPD | (Clinical and Epidemiology Project Lead) (Clinical Research and Development (Lead statistician) (Lead statistical analyst) (Scientific writer) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | ABBREVIATIONS | 6 |
| 1. | DOC | UMENT HISTORY | 7 |
| 2. | STUD | DY DESIGN | 7 |
| 2 | 0D IE | -CTN/F0 | 44 |
| 3. | | | 11 |
| | 3.1.<br>3.2. | | 11<br>11 |
| 4. | ENDE | POINTS | 12 |
| →. | 4.1. | | 12 |
| | 4.2. | | 12 |
| 5. | ANAL | YSIS SETS | 13 |
| | 5.1. | Definitions | 13 |
| | | | 13 |
| | | 5.1.2. Per-Protocol analysis Set o | f immunogenicity (PPS)13 |
| | 5.2. | Criteria for eliminating data from ana | yses sets14 |
| | | | et (ES)14 |
| | | | col analysis Set (PPS)14 |
| | | | 15 |
| | | | a16 |
| | 5.3. | Important protocol deviation not lead protocol analysis set | ng to elimination from per- |
| ^ | $\circ$ | • | |
| 6. | | | 16 |
| | 6.1. | | |
| | | | paseline characteristics planned16 |
| | | | 17 |
| | 6.2. | | 17 |
| | 0.2. | | ed in the protocol17 |
| | | | 17 |
| | 6.3. | | 17 |
| | 0.5. | | planned in the protocol17 |
| | | | ssessment17 |
| | | 6 3 1 2 Retween groups a | assessment |
| | | 6.3.1.3. Statistical Metho | ods |
| | | | 18 |
| | 6.4. | | 19 |
| | 0.4. | | n the protocol19 |
| | | | 20 |
| 7. | ANAL | YSIS INTERPRETATION | 20 |
| 0 | CONT | DUCT OF ANALYSES | 04 |
| 8. | | | 21 |
| | O. I. | Sequence of analyses | |

| | | | | 115461 (ROTA-081) |
|---|---|---|---|---|
| | | | Statis | tical Analysis Plan Final |
| | | 8.1.1. | Final analysis up to Visit 3: | 21 |
| | 8.2. | | alysis | |
| | 8.3. | | al considerations for interim analyses | |
| 9. | CHAN | GES FRO | OM PLANNED ANALYSES | 22 |
| 10 | LICT | | DEDORT TARLES LISTINGS AND FIGURES | 22 |
| 10. | LIST | OF FINAL | REPORT TABLES, LISTINGS AND FIGURES | 22 |
| 11. | | | IDARD DATA DERIVATION RULE AND STAT | |
| | METH | | | |
| | 11.1. | Statistica | al Method References | <mark>23</mark> |
| | | 11.1.1. | Date derivation | <mark>23</mark> |
| | | 11.1.2. | Dose number | <mark>23</mark> |
| | | 11.1.3. | Demography | <mark>24</mark> |
| | | 11.1.4. | Immunogenicity | 24 |
| | | 11.1.5. | Safety | |
| | | 11.1.6. | Management of missing data | |
| | | 11.1.7. | Data presentation description | |
| 12. | ANNE | X 2: SUM | MARY ON ELIMINATION CODES | 28 |

115461 (ROTA-081) Statistical Analysis Plan Final

## **LIST OF TABLES**

| | | PAGE |
|---------|---------------------------------------------------|------|
| Table 1 | Study groups and epoch foreseen in the study | 8 |
| Table 2 | Study groups and treatments foreseen in the study | 8 |
| Table 3 | Blinding of study epoch | 9 |

115461 (ROTA-081) Statistical Analysis Plan Final

# **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Sequence for evaluating the study objectives in order to control the overall type I error below 2.5% | 21 |

115461 (ROTA-081) Statistical Analysis Plan Final

## **LIST OF ABBREVIATIONS**

AE Adverse event

ANOVA Analysis of Variance

cDISCI Clinical Data Interchange Standards Consortium

CI Confidence Interval
CRF Case Report Form

CTRS Clinical Trial Registry Summary

EL.U/ml ELISA unit per milliliter

Eli Type Internal GSK database code for type of elimination code

ELISA Enzyme-linked immunosorbent assay

ES Exposed Set
GE Gastroenteritis
GSK GlaxoSmithKline

iDMC Independent Data Monitoring Committee

IU/ml International units per milliliter

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not Applicable

PD Protocol Deviation

PPS Per Protocol Set

RV RotaVirus

SAE Serious adverse event SAP Statistical Analysis Plan

SAS Statistical Analysis Software

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

## 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|----------------------|
| 30 May 2017 | first version | Amendment 1 (09March |
| | | 2017) |

## 2. STUDY DESIGN



N: Number of subjects planned to be enrolled, n = number of subjects in each group

Review of the safety data for the first 800 enrolled subjects (50% of total enrolment) will be conducted as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available for 800 subjects.

Protocol waivers or exemptions are not allowed with the exception of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the outline of study procedures (Section 5.5 of protocol), are essential and required for study conduct.

• Experimental design: Phase IIIA, observer-blind, randomised (1:1:1:1), controlled, multi-centric, with four parallel groups and a staggered enrolment (Part A and Part B).

<sup>\*</sup> Contact (by telephone call or any other convenient procedure) for the safety follow-up will take place 6 months after the last dose of HRV vaccine.

<sup>\*\*</sup> Two oral doses of the study vaccines will be administered at an approximate 1-month or 2-months interval to subjects, according to the immunisation schedule for RV vaccine administration in participating countries. #Blood samples will be taken before the first dose and 1 to 2 months after the second dose.

<sup>\$</sup> An IDMC will review the safety data for the first 80 enrolled subjects (5% of total enrolment) and first 160 enrolled subjects (10% of total enrolment) as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available. Enrolment will be paused when first 10% of the subjects are enrolled for the purpose of the IDMC review of the safety data and will only resume if the outcome of the IDMC review is positive.

- Duration of the study: The intended duration of the study, per subject, will be approximately 7-8 months including the 6 months of extended safety follow-up period after the last dose of HRV vaccine.
  - Epoch 001: Primary starting at Visit 1 (Day 0) and ending at the safety follow-up contact (Month 7-8).
- Primary completion Date (PCD): Visit 3 (Month 2-4).

Refer to protocol glossary for the definition of PCD.

• End of Study (EoS): Last testing results released of samples collected at Visit 3 or Last Subject Last Visit (LSLV) (Follow up contact at month 7-8).

Refer to protocol glossary for the definition of EoS.

• Study groups: The study groups and epoch foreseen in the study are provided in Table 1.

Table 1 Study groups and epoch foreseen in the study

| Study Groups | Number of subjects | Age at Dose 1 (Min-Max) | Epoch<br>Epoch 001 |
|---|---|---|---|
| Liq_A | 400 | 6 weeks-12 weeks | • |
| Liq_B | 400 | 6 weeks-12 weeks | • |
| Liq_C | 400 | 6 weeks-12 weeks | • |
| Lyo | 400 | 6 weeks-12 weeks | • |

The study groups and treatments foreseen in the study are given in Table 2.

Table 2 Study groups and treatments foreseen in the study

| _ | Vaccina nama | | Study Groups | | |
|-----------------|----------------|-------|--------------|-------|-----|
| Treatment name | Vaccine name | Liq_A | Liq_B | Liq_C | Lyo |
| HRV Liquid | HRV PCV-free ‡ | Х | Х | Х | |
| HRV Lyophilised | HRV * | | | | Х |

<sup>‡</sup>PCV-free HRV liquid vaccine

- PCV-free HRV liquid formulation lot A (also referred to as Liq A group)
- PCV-free HRV liquid formulation lot B (also referred to as Liq\_B group)
- PCV-free HRV liquid formulation lot C (also referred to as Liq C group)
- GSK Biologicals' currently licensed lyophilised HRV formulation (also referred to as Lyo group)
- Control: active control-GSK Biologicals' currently licensed lyophilised HRV vaccine.

<sup>\*</sup> Licensed formulation of HRV lyophilised vaccine

- Vaccination schedule: Two doses of HRV vaccine to be administered according to a
  0, 1-2 month schedule according to the immunisation schedule for RV vaccine
  administration in participating countries.
  - Concomitant administration of routine childhood vaccines will be allowed according to local immunisation practices in each participating country.
- Treatment allocation: Randomised 1:1:1:1 using GSK Biologicals' central randomisation system on Internet (SBIR).
- Blinding: observer-blind

The blinding in the study is given in Table 3.

Table 3 Blinding of study epoch

| Study Epoch | Blinding* |
|-------------|----------------|
| Epoch 001 | Double-blind |
| Epoch 001 | Observer-blind |

<sup>\*</sup>Double blind for the three lots of PCV-free HRV liquid vaccine and observer-blind for the liquid formulation versus the lyophilised formulation.

- Sampling schedule: Blood samples will be collected from all subjects at Visit 1 and Visit 3 to measure serum anti-RV IgA antibody concentrations using Enzyme Linked Immunosorbent Assay (ELISA).
- Recording of GE episodes: Any GE episodes occurring from Dose 1 of HRV vaccine up to Visit 3 will be recorded for all subjects in the diary card. Parents/Legally Acceptable Representative(s) (LARs) will be instructed to collect stool sample(s) if the subject develops GE during the period from Dose 1 of HRV vaccine up to Visit 3. A stool sample should be collected as soon as possible after illness begins and preferably not later than 7 days after the start of GE symptoms. Two occurrences of diarrhoea will be classified as separate episodes if there will be five or more diarrhoea-free days between the episodes. Refer to the protocol glossary for definitions of GE and diarrhoea.
- Recording of Solicited AEs: Solicited AEs (fever, fussiness/irritability, loss of appetite, cough/runny nose, diarrhoea and vomiting) occurring between the day of each HRV vaccine dose and the following 7 days (Day 0-Day 7) will be recorded daily using diary cards for all subjects.
- Recording of Unsolicited AEs: Unsolicited AEs occurring within 31 days (Day 0-Day 30) after each dose of HRV vaccine will be recorded using diary cards for all subjects.
- Recording of SAEs: SAEs will be recorded from Visit 1 (Day 0) up to 6 months after Dose 2 of HRV vaccine.
- Type of study: self-contained
- Data collection: Electronic Case Report Form (eCRF)
- Safety monitoring: An IDMC comprising of clinical experts and a biostatistician, will review the safety data accrued during the study and the details of the review will be

115461 (ROTA-081) Statistical Analysis Plan Final

described in an IDMC charter. The IDMC review will happen after enrolment of 5%, 10% and 50% of subjects. The IDMC review will happen at the following stages:

Review of all safety data for the first 80 enrolled subjects (5% of total enrolment) as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available for 80 subjects.

- any available data beyond 8 days post Dose 2 will also be reviewed.
- during this IDMC review, enrolment of subjects will continue.

Review of all safety data for the first 160 enrolled subjects (10% of total enrolment) as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available for 160 subjects.

- any available data beyond 8 days post Dose 2 will also be reviewed.
- until this IDMC review, enrolment of subjects will pause. Enrolment will resume only if no safety concerns are raised by IDMC.

Review of all safety data for the first 800 enrolled subjects (50% of total enrolment) as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available for 800 subjects.

- any available data beyond 8 days post Dose 2 will also be reviewed.
- during this IDMC review, enrolment of subjects will continue.

## 3. OBJECTIVES

# 3.1. Co-Primary

• To demonstrate the lot-to-lot consistency of the PCV-free liquid HRV vaccine in terms of immunogenicity as measured by serum anti-RV IgA antibody concentrations 1-2 months after Dose 2.

Consistency will be demonstrated if, for all pairs of lots, the two-sided 95% confidence intervals (CIs) for the ratio of anti-RV IgA antibody GMCs 1-2 months after Dose 2 are within the [0.5; 2] clinical limit interval.

• To demonstrate the immunological non-inferiority of PCV-free liquid HRV vaccine as compared to the currently licensed lyophilised HRV vaccine in terms of seroconversion rates 1-2 months after Dose 2.

Non-inferiority will be demonstrated if the lower limit of the two-sided asymptotic standardized 95% CI for the difference in seroconversion rate between the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and licensed lyophilised HRV vaccine is greater than or equal to -10%.

• To demonstrate the non-inferiority of the PCV-free liquid HRV vaccine to that of the currently licensed lyophilised HRV vaccine in terms of serum anti-RV IgA antibody concentrations 1-2 months after Dose 2.

Non-inferiority will be demonstrated if the lower limit of the two-sided 95% CI for the ratio of anti-RV IgA antibody GMCs 1-2 months after Dose 2 between the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and the lyophilised HRV vaccine is greater than or equal to 0.67.

## 3.2. Secondary

#### Reactogenicity and safety

- To evaluate the reactogenicity of the liquid HRV vaccine and currently licensed lyophilised HRV vaccine in terms of solicited AEs during the 8 days (Day 0-Day 7) follow-up period after each vaccination.
- To assess the safety of the study vaccines in terms of unsolicited AEs during the 31 days (Day 0-Day 30) follow-up period after each vaccination and Serious Adverse Events (SAEs) during the entire study period.

#### **Immunogenicity**

• To assess the immunogenicity of the PCV-free liquid HRV vaccine and the currently licensed lyophilised HRV vaccine, in terms of percentage of subjects with anti-RV IgA antibody concentrations ≥ 90 U/mL 1-2 months after Dose 2.

## 4. ENDPOINTS

# 4.1. Primary

- Evaluation of immunogenicity in terms of anti-RV antibody concentrations
  - Serum anti-RV IgA antibody concentrations expressed as GMCs 1-2 months after Dose 2 in each of the HRV liquid formulation groups (Liq\_A, Liq\_B and Liq\_C).
  - Anti-RV IgA antibody seroconversion rate\* 1-2 months after Dose 2 in the lyophilised and pooled liquid groups.
  - Serum anti-RV IgA antibody concentrations expressed as GMCs 1-2 months after Dose 2 in the lyophilised and pooled liquid groups.

## 4.2. Secondary

- Solicited adverse events
  - Occurrence of each general solicited symptom within the 8 days (Day 0-Day 7) follow-up period after each dose of the lyophilised and PCV-free HRV liquid vaccine
- Unsolicited adverse events.
  - Occurrence of unsolicited AEs within 31 days (Day 0-Day 30) after any dose of HRV vaccine, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification.
- Serious adverse events
  - Occurrence of serious adverse events from Dose 1 up to study end.
- Evaluation of immunogenicity in terms of anti-RV antibody concentrations.
  - Serum anti-RV IgA antibody concentrations ≥ 90 U/mL 1-2 months after Dose 2 in the lyophilised and pooled liquid groups.

<sup>\*</sup>Seroconversion rate is defined as the percentage of subjects who were initially seronegative (i.e., with anti-RV IgA antibody concentration < 20 U/mL prior the first dose of HRV vaccine) and developed anti-RV IgA antibody concentration  $\ge 20$  U/mL at Visit 3.

## 5. ANALYSIS SETS

## 5.1. Definitions

## 5.1.1. Exposed Set

The ES will include all subjects with at least one study vaccine administration documented:

- a safety analysis based on the ES will include all vaccinated subjects,
- an immunogenicity analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available.

The ES analysis will be performed per treatment actually administered at dose 1.

## 5.1.2. Per-Protocol analysis Set of immunogenicity (PPS)

The PPS for immunogenicity will include all subjects from the ES:

- who have received all doses of study vaccine,
- for whom the HRV vaccine liquid or lyophilised formulation was administered according to protocol and subjects did not regurgitate after vaccination,
- who have not received a vaccine prohibited by the protocol up to Visit 3,
- for whom the randomisation code has not been broken
- who were seronegative for serum anti-RV IgA antibodies on the day of Dose 1
- who have not received medication prohibited by the protocol up to Visit 3 as listed in Section 6.7.2 of the study protocol,
- whose underlying medical condition was not prohibited by the protocol up to Visit 3 as listed in Section 6.8 of the study protocol,
- who comply with the vaccination schedule (Table 5 of the study protocol),
- who comply with blood sampling schedule (Table 5 of the study protocol),
- for whom immunogenicity data are available at the post-vaccination sampling time point,
- who have no RV other than vaccine strain in Gastroenteritis (GE) stool samples collected up to Visit 3,
- who have no concomitant infection unrelated to the vaccine up to Visit 3, which may influence the immune response.

## 5.2. Criteria for eliminating data from analyses sets

# 5.2.1. Elimination from Exposed set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES.

# 5.2.2. Elimination from Per-Protocol analysis Set (PPS)

A subject will be excluded from the PPS analysis under the following conditions

| Code | Decode => Condition under which the code is used |
|---|---|
| 900 | Questionable subject => subjects with invalid informed consent or fraudulent data Study vaccine dose not administrated but subject number allocated => subjects enrolled but not vaccinated |
| 1040 | Administration of vaccine(s) forbidden in the protocol => Administration of a vaccine not foreseen by the study protocol and administered during the period starting from 30 days before the first vaccination and ending at Visit 3, with the exception of the inactivated influenza vaccine, which is allowed at any time during the study, and other licensed routine childhood vaccinations. |
| 1060 | Randomisation code broken at the investigator site => Subjects unblinded in SBIR or unblinding reported as protocol deviation |
| 1070 | <ul> <li>Study vaccine dose not administered according to protocol =&gt;</li> <li>Subjects vaccinated with the correct vaccine but who regurgitated for one of the 2 doses;</li> <li>subjects for whom the second administered dose is not aligned with the first dose (e.g. lyo as second dose after a first dose with liquid from lot A; or liquid from lot B as second dose after a first dose with liquid from lot A)</li> <li>Subject who did not receive the second dose and return to visit 3 blood sample</li> <li>Subject who was given multiple doses at one visit</li> <li>Route of vaccination which is not oral</li> </ul> |
| 1080 | Vaccine temperature deviation => Subjects who have received a vaccine which had a temperature deviation qualified as inappropriate for use by Quality Assurance. |
| 1090 | Expired vaccine administered => Subjects who received an expired vaccine |

115461 (ROTA-081) Statistical Analysis Plan Final

| Code | Decode => Condition under which the code is used |
|---|---|
| N N | Protocol violation (inclusion/exclusion criteria) => Ineligible subjects who was vaccinated (i.e. Age at dose 1 is not between 42-90 days, gestational age is < 37 weeks 0 day or > 41 weeks 6 days or other eligibility criteria – see section 4.2 and 4.3 of the protocol) |
| | Initially seropositive or initially unknown antibody status => Anti-HRV concentration ≥ 20 U/mL or unknown at pre-dose 1 blood sample |
| | study vaccines used between Visit 1 and Visit 3 during the study period. Immunosuppressants or other immune-modifying drugs administered chronically (i.e., more than 14 days) during the study period between Visit 1 to Visit 3. For corticosteroids, this will mean prednisone (0.5 mg/kg/day, or equivalent). Inhaled and topical steroids are allowed. |
| r | Concomitant infection related to the vaccine which may influence immune response => Subjects with non-vaccine type RV detected in GE stool samples that may impact immunogenicity at Visit 3. |
| r | Concomitant infection not related to the vaccine which may influence immune response => Condition that has the capability of altering their immune response at visit 3 such autoimmune disease. |
| | Non-compliance with vaccination schedule (including wrong and unknown dates ) => Subjects who did not comply with the interval for dose 2 (Dose 2 should be between 28-83 days after Dose 1). |
| S | Non-compliance with blood sampling schedule (including wrong and unknown dates => Subjects who did not comply with the blood sample interval (blood sample post dose 2 should be between 28-83 days after Dose 2); subjects with a blood sample at visit 3 and without a second HRV vaccine administered |
| | Essential serological data missing => Anti-HRV results not available post-vaccination |
| | Obvious incoherence or abnormality or error in data => subjects without blood sample at visit 3 for whom a sample post-vaccination is found. |

# 5.2.3. Right censored Data

Not applicable

## 5.2.4. Visit-specific censored Data

Not applicable

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

- Forced randomization: In case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event.
- Manual randomization: In case the randomization system is unavailable, the investigator has the option to perform randomization by selecting supplies available at the site according to a pre-defined rule. In case the randomization system is available, a vaccine different from the randomized treatment may have been administered at dose 1.
- Short follow-up: subjects with a safety follow-up period after the last dose of HRV vaccine that is less than 180 days.
- Vaccinated subjects without documentation of solicited symptoms i.e. for a vaccine dose administered, at least one solicited symptom is not documented as being present or absent.

## 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in annex 1 and will not be repeated below. All Confidence Interval (CI) will be two-sided 95% CI.

# 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The following calculations will be performed for each group and for the pooled liquid vaccine group:

- The distribution of subjects enrolled among the study centres and countries will be tabulated as a whole and for each group.
- The numbers of subjects who withdraw from the study will be tabulated by group according to the reason for drop-out.
- The deviations from specifications for age and intervals between study visits will be tabulated by group.

- The median, mean, range and standard deviation of age (in weeks) at each HRV vaccine dose and of the gestational age will be computed by group. The median, mean and standard deviation of height (in centimetres) and weight (in kilograms) at Visit 1 will be computed by group. The racial and sex composition will be presented. These calculations will also be performed by country.
- Summary of co-administered vaccinations (i.e., vaccinations given on the day of each HRV vaccine dose) and intercurrent vaccinations (i.e., vaccinations from birth up to Visit 3, excluding vaccination given on the day of HRV vaccine doses) will be summarized by group for the ES.

#### 6.1.2. Additional considerations

All demography summaries will be generated for the ES. The summary of age, height, weight, race and sex will also be provided for the PPS. Number and reason for elimination from PPS will be tabulated by group. Summary of important protocol deviations not leading to elimination will be provided by groups for the PPS.

## 6.2. Exposure

## 6.2.1. Analysis of exposure planned in the protocol

Not applicable

#### 6.2.2. Additional considerations

The number of doses administered will be tabulated for each group.

## 6.3. Immunogenicity

#### 6.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the PPS for analysis of immunogenicity. If, in any vaccine group, the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is 5% or more, a second analysis based on the ES will be performed to complement the PPS analysis.

#### 6.3.1.1. Within groups assessment

The following calculations will be performed for each group and for the pooled liquid vaccine group.

- For each group, at each time point that anti-rotavirus IgA is measured,
  - Seropositivity/seroconversion rates and their exact 95% CI will be computed,
  - Percentage of subjects with anti-RV IgA antibody concentrations ≥ 90 U/mL and their exact 95% CI will be computed.

- GMCs and their 95% CIs will be computed.
- The above mentioned descriptive analyses will also be performed by country.
- The distribution of anti-RV IgA antibody concentrations at Visit 3 will be displayed using Reverse Cumulative Curves (RCCs).

#### 6.3.1.2. Between groups assessment

- The 95% CI for the ratio of anti-RV IgA antibody GMCs at Visit 3 between any pair of the three lots of the HRV liquid vaccine will be computed (first co-primary objective).
- The asymptotic standardized 95% CI for the difference in seroconversion rate at Visit 3 between the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and lyophilised HRV vaccine will be computed (second co-primary objective).
- The 95% CI for the ratio of anti-RV IgA antibody GMCs at Visit 3 between the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and lyophilised HRV vaccine will be computed (third co-primary objective).

#### 6.3.1.3. Statistical Methods

- The exact CIs for a proportion within a group will be calculated using SAS [see section 11.1].
- The standardized asymptotic CI for the group difference in proportion will be calculated using SAS [see section 11.1].
- The CI for GMCs will be obtained within each group separately. The CI for the mean of log-transformed concentration will be first obtained assuming that log-transformed values were normally distributed with unknown variance. The CI for the GMCs will then be obtained by exponential-transformation of the CI for the mean of log-transformed concentration.
- The GMC group ratio will be obtained using an ANOVA model on the logarithm-transformed concentrations. The ANOVA model will include the vaccine group and the country as fixed effects. The GMC ratio and their 95% CI will be derived by exponential-transformation of the corresponding group contrast in the model.

#### 6.3.2. Additional considerations

The ANOVA model for the lot-to-lot GMC ratio will include the data from the 3 HRV liquid groups only.

The country effect for the ANOVA model will be accounted by country indicator variables that will be treated as continuous variable in order to obtain adjusted GMCs that reflect the distribution of subjects between countries.

Summaries planned per countries will be limited to the PPS. These summaries will also be generated by frequent race and by gender. Note that a race category is considered if it

includes more than 40 subjects. Infrequent race categories will be combined together and summarized if it includes more than 40 subjects.

## 6.4. Analysis of safety

## 6.4.1. Analysis of safety planned in the protocol

The ES will be used for the analysis of safety.

The following calculations will be performed for each group and for the pooled liquid vaccine group:

The percentage of doses and of subjects reporting at least one symptom (solicited or unsolicited) during the 8 days (Day 0-Day 7) solicited follow-up period post vaccination will be computed, along with exact 95% CI. The same calculations will be done for symptoms (solicited or unsolicited) rated as grade 3 in intensity and for symptoms (solicited or unsolicited) assessed as causally related to vaccination.

The percentage of doses and of subjects reporting each individual solicited general symptom will be computed, over the 8 days (Day 0-Day 7) solicited follow-up period post vaccination, along with exact 95% CI. The same calculations will be done for each individual general solicited symptom rated as grade 3 in intensity, for each individual solicited general symptom assessed as causally related to vaccination and those that resulted in a medically attended visit.

The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to MedDRA. Every verbatim term will be matched with the appropriate Preferred Term. The percentage of subjects with unsolicited AEs occurring within 31 days (Day 0-Day 30) follow-up period after any dose with its exact 95% CI will be tabulated by group, and by preferred term. Similar tabulation will be done for unsolicited AEs rated as grade 3, for unsolicited AEs with causal relationship to vaccination and those that resulted in a medically attended visit.

The percentage of subjects reporting GE episodes from Dose 1 of HRV vaccine up to Visit 3 will be tabulated by group.

The percentage of subjects with presence of RV in GE stool samples collected from Dose 1 of HRV vaccine up to Visit 3 will be tabulated by group.

The percentage of GE episodes with no available stool results from Dose 1 of HRV vaccine up to Visit 3 will be tabulated.

The percentage of subjects who started taking at least one concomitant medication from HRV vaccination to Day 7 after vaccinations will be tabulated with exact 95% CI. The percentages of subjects who started taking at least one concomitant medication during the study period will be tabulated with exact 95% CI.

SAEs reported during the study period will be described in detail.

#### 6.4.2. Additional considerations

As indicated in section 10.5 of the protocol and in line with the project history, analysis of safety will be primarily performed per dose administered and subjects who missed reporting symptoms (solicited/unsolicited or concomitant medications) will be treated as subjects without symptoms (solicited/unsolicited or concomitant medications, respectively). A sensitivity analysis will be performed on documented doses i.e. accounting only for doses where solicited symptoms are indicated as being absent/present in case more than 5% of the doses are not documented.

Summary of temperature will be provided by  $0.5^{\circ}$  increment (i.e.  $\geq 38.0^{\circ}$ C, >38.5; >39, >39.5, >40).

Summary of solicited symptoms will also be provided by country, gender and frequent race(s) while summary of unsolicited symptoms within 31 days post-vaccination will be provided by country – see section 6.3.2 for the definition of frequent race.

Summary of solicited symptoms will also be provided for each individual general solicited symptom causally related to vaccination and rated as grade 3 in intensity. Likewise the percentage of subjects and of doses with grade 3 causally related unsolicited AEs occurring within 31 days (Day 0-Day 30) follow-up period after any dose with its exact 95% CI will be tabulated by group, and by preferred term. These summaries will not be provided by country, gender or frequent race(s).

Note that the study will be converted in cDISC. Accordingly Day 0-Day 7 and Day 0-Day 30 will be replaced by Day 1-Day 8 and Day 1-Day 31 for the statistical analysis.

### 7. ANALYSIS INTERPRETATION

Except for analyses addressing criteria specified in the co-primary objectives referred as confirmatory analyses, all the analyses will be descriptive/exploratory in nature. The use of these descriptive/exploratory analyses should be limited to support the confirmatory analyses or to generate hypothesis.

To control the overall type I error below 2.5%, the confirmatory objectives will be evaluated using a hierarchical procedure as shown in Figure 1. A confirmatory objective will be reached if the associated criteria are met and the previous objectives have been met.

Figure 1 Sequence for evaluating the study objectives in order to control the overall type I error below 2.5%



### 8. CONDUCT OF ANALYSES

## 8.1. Sequence of analyses

Safety data that is as clean as possible will be analysed for IDMC review. Details of the review are described in an IDMC charter.

### 8.1.1. Final analysis up to Visit 3:

An analysis will be conducted once all the study data up to Visit 3 are available and cleaned and Rota-IgA ELISA testing at 1-2 month post-dose 2 has been fully completed. The Clinical Study Report (CSR) with data up to Visit 3 will be used for the registration of PCV-free liquid vaccine in European Union (EU) and 'rest of world' countries.

The study report will include the following:

- All analysis of the serum anti-RV IgA antibody concentrations, 1-2 months after Dose 2 in the lyophilised and pooled liquid groups.
- All analyses of safety up to visit 3 and analysis of SAEs and AEs leading to drop out based on the database lock for the analysis.

# 8.2. Final analysis

If the previous analysis does not cover all study data, the study report will be amended when all data will be available. The study report amendment will include the additional safety information

The following table provides the plan for analyses excluding analyses dedicated to IDMC

| Description | Analysis<br>ID | Disclosure Purpose (IN=internal, CTRS=public posting, SR=study report and public posting) | Dry run<br>review<br>needed (Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final analysis up to Visit 3 | E1_05 | SR | Yes | Yes | TFL TOC first<br>version – All TFLs<br>as per database<br>lock date |
| Final | E1_01 | SR | No | Yes | TFL TOC first<br>version - All TFLs |

## 8.3. Statistical considerations for interim analyses

All confirmatory analyses will be conducted for the Final analysis up to Visit 3 and therefore no statistical adjustment for interim analyses is required.

### 9. CHANGES FROM PLANNED ANALYSES

Not applicable

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS,...). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The mock tables referred under column named 'layout' can be found in Annex 3 of this SAP

The following group names will be used in the TFLs, to be in line with the T-domains:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | Liq_A | PCV-free HRV liquid vaccine - lot A |
| 2 | Liq_B | PCV-free HRV liquid vaccine - lot B |
| 3 | Liq_C | PCV-free HRV liquid vaccine - lot C |
| 4 | Liq pooled | PCV-free HRV liquid vaccine - Pooled Lot |
| 5 | Lyo | HRV Lyophilised vaccine |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413. The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper: Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890. The standardised asymptotic method used is the method six.

#### 11.1.1. Date derivation

- SAS date derived from a character date: in case day is missing, PP is used. In case day & month are missing, PPD is used.
- Onset day for an event (ae, medication, vaccination, ...): the onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 1 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.

#### 11.1.2. Dose number

• The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.

- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered and an event occurs after the subsequent study dose (e.g. 2<sup>nd</sup> study dose), the relative dose of the event will be study dose associated to the subsequent study dose (e.g. dose 2).
- The number of doses for a product is the number of time the product was administered to a subject.
- The incidence per dose is the number of vaccination visits at which an event was reported among all vaccination visits.

## 11.1.3. Demography

Age: Age at the reference activity, computed as the number of complete weeks between the date of birth and the reference activity.

Conversion of weight to kg: the following conversion rule is used:

Weight in Kilogram= weight in Pounds / 2.2

Weight in Kilogram = weight in ounces / 35.2

The result is rounded to 2 decimals.

Conversion of height to cm: the following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48

Height in Centimetres = Height in Inch \* 2.54

The result is rounded to the unit (i.e. no decimal).

Conversion of temperature to °C: the following conversion rule is used:

Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

## 11.1.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced.
- The Geometric Mean Concentrations (GMCs) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in Section 5.7.3 of the protocol.

- A seronegative subject is a subject whose antibody concentration is below the cut-off value of the assay. A seropositive subject is a subject whose antibody concentration is greater than or equal to the cut-off value of the assay.
- The assay cut-off is the value under which there is no quantifiable result available. For an assay with a specific 'cut\_off', numerical immuno result is derived from a character field (rawres):
  - If rawres is 'NEG' or '-' or '(-)', numeric result= cut off/2,
  - if rawres is 'POS' or '+' or '(+)', numeric result = cut off,
  - if rawres is '< value' and value<=cut off, numeric result =cut off/2,
  - if rawres is '< value' and value>cut off, numeric result =value,
  - if rawres is '> value' and value<cut\_off, numeric result =cut\_off/2,</p>
  - if rawres is '> value' and value>=cut off, numeric result =value,
  - if rawres is '<= value' or '>= value' and value<cut\_off, numeric result =cut\_off/2,</p>
  - if rawres is '<= value' or '>= value' and value>=cut off, numeric result =value,
  - if rawres is a value < cut off, numeric result = cut off/2,
  - if rawres is a value >= cut off, numeric result = rawres,
  - if rawres is a value >= cut off, numeric result = rawres,
  - else numeric result is left blank.

### 11.1.5. Safety

- For analysis of solicited, unsolicited adverse events (such as serious adverse events or adverse events by primary MedDRA term) and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report the event or the concomitant medication will be considered as subjects without the event or the concomitant medication respectively.
- In case there will be more than 5% of subjects without documented dose for solicited symptoms (i.e., symptom screen not completed), sensitivity analysis will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed).
- The following rules will be used for the analysis of solicited symptoms:
  - Subject who didn't document the presence or absence of a solicited symptom
    after one dose will be considered not having that symptom after that dose in the
    analysis done on "administrated dose"
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
  - Subjects who documented the presence of a solicited symptom and fully or
    partially recorded daily measurement over the solicited period will be included in
    the summaries at that dose and classified according to their maximum observed
    daily recording over the solicited period.

115461 (ROTA-081) Statistical Analysis Plan Final

- Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be considered as having that symptom after that dose).
- For the analysis, temperatures will be coded as follows for oral, axillary or tympanic route:

| Grade | Temperature |
|-------|---------------------|
| 0 | < 38.0°C |
| 1 | ≥ 38.0°C - ≤ 38.5°C |
| 2 | > 38.5°C - ≤ 39.5°C |
| 3 | > 39.5°C |

• Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for<br>Vaccination phase | N used for deriving % per dose for<br>Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited general symptom | Primary analysis: all subjects with study vaccine administered | Primary analysis: all study visits with study vaccine administered |
| | Sensitivity analysis as applicable (see section 6.4.2): all subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) | Sensitivity analysis: all study visits with study vaccine administered and with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

115461 (ROTA-081) Statistical Analysis Plan Final

For summaries by MedDRA primary preferred term combining solicited and unsolicited adverse events, solicited adverse events will be coded as per the following MedDRA codes

| Solicited symptom | Lower level term code | Corresponding<br>Lower level term<br>decode |
|---|---|---|
| Fever | 10016558 | Fever |
| Irritability/Fussiness | 10022998 | Irritability |
| Diarrhoea | 10012727 | Diarrhoea |
| Vomiting | 10047700 | Vomiting |
| Loss of appetite | 10003028 | Appetite lost |
| Cough/runny nose | 10011224 | Cough |

## 11.1.6. Management of missing data

## **Demography:**

• For a given subject and a given demographic variable, missing measurements will not be replaced.

## **Immunogenicity:**

• For a given subject and a given immunogenicity measurement time point, missing or non-evaluable measurements will not be replaced.

## Reactogenicity and safety:

• Subjects who missed reporting symptoms (solicited/unsolicited or concomitant medications) will be treated as subjects without symptoms (solicited/unsolicited or concomitant medications, respectively).

# 11.1.7. Data presentation description

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| All summaries | % of count, including LL & UL of CI | 1 |
| Demographic characteristics | Mean, median, SD | 1 |
| Immunogenicity | % of difference, including LL & UL of CI | 2 |
| Immunogenicity | GMC group ratio, including LL & UL of CI | 2 |
| Immunogenicity | Anti-RV IgA GMC | 1 |

## 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to Section 5.2.

## 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following draft study specific mock TFLs will be used.

The data display, title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

These templates were copied from ROTA-061 and additional tables required for public disclosure were added. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

Note that all tables will include the pooled lot group for HRV liquid as shown in Template 2.

| Template 1 | Minimum and maximum activity dates (Exposed Set) | 32 |
|---|---|---|
| Template 2 | Number of subjects enrolled by center - Exposed Set | 32 |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal entire study period- Exposed Set | 33 |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Exposed Set) | 34 |
| Template 5 | Number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses with reasons for exclusion | 35 |
| Template 6 | Summary of demographic characteristics (Per Protocol Analysis Set of Immunogenicity) | 36 |
| Template 7 | Deviations from specifications for age and intervals between study visits - Exposed Set | 38 |
| Template 8 | Summary of co-administered vaccination by dose - Exposed Set | 39 |
| Template 9 | Summary of vaccinations other than HRV vaccine administered from birth until Visit 3, excluding vaccination given on the day of HRV doses - Exposed Set | 40 |
| Template 10 | Anti-rotavirus IgA antibody GMC and seroconversion rates – Per Protocol Analysis Set of Immunogenicity | 41 |
| Template 11 | Anti-rotavirus IgA antibody GMC calculated on subjects seropositive for anti-rotavirus IgA antibodies – Per Protocol Analysis Set of Immunogenicity | 41 |
| Template 12 | Ratio of anti-rotavirus IgA antibody GMCs 1-2 months after Dose 2 of the HRV vaccine between each pair of the three lots of | |

CONFIDENTIAL 115461 (ROTA-081) Statistical Analysis Plan Final the HRV PCV-free liquid vaccine - Per Protocol Analysis Set of Immunogenicity......42 Template 13 Difference between groups in the percentage of subjects who seroconverted for anti-rotavirus IgA antibody 1-2 months after Dose 2 of the HRV vaccine – Per Protocol Analysis Set of Ratio of anti-rotavirus IgA antibody GMCs 1-2 months after Dose Template 14 2 of the HRV vaccine between the HRV lyophilised vaccine group and the pooled HRV PCV-free liquid vaccine - Per Protocol Analysis Set of Immunogenicity......42 Template 15 Reverse cumulative distribution curve for anti-rotavirus IgA antibody concentrations at Visit 3 - Per Protocol Analysis Set of Immunogenicity......43 Template 16 Number and percentage of subjects who received study vaccine doses - Exposed Set ......43 Template 17 Compliance in returning symptom sheets - Exposed Set......44 Template 18 Percentage of doses and of subjects reporting symptoms (solicited or unsolicited) reported during the 8-day (Day 0 to Day 7) follow-up period - Exposed Set ......45 Template 19 Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, after each dose of the HRV lyophilised and HRV PCVfree liquid vaccine for all groups. - Exposed Set......46 Percentage of subjects reporting each solicited general symptom Template 20 including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each dose in the pooled HRV PCV-free liquid vaccine group and the HRV vaccine lyophilised formulation group -Exposed Set......48 Template 21 Percentage of doses and subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, after each dose of the HRV lyophilised and HRV PCV-free HRV liquid vaccine for all groups.

Template 22

Percentage of subjects with unsolicited symptoms classified by

MedDRA SOC and PT from Day 0 to Day 30 after any vaccination in each HRV PCV-free vaccine liquid group -

- Exposed Set ......49

115461 (ROTA-081) Statistical Analysis Plan Final

| Template 23 | Percentage of doses with unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after vaccination in each HRV PCV-free liquid vaccine group - Exposed Set | 53 |
|---|---|---|
| Template 24 | Percentage of subjects reporting any GE episodes from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set | 54 |
| Template 25 | Percentage of subjects reporting RV (vaccine strain or wild type RV) GE episodes from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set | 55 |
| Template 26 | Summary of RV GE episodes reported from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set | 56 |
| Template 27 | Number and percentage of doses and of subjects who took at least one concomitant medication from Day 0 to Day 7 after vaccination by type in each HRV PCV-free vaccine liquid group - Exposed Set | 56 |
| Template 28 | Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each documented dose in each HRV PCV-free liquid group - Exposed Set | 57 |
| Template 29 | Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort) | 58 |
| Template 30 | Subjects with Serious Adverse Events reported up to Visit 3 - Exposed Set | 58 |
| Template 31 | Number (%) of subjects with serious adverse events from Dose 1 up to study end, including number of events reported (Exposed Set) | 58 |
| Template 32 | Solicited and unsolicited symptoms experienced by at least 5 % of subjects classified by MedDRA Primary System Organ Class and Preferred Term within 31-day (Days 0-30) post-vaccination period after any dose of HRV PCV-free liquid vaccine - SAE excluded (Exposed Set) | 59 |
| Template 33 | Number of subjects by country | 59 |
| Template 34 | Number of enrolled subjects by age category (Exposed Set) | 60 |
| Template 35 | Study population (Exposed Set) | 60 |

Template 1 Minimum and maximum activity dates (Exposed Set)

| Visit | Minimum date | Maximum date |
|-------|--------------|--------------|
| 1 | 19JUN2007 | 29DEC2007 |
| 2 | 24JUL2007 | 08FEB2008 |
| 3 | 24AUG2007 | 18MAR2008 |
| 4 | 25MAR2008 | 22NOV2008 |
| 5 | 24MAR2009 | 31MAR2009* |

<sup>\*</sup>Database Lock Date = 31MAR2009

Template 2 Number of subjects enrolled by center - Exposed Set

| | | LIQ_A | LIQ_B | LIQ_C | LIQ_pool | LYO | Total | |
|---------|--------|-------|-------|-------|----------|-----|-------|------|
| Country | Center | n | n | n | n | n | n | % |
| XXXX | PPD | 38 | 38 | 38 | | 37 | 151 | 12.6 |
| | PPD | 20 | 20 | 20 | | 20 | 80 | 6.7 |
| | PPD | 30 | 30 | 29 | | 29 | 118 | 9.8 |
| | PPD | 19 | 19 | 20 | | 20 | 78 | 6.5 |
| | All | | | | | | | |
| YYYYY | PPD | 15 | 15 | 15 | | 15 | 60 | 5.0 |
| | PPD | 22 | 22 | 23 | | 22 | 89 | 7.4 |
| | PPD | 35 | 36 | 36 | | 35 | 142 | 11.8 |
| | PPD | 28 | 28 | 28 | | 28 | 112 | 9.3 |
| | PPD | 20 | 21 | 20 | | 21 | 82 | 6.8 |
| | PPD | 22 | 23 | 22 | | 23 | 90 | 7.5 |
| | PPD | 22 | 23 | 22 | | 23 | 90 | 7.5 |
| | PPD | 27 | 27 | 27 | | 27 | 108 | 9.0 |
| | All | | | | | | | |
| All | All | 298 | 302 | 300 | | 300 | 1200 | 100 |

<sup>&</sup>lt;group description >

n = n number of subjects included in each group or in total for a given center or for all centers All = sum of all subjects in each group or in total (sum of all groups)

 $<sup>% =</sup> n/AII \times 100$ 

# Template 3 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal entire study period- Exposed Set

| | LIQ_A | LIQ_B | LIQ_C | LYO | Total |
|---|---|---|---|---|---|
| Number of subjects vaccinated | 298 | 302 | 300 | 300 | 1200 |
| Number of subjects completed | 297 | 301 | 298 | 297 | 1193 |
| Number of subjects withdrawn | 1 | 1 | 2 | 3 | 7 |
| Reasons for withdrawal : | | | | | |
| Serious Adverse Event | 0 | 0 | 0 | 1 | 1 |
| Non-serious adverse event | 0 | 0 | 0 | 0 | 0 |
| Protocol violation | 0 | 0 | 0 | 0 | 0 |
| Consent withdrawal (not due to an adverse event) | 1 | 0 | 1 | 2 | 4 |
| Migrated/moved from study area | 0 | 1 | 1 | 0 | 2 |
| Lost to follow-up (subjects with incomplete vaccination course) | 0 | 0 | 0 | 0 | 0 |
| Lost to follow-up (subjects with complete vaccination course) | 0 | 0 | 0 | 0 | 0 |
| Others | 0 | 0 | 0 | 0 | 0 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LYO = HRV vaccine lyophilised formulation

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed study visit 3

Withdrawn = number of subjects who did not come for study visit 3

115461 (ROTA-081) Statistical Analysis Plan Final

# Template 4 Number of subjects at each visit and list of withdrawn subjects (Exposed Set)

| Group | VISIT | N | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| Liq_A | VISIT 1 508 | | | |
| | - | | no. PP | CONSENT WITHDRAWAL |
| | | | no PP | CONSENT WITHDRAWAL |
| | | | no PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 504 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | SERIOUS ADVERSE EXPERIENCE |
| | VISIT 3 | 501 | | |
| | | | no. | MIGRATION FROM STUDY AREA |
| | | | no. P | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no.PPD | MIGRATION FROM STUDY AREA |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no PPD | MIGRATION FROM STUDY AREA |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | VISIT 4 | 492 | | |
| Lyo | VISIT 1 | 257 | | |
| | | | no. PP | PROTOCOL VIOLATION |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 255 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 3 | 254 | | |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | LOST TO FOLLOW-UP |
| | | | no. PP | LOST TO FOLLOW-UP |
| - | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | LOST TO FOLLOW-UP |
| | | | no. PPD | ADVERSE EXPERIENCE |
| | VISIT 4 | 247 | | |

Template 5 Number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses with reasons for exclusion

| | | То | tal | | LIQ_A | | | I | LIQ_B | | | LIQ_C | | | LYO | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Title | N | n | S | % | N | n | S | N | n | s | N | n | s | N | n | s |
| Total enrolled cohort | 1200 | | | | 298 | | | 302 | | | 300 | | | 300 | | |
| Exposed Set | 1200 | | | 100 | 298 | | | 302 | | | 300 | | | 300 | | |
| Administration of vaccine(s) forbidden in the protocol (code 1040) | | 2 | 2 | | | 1 | 1 | | 1 | 1 | | 0 | 0 | | 0 | 0 |
| Study vaccine dose not administered according to protocol (code 1070) | | 73 | 73 | | | 21 | 21 | | 13 | 13 | | 23 | 23 | | 16 | 16 |
| Initially seropositive or unknown anti-rotavirus IgA antibody on day of dose 1 (code 1500) | | 10 | 11 | | | 3 | 4 | | 3 | 3 | | 3 | 3 | | 1 | 1 |
| Protocol violation<br>(inclusion/exclusion criteria)<br>(code 2010) | | 1 | 1 | | | 0 | 0 | | 0 | 0 | | 1 | 1 | | 0 | 0 |
| Administration of any medication forbidden by the protocol (code 2040) | | 1 | 1 | | | 0 | 0 | | 0 | 0 | | 0 | 0 | | 1 | 1 |
| Underlying medical condition forbidden by the protocol (code 2050) | | 1 | 1 | | | 1 | 1 | | 0 | 0 | | 0 | 0 | | 0 | 0 |
| Concomitant infection not related to the vaccine which may influence immune response (code 2070) | | 0 | 1 | | | 0 | 0 | | 0 | 0 | | 0 | 0 | | 0 | 1 |
| Non-compliance with vaccination schedule (including wrong and unknown dates ) (code 2080) | | 14 | 16 | | | 5 | 5 | | 0 | 0 | | 6 | 7 | | 3 | 4 |
| Non-compliance with blood<br>sampling schedule (including<br>wrong and unknown dates)<br>(code 2090) | | 12 | 16 | | | 2 | 3 | | 3 | 3 | | 3 | 5 | | 4 | 5 |
| Essential serological data missing (code 2100) | | 87 | 95 | | | 23 | 25 | | 21 | 22 | | 20 | 22 | | 23 | 26 |
| Subjects with incomplete study vaccination schedule but with post serological result (code 2500) Per protocol set | 998 | 1 | 1 | 83.2 | 242 | 0 | 0 | 260 | 1 | 1 | 244 | 0 | 0 | 252 | 0 | 0 |

LIQ\_A = HRV vaccine liquid formulation Lot A LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C LYO = HRV vaccine lyophilised formulation

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

<sup>% =</sup> percentage of subjects in the per protocol set (PPS) relative to the exposed set (ES)

115461 (ROTA-081) Statistical Analysis Plan Final

Template 6 Summary of demographic characteristics (Per Protocol Analysis Set of Immunogenicity)

| | | LIQ_A<br>N = 242 | | LIQ_B<br>N = 260 | | LIQ_C<br>N = 244 | | LYO<br>N = 252 | | Total<br>N = 998 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Value | % | Value | | Value | | Value | | Value | |
| Characteristics | Parameters or Categories | or n | /6 | or n | /0 | or n | 70 | or n | /0 | or n | /6 |
| Age at Dose 1 | Mean | 11.6 | - | 11.5 | - | 11.5 | - | 11.6 | - | 11.6 | - |
| of HRV vaccine<br>(weeks) | SD | 1.32 | - | 1.16 | - | 1.19 | - | 1.20 | - | 1.22 | - |
| | Median | 11.0 | - | 11.0 | - | 11.0 | - | 11.0 | - | 11.0 | - |
| | Minimum | 10 | - | 10 | - | 10 | - | 10 | - | 10 | - |
| | Maximum | 17 | - | 15 | - | 15 | - | 16 | - | 17 | - |
| Age at Dose 2 | Mean | 16.6 | - | 16.5 | - | 16.5 | - | 16.7 | - | 16.6 | - |
| of HRV vaccine | SD | 1.48 | - | 1.40 | - | 1.37 | - | 1.34 | - | 1.40 | - |
| (weeks) | Median | 17.0 | - | 16.0 | - | 16.0 | - | 17.0 | - | 17.0 | - |
| | Minimum | 14 | - | 14 | - | 14 | - | 14 | - | 14 | - |
| | Maximum | 22 | - | 20 | - | 20 | - | 21 | - | 22 | - |
| Gender | Female | 122 | 50.4 | 121 | 46.5 | 120 | 49.2 | 120 | 47.6 | 483 | 48.4 |
| | Male | 120 | 49.6 | 139 | 53.5 | 124 | 50.8 | 132 | 52.4 | 515 | 51.6 |
| Ethnicity | American Hispanic or Latino | 0 | 0.0 | 2 | 0.8 | 1 | 0.4 | 0 | 0.0 | 3 | 0.3 |
| | Not American Hispanic or Latino | 242 | 100.<br>0 | 258 | 99.2 | 243 | 99.6 | 252 | 100.<br>0 | 995 | 99.7 |
| Race | African heritage / African<br>American | 1 | 0.4 | 0 | 0.0 | 1 | 0.4 | 0 | 0.0 | 2 | 0.2 |
| | American Indian or Alaskan native | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - central/south Asian<br>heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - east Asian heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - Japanese heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - south east Asian<br>heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Native Hawaiian or other pacific islander | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | White - Arabic / north African<br>heritage | 0 | 0.0 | 0 | 0.0 | 2 | 8.0 | 0 | 0.0 | 2 | 0.2 |
| | White - Caucasian / European heritage | 239 | 98.8 | 258 | 99.2 | 240 | 98.4 | 247 | 98.0 | 984 | 98.6 |
| | Other | 2 | 8.0 | 2 | 0.8 | 1 | 0.4 | 5 | 2.0 | 10 | 1.0 |
| Height at Visit<br>1 (cm) | Mean | 60.4 | - | 60.5 | - | 60.7 | <u> -</u> | 60.6 | - | 60.5 | - |
| | SD | 2.35 | - | 2.37 | - | 2.32 | - | 2.22 | - | 2.32 | - |
| | Median | 61.0 | - | 60.0 | - | 61.0 | <u> -</u> | 61.0 | - | 61.0 | - |
| | Unknown | 0 | - | 1 | - | 2 | - | 0 | - | 3 | - |
| Weight at Visit<br>1 (kg) | Mean | 6.0 | - | 6.1 | - | 6.2 | - | 6.1 | - | 6.1 | - |
| | SD | 0.77 | - | 0.76 | - | 0.77 | <u> -</u> | 0.75 | - | 0.76 | - |
| | Median | 6.0 | - | 6.0 | - | 6.2 | - | 6.1 | - | 6.1 | - |
| BMI at Visit 1<br>(kg/m²) | Mean | 16.5 | - | 16.6 | - | 16.7 | - | 16.7 | - | 16.6 | - |
| | SD | 1.49 | - | 1.46 | - | 1.46 | - | 1.46 | - | 1.47 | - |
| | Median | 16.3 | - | 16.5 | - | 16.5 | - | 16.7 | - | 16.5 | - |
| | Unknown | 0 | - | 1 | - | 2 | - | 0 | - | 3 | - |
115461 (ROTA-081) Statistical Analysis Plan Final

LIQ\_A = HRV vaccine liquid formulation Lot A LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C LYO = HRV vaccine lyophilised formulation

N = total number of subjects

n (%) = number / percentage of subjects in a given category Value = value of the considered parameter

SD = standard deviation

# Template 7 Deviations from specifications for age and intervals between study visits - Exposed Set

| | | Age | PRE-Dose:1 | Dose:1 | -Dose:2 | Dose:2 | -PII(M2) |
|---|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Adapted | Protocol | Adapted |
| • | | from 10 to 17 | from 0 to 0 days | from 30 to 48 | from 21 to 48 | from 30 to 48 | from 21 to 48 |
| | | weeks | | days | days | days | days |
| LIQ_A | N | 298 | 298 | 297 | 297 | 287 | 287 |
| | n | 0 | 2 | 8 | 7 | 1 | 1 |
| | % | 0.0 | 0.7 | 2.7 | 2.4 | 0.3 | 0.3 |
| | range | 10 to 17 | 0 to 4 | 29 to 76 | 29 to 76 | 30 to 55 | 30 to 55 |
| LIQ_B | N | 302 | 302 | 301 | 301 | 294 | 294 |
| | n | 0 | 1 | 0 | 0 | 4 | 2 |
| | % | 0.0 | 0.3 | 0.0 | 0.0 | 1.4 | 0.7 |
| | range | 10 to 15 | 0 to 3 | 30 to 48 | 30 to 48 | 24 to 56 | 24 to 56 |
| LIQ_C | N | 300 | 300 | 300 | 300 | 291 | 291 |
| | n | 1 | 1 | 8 | 7 | 4 | 4 |
| | % | 0.3 | 0.3 | 2.7 | 2.3 | 1.4 | 1.4 |
| | range | 9 to 17 | 0 to 9 | 27 to 76 | 27 to 76 | 30 to 56 | 30 to 56 |
| LYO | N | 300 | 300 | 299 | 299 | 289 | 289 |
| | n | 0 | 2 | 4 | 4 | 5 | 3 |
| | % | 0.0 | 0.7 | 1.3 | 1.3 | 1.7 | 1.0 |
| | range | 10 to 16 | 0 to 3 | 30 to 61 | 30 to 61 | 28 to 61 | 28 to 61 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LYO = HRV vaccine lyophilised formulation

PRE = pre-vaccination

PII (M2) = blood sample taken one month after Dose 2 of the HRV vaccine (Visit 3)

Adapted = interval used for defining the ATP cohorts for immunogenicity

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

#### Summary of co-administered vaccination by dose - Exposed Set Template 8

| Dose1 | LIQ_A<br>N = 298 | _ | | _ | | LIQ_C<br>N = 300 | | LYO<br>N = 300 | | 00 |
|---|---|---|---|---|---|---|---|---|---|---|
| | Value | % | Value | % | Value | % | Value | % | Value | % |
| Characteristics | or n | | or n | | or n | | or n | | or n | |
| Any | 298 | 100 | 302 | 100 | 299 | 99.7 | 300 | 100 | 1199 | 99.9 |
| Infanrix hexa | 298 | 100 | 302 | 100 | 299 | 99.7 | 300 | 100 | 1199 | 99.9 |
| Dose 2 | LIQ_A<br>N = 297 | , | LIQ_B<br>N = 301 | | LIQ_C<br>N = 300 | ) | LYO<br>N = 299 | | Total<br>N = 1197 | |
| | Value | % | Value | % | Value | % | Value | % | Value | % |
| Characteristics | or n | | or n | | or n | | or n | | or n | |
| Any | 297 | 100 | 301 | 100 | 298 | 99.3 | 299 | 100 | 1195 | 99.8 |
| Infanrix hexa | 297 | 100 | 301 | 100 | 298 | 99.3 | 299 | 100 | 1195 | 99.8 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LYO = HRV vaccine lyophilised formulation

N = total number of subjects having received the considered dose of HRV n/% = number/percentage of subjects who received the specified vaccination on the same day as the considered dose of HRV vaccine

Template 9 Summary of vaccinations other than HRV vaccine administered from birth until Visit 3, excluding vaccination given on the day of HRV doses - Exposed Set

| Before Dose 1 | | LIQ_ | Α | | LIQ_I | В | | LIQ_ | C | | LYC | ) | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N = 2 | 98 | | N = 30 | )2 | | N = 3 | 00 | | N = 3 | 00 | ı | N = 120 | 00 |
| | # | n | % | # | n | % | # | n | % | # | n | % | # | n | % |
| Characteristics | | | | | | | | | | | | | | | |
| Any | 18 | 18 | 6.0 | 11 | 11 | 3.6 | 13 | 13 | 4.3 | 25 | 25 | 8.3 | 67 | 67 | 5.6 |
| BCG | 18 | 18 | 6.0 | 11 | 11 | 3.6 | 12 | 12 | 4.0 | 25 | 25 | 8.3 | 66 | 66 | 5.5 |
| Infanrix hexa™ | 0 | 0 | 0.0 | 0 | 0 | 0.0 | 1 | 1 | 0.3 | 0 | 0 | 0.0 | 1 | 1 | 0.1 |
| Between Dose 1 and | | LIQ | Α | | LIQ_I | В | | LIQ C | | | LYC | ) | | Total | • |
| Dose 2§ | | N = 298 | | | N = 302 | | | N = 3 | 00 | | N = 3 | 00 | ı | N = 120 | 00 |
| | # | n | % | # | n | % | # | n | % | # | n | % | # | n | % |
| Characteristics | | | | | | | | | | | | | | | |
| Any | 0 | 0 | 0.0 | 2 | 1 | 0.3 | 0 | 0 | 0.0 | 0 | 0 | 0.0 | 2 | 1 | 0.1 |
| Infanrix hexa™ | 0 | 0 | 0.0 | 2 | 1 | 0.3 | 0 | 0 | 0.0 | 0 | 0 | 0.0 | 2 | 1 | 0.1 |
| Between Dose 2 and | | LIQ_ | Α | | LIQ_I | В | | LIQ_ | С | | LYC | ) | | Total | • |
| Visit 3* | | N = 2 | 97 | | N = 30 | )1 | | N = 3 | 00 | | N = 2 | 99 | ı | N = 119 | 97 |
| | # | n | % | # | n | % | # | n | % | # | n | % | # | n | % |
| Characteristics | | | | | | | | | | | | | | | |
| Any | 291 | 291 | 98.0 | 295 | 295 | 98.0 | 287 | 286 | 95.3 | 290 | 290 | 97.0 | 1163 | 1162 | 97.1 |
| DTPa+IPV+Hib | 0 | 0 | 0.0 | 1 | 1 | 0.3 | 0 | 0 | 0.0 | 0 | 0 | 0.0 | 1 | 1 | 0.1 |
| Infanrix hexa™ | 291 | 291 | 98.0 | 294 | 294 | 97.7 | 287 | 286 | 95.3 | 290 | 290 | 97.0 | 1162 | 1161 | 97.0 |

LIQ\_A = HRV vaccine liquid formulation Lot A

§= up to last contact of conclusion at Visit 3 if dose 2 of HRV was not administered

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LYO = HRV vaccine lyophilised formulation

N = Before Dose 1 and between Dose 1 and Dose 2: total number of subjects having received dose 1 of HRV Between Dose 2 and visit 3: total number of subjects having received dose 2 of HRV

<sup>#=</sup> number of doses administered of the specified vaccination excluding vaccination given on the day of HRV doses n/% = number/percentage of subjects who received at least one specified vaccination between the considered visits excluding vaccination given on the day of HRV doses

<sup>\*=</sup> up to last contact of conclusion at Visit 3 if visit 3 was not done

# Template 10 Anti-rotavirus IgA antibody GMC and seroconversion rates – Per Protocol Analysis Set of Immunogenicity

| | | | | ≥ 20 | J/ml | | | GMC (U/ml) | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% | 6 CI | | 95% | 6 CI |
| Group | Timing | N | n | % | LL | UL | value | LL | UL |
| LIQ_A | PRE | 242 | 0 | 0.0 | 0.0 | 1.5 | <20 | - | - |
| | PII(M2) | 242 | 220 | 90.9 | 86.6 | 94.2 | 384.4 | 309.1 | 478.2 |
| LIQ_B | PRE | 260 | 0 | 0.0 | 0.0 | 1.4 | <20 | - | - |
| | PII(M2) | 260 | 235 | 90.4 | 86.1 | 93.7 | 418.8 | 337.8 | 519.1 |
| LIQ_C | PRE | 244 | 0 | 0.0 | 0.0 | 1.5 | <20 | - | - |
| | PII(M2) | 244 | 206 | 84.4 | 79.3 | 88.7 | 324.4 | 253.4 | 415.3 |
| LIQPOOL | PRE | 746 | 0 | 0.0 | 0.0 | 0.5 | <20 | - | - |
| | PII(M2) | 746 | 661 | 88.6 | 86.1 | 90.8 | 374.7 | 328.8 | 426.9 |
| LYO | PRE | 252 | 0 | 0.0 | 0.0 | 1.5 | <20 | - | - |
| | PII(M2) | 252 | 228 | 90.5 | 86.2 | 93.8 | 331.8 | 265.0 | 415.4 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects with available results

n (%) = number/percentage of subjects with concentration above the cut-off

95% CI = 95% Confidence Interval; L.L =Lower limit; U.L = upper limit

Pre = pre-vaccination

PII (M2) = blood sample taken one month after Dose 2 of HRV vaccine (Visit 3)

Template 11 Anti-rotavirus IgA antibody GMC calculated on subjects seropositive for anti-rotavirus IgA antibodies – Per Protocol Analysis Set of Immunogenicity

| | | | | GMC | |
|---------|---------|-----|-------|-------------|-------|
| | | | | 95% CI | |
| Group | Timing | N | value | LL | UL |
| LIQ_A | PII(M2) | 220 | 553.8 | 463.4 | 661.7 |
| LIQ_B | PII(M2) | 235 | 623.0 | 525.0 | 739.4 |
| LIQ_C | PII(M2) | 206 | 616.4 | 510.4 | 744.4 |
| LIQPOOL | PII(M2) | 661 | 597.1 | 538.7 | 661.8 |
| LYO | PII(M2) | 228 | 479.7 | 395.4 582.0 | |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects who were seropositive for anti-rotavirus IgA antibodies

95% CI = 95% Confidence Interval; LL = Lower Limit; UL = Upper Limit

PII(M2) = blood sample taken one month after Dose 2 of HRV vaccine (Visit 3)

Template 12 Ratio of anti-rotavirus IgA antibody GMCs 1-2 months after Dose 2 of the HRV vaccine between each pair of the three lots of the HRV PCV-free liquid vaccine – Per Protocol Analysis Set of Immunogenicity

| | | | | | | GMC ratio | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 95% | |
| Group | N | GMC | Group | N | GMC | Ratio order | Value | LL | UL |
| LIQ_A | 242 | 384.4 | LIQ_B | 260 | 418.8 | LIQ_A /LIQ_B | 0.92 | 0.67* | 1.26* |
| LIQ_A | 242 | 384.4 | LIQ_C | 244 | 324.4 | LIQ_A /LIQ_C | 1.19 | 0.86* | 1.64* |
| LIQ_B | 260 | 418.8 | LIQ_C | 244 | 324.4 | LIQ_B /LIQ_C | 1.29 | 0.94* | 1.77* |

LIQ A = HRV vaccine liquid formulation Lot A LIQ B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = number of subjects with available results

95% CI = 95% Confidence Interval (one-way ANOVA model with pooled variance from the four groups)

L.L. = Lower Limit, U.L. = Upper Limit

\*The two-sided 95% CIs are within [0.5; 2] (the pre-defined clinical limit interval for consistency)

Template 13 Difference between groups in the percentage of subjects who seroconverted for anti-rotavirus IgA antibody 1-2 months after Dose 2 of the HRV vaccine – Per Protocol Analysis Set of Immunogenicity

| | | | | | Difference in seroconversion rate | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | 95 % ( | | | | | | | | |
| Group | N | % | Group | N | % | Difference | % | LL | UL |
| LIQPOOL | 746 | 88.6 | LY0 | 252 | 90.5 | LYO - LIQPOOL | 1.87 | -2.85 | 5.83* |

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects with available results

% = percentage of subjects who seroconverted at visit 3

95% CI = asymptotic standardised 95% Confidence Interval; LL = Lower Limit; UL = Upper Limit

\*Lower limit of the 95% Cl ≥-10% (the pre-defined clinical limit for non-inferiority)

Template 14 Ratio of anti-rotavirus IgA antibody GMCs 1-2 months after Dose 2 of the HRV vaccine between the HRV lyophilised vaccine group and the pooled HRV PCV-free liquid vaccine – Per Protocol Analysis Set of Immunogenicity

| | | | | | | GMC ratio | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% CI | | | |
| Group | N | GMC | Group | N | GMC | Ratio order | Value | LL | UL |
| LIQPOOL | 746 | 373.8† | LYO | 252 | 331.8 | LYO /LIQPOOL | 0.89 | 0.68 | 1.15* |

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects with available results

†geometric mean of the 3 GMC from the HRV liquid formulation groups

95% CI = 95% Confidence Interval (one-way ANOVA model using the group contrast between the HRV lyophilised formulation group and average of the HRV liquid formulation groups)

L.L. = Lower Limit, U.L. = Upper Limit

\*Lower limit of the 95% CI ≥ 0.67 (the pre-defined clinical limit for non-inferiority)

Template 15 Reverse cumulative distribution curve for anti-rotavirus IgA antibody concentrations at Visit 3 - Per Protocol Analysis Set of Immunogenicity



Template 16 Number and percentage of subjects who received study vaccine doses - Exposed Set

| | LIQ_A<br>N = 298 | | LIQ_B<br>N = 302 | | LIC<br>N = | )_C<br>300 | LY<br>N = | | Total<br>N = 1200 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Total number of doses received | n | % | n | % | n | % | n | % | n | % |
| 1 | 1 | 0.3 | 1 | 0.3 | 0 | 0.0 | 1 | 0.3 | 3 | 0.3 |
| 2 | 297 | 99.7 | 301 | 99.7 | 300 | 100 | 299 | 99.7 | 1197 | 99.8 |
| Anv | 298 | 100 | 302 | 100 | 300 | 100 | 300 | 100 | 1200 | 100 |

LIQ\_A = HRV vaccine Liquid formulation lot A

LIQ\_B = HRV vaccine Liquid formulation lot B

LIQ\_C = HRV vaccine Liquid formulation lot C

LYO = HRV vaccine lyophilised formulation

N = number of subjects in each group or in total included in the considered cohort

n (%) = number/percentage of subjects receiving the specified total number of doses

Any = number and percentage of subjects receiving at least one dose

# Template 17 Compliance in returning symptom sheets - Exposed Set

| Dose | GROUP | Number of doses | Doses NOT according to protocol | Number of general SS | Compliance<br>% general SS |
|---|---|---|---|---|---|
| 1 | LIQ_A | 298 | 10 | 298 | 100 |
| | LIQ_B | 302 | 7 | 302 | 100 |
| | LIQ_C | 300 | 6 | 300 | 100 |
| | LIQPOOL | 900 | 23 | 900 | 100 |
| | LYO | 300 | 6 | 299 | 99.7 |
| 2 | LIQ_A | 297 | 12 | 296 | 99.7 |
| | LIQ_B | 301 | 6 | 301 | 100 |
| | LIQ_C | 300 | 13 | 299 | 99.7 |
| | LIQPOOL | 898 | 31 | 896 | 99.8 |
| | LYO | 299 | 9 | 297 | 99.3 |
| Total | LIQ_A | 595 | 22 | 594 | 99.8 |
| | LIQ_B | 603 | 13 | 603 | 100 |
| | LIQ_C | 600 | 19 | 599 | 99.8 |
| | LIQPOOL | 1798 | 54 | 1796 | 99.9 |
| | LYO | 599 | 15 | 596 | 99.5 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

SS = Symptom sheets used for the collection of solicited AEs

Compliance % = (number of doses with symptom sheet return / number of administered doses) X 100

Doses not according to protocol = number of doses with regurgitation or vomiting

Template 18 Percentage of doses and of subjects reporting symptoms (solicited or unsolicited) reported during the 8-day (Day 0 to Day 7) follow-up period - Exposed Set

| | | | Any | symptom | | |
|-----------------|---------|------|------|---------|------|------|
| | | | | | 95% | % CI |
| | Group | N | n | % | LL | UL |
| Dose 1 | LIQ_A | 298 | 251 | 84.2 | 79.6 | 88.2 |
| | LIQ_B | 302 | 267 | 88.4 | 84.3 | 91.8 |
| | LIQ_C | 300 | 247 | 82.3 | 77.5 | 86.5 |
| | LIQPOOL | 900 | 765 | 85.0 | 82.5 | 87.3 |
| | LYO | 300 | 249 | 83.0 | 78.3 | 87.1 |
| Dose 2 | LIQ_A | 297 | 247 | 83.2 | 78.4 | 87.2 |
| | LIQ_B | 301 | 260 | 86.4 | 82.0 | 90.0 |
| | LIQ_C | 300 | 236 | 78.7 | 73.6 | 83.2 |
| | LIQPOOL | 898 | 743 | 82.7 | 80.1 | 85.2 |
| | LYO | 299 | 247 | 82.6 | 77.8 | 86.7 |
| Overall/dose | LIQ_A | 595 | 498 | 83.7 | 80.5 | 86.6 |
| | LIQ_B | 603 | 527 | 87.4 | 84.5 | 89.9 |
| | LIQ_C | 600 | 483 | 80.5 | 77.1 | 83.6 |
| | LIQPOOL | 1798 | 1508 | 83.9 | 82.1 | 85.5 |
| | LYO | 599 | 496 | 82.8 | 79.5 | 85.7 |
| Overall/subject | LIQ_A | 298 | 283 | 95.0 | 91.8 | 97.2 |
| _ | LIQ_B | 302 | 287 | 95.0 | 91.9 | 97.2 |
| | LIQ_C | 300 | 275 | 91.7 | 87.9 | 94.5 |
| | LIQPOOL | 900 | 845 | 93.9 | 92.1 | 95.4 |
| | LYO | 300 | 279 | 93.0 | 89.5 | 95.6 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

For each dose:

N = number of subjects having received the considered dose

n% = number/percentage of subjects reporting at least one symptom for the considered dose

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses followed by at least one symptom

For overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least one symptom

Template 19 Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, after each dose of the HRV lyophilised and HRV PCV-free liquid vaccine for all groups. - Exposed Set

| | | | L | IQ_A | | | | | LIQ_I | В | | | | LIQ | С | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 % | 6 CI | | | | 95 % | 6 CI | | | | | % CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| • | | | | u. | ļ. | Dos | se 1 | | | | | | | ļ. | ļ. | ļ. |
| Cough/runny | All | 298 | 72 | 24.2 | 19.4 | 29.4 | 302 | 90 | 29.8 | 24.7 | 35.3 | 300 | 71 | 23.7 | 19.0 | 28.9 |
| nose | Grade<br>3 | 298 | 1 | 0.3 | 0.0 | 1.9 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 62 | 20.8 | 16.3 | 25.9 | 302 | 76 | 25.2 | 20.4 | 30.5 | 300 | 49 | 16.3 | 12.3 | 21.0 |
| Diarrhoea | All | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 9 | 3.0 | 1.4 | 5.6 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| | Grade<br>3 | 298 | 3 | 1.0 | 0.2 | 2.9 | 302 | 2 | 0.7 | 0.1 | 2.4 | 300 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 9 | 3.0 | 1.4 | 5.6 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| Fever(°C) | All | 298 | 63 | 21.1 | 16.6 | 26.2 | 302 | 59 | 19.5 | 15.2 | 24.5 | 300 | 57 | 19.0 | 14.7 | 23.9 |
| | Grade<br>3 | 298 | 1 | 0.3 | 0.0 | 1.9 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 61 | 20.5 | 16.0 | 25.5 | 302 | 58 | 19.2 | 14.9 | 24.1 | 300 | | 18.3 | 14.1 | 23.2 |
| Irritability | All | 298 | 213 | 71.5 | 66.0 | 76.5 | 302 | 225 | 74.5 | 69.2 | 79.3 | 300 | | 63.7 | 57.9 | 69.1 |
| | Grade<br>3 | 298 | 12 | 4.0 | 2.1 | 6.9 | 302 | 17 | 5.6 | 3.3 | 8.9 | 300 | 9 | 3.0 | 1.4 | 5.6 |
| | Related | 298 | 203 | 68.1 | 62.5 | 73.4 | 302 | 220 | 72.8 | 67.5 | 77.8 | 300 | | | 55.6 | 66.9 |
| Loss of appetite | All | 298 | 79 | 26.5 | 21.6 | 31.9 | 302 | 79 | 26.2 | 21.3 | 31.5 | 300 | 73 | 24.3 | 19.6 | 29.6 |
| | Grade<br>3 | 298 | 0 | 0.0 | 0.0 | 1.2 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 75 | 25.2 | 20.3 | 30.5 | 302 | 78 | 25.8 | 21.0 | 31.2 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| Vomiting | All | 298 | 47 | 15.8 | 11.8 | 20.4 | 302 | 45 | 14.9 | 11.1 | 19.4 | 300 | 44 | 14.7 | 10.9 | 19.2 |
| | Grade<br>3 | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | 7 | 2.3 | 0.9 | 4.7 | 300 | 7 | 2.3 | 0.9 | 4.7 |
| | Related | 298 | 45 | 15.1 | 11.2 | 19.7<br><b>Dos</b> | 302<br>se <b>2</b> | 43 | 14.2 | 10.5 | 18.7 | 300 | 39 | 13.0 | 9.4 | 17.3 |
| Cough/runny | All | 297 | 92 | 31.0 | 25.8 | 36.6 | 301 | 104 | 34.6 | 29.2 | 40.2 | 300 | 95 | 31.7 | 26.4 | 37.3 |
| nose | Grade<br>3 | 297 | 2 | 0.7 | 0.1 | 2.4 | 301 | 2 | 0.7 | 0.1 | 2.4 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Related | 297 | 79 | 26.6 | 21.7 | 32.0 | 301 | 84 | 27.9 | 22.9 | 33.3 | 300 | 79 | 26.3 | 21.4 | 31.7 |
| Diarrhoea | All | 297 | 3 | 1.0 | 0.2 | 2.9 | 301 | 7 | 2.3 | 0.9 | 4.7 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| | Grade<br>3 | 297 | 1 | 0.3 | 0.0 | 1.9 | 301 | 2 | 0.7 | 0.1 | 2.4 | 300 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 297 | 3 | 1.0 | 0.2 | 2.9 | 301 | 7 | 2.3 | 0.9 | 4.7 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| Fever(°C) | All | 297 | 80 | 26.9 | 22.0 | 32.4 | 301 | 79 | 26.2 | 21.4 | 31.6 | | | 31.3 | 26.1 | 36.9 |
| | Grade<br>3 | 297 | 2 | 0.7 | 0.1 | 2.4 | 301 | 1 | 0.3 | 0.0 | 1.8 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 297 | 79 | 26.6 | 21.7 | 32.0 | 301 | 76 | 25.2 | 20.4 | 30.6 | | | 30.3 | 25.2 | 35.9 |
| Irritability | All | 297 | 201 | 67.7 | 62.0 | 73.0 | 301 | 224 | | 69.1 | | | | 67.3 | 61.7 | 72.6 |
| - | Grade<br>3 | 297 | 11 | 3.7 | 1.9 | 6.5 | 301 | 18 | 6.0 | 3.6 | 9.3 | 300 | | 4.7 | 2.6 | 7.7 |
| | Related | 297 | 195 | 65.7 | 60.0 | 71.0 | 301 | 220 | 73.1 | 67.7 | 78.0 | | 200 | | 61.0 | 72.0 |
| Loss of appetite | All | 297 | 69 | 23.2 | 18.5 | 28.5 | 301 | 63 | 20.9 | 16.5 | 26.0 | | | 23.3 | 18.7 | 28.5 |
| | Grade<br>3 | 297 | 1 | 0.3 | 0.0 | 1.9 | 301 | 0 | 0.0 | 0.0 | 1.2 | 300 | 0 | 0.0 | 0.0 | 1.2 |

115461 (ROTA-081) Statistical Analysis Plan Final

| | | | L | IQ_A | | | | | LIQ_E | 3 | | | | LIQ | С | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 % | 6 CI | | | | 95 % | 6 CI | | | | 95 9 | % CI |
| Symptom | Type | N | | | | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | Related | 297 | 67 | 22.6 | 17.9 | 27.7 | 301 | 59 | 19.6 | 15.3 | 24.5 | 300 | 68 | 22.7 | 18.1 | 27.8 |
| Vomiting | All | 297 | 43 | 14.5 | 10.7 | 19.0 | 301 | 40 | 13.3 | 9.7 | 17.7 | 300 | 33 | 11.0 | 7.7 | 15.1 |
| | Grade<br>3 | 297 | 7 | 2.4 | 1.0 | 4.8 | 301 | 8 | 2.7 | 1.2 | 5.2 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| | Related | 297 | 40 | 13.5 | 9.8 | 17.9 | 301 | 40 | 13.3 | 9.7 | 17.7 | 300 | 32 | 10.7 | 7.4 | 14.7 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = number of subjects having received the considered dose

n/% = number/percentage of subjects reporting the specified symptom for the considered dose

All = any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination

Grade 3 = any occurrence of the specified symptom rated as grade 3

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

Template 20 Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each dose in the pooled HRV PCV-free liquid vaccine group and the HRV vaccine lyophilised formulation group - Exposed Set

| | | | | LIQPO | OL | | | | LYO | ) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 9 | % CI | | | | 95 9 | % CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | | Dose 1 | | | | | | | |
| Cough/runny nose | All | 900 | 233 | 25.9 | 23.1 | 28.9 | 300 | 79 | 26.3 | 21.4 | 31.7 |
| | Grade 3 | 900 | 2 | 0.2 | 0.0 | 8.0 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Related | 900 | 187 | 20.8 | 18.2 | 23.6 | 300 | 64 | 21.3 | 16.8 | 26.4 |
| Diarrhoea | All | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Grade 3 | 900 | 7 | 8.0 | 0.3 | 1.6 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 3 | 1.0 | 0.2 | 2.9 |
| Fever(°C) | All | 900 | 179 | 19.9 | 17.3 | 22.6 | 300 | 68 | 22.7 | 18.1 | 27.8 |
| | Grade 3 | 900 | 2 | 0.2 | 0.0 | 8.0 | 300 | 0 | 0.0 | 0.0 | 1.2 |
| | Related | 900 | 174 | 19.3 | 16.8 | 22.1 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| Irritability | All | 900 | 629 | 69.9 | 66.8 | 72.9 | 300 | 207 | 69.0 | 63.4 | 74.2 |
| | Grade 3 | 900 | 38 | 4.2 | 3.0 | 5.7 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 900 | 607 | 67.4 | 64.3 | 70.5 | 300 | 201 | 67.0 | 61.4 | 72.3 |
| Loss of appetite | All | 900 | 231 | 25.7 | 22.8 | 28.7 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| | Grade 3 | 900 | 1 | 0.1 | 0.0 | 0.6 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 900 | 220 | 24.4 | 21.7 | 27.4 | 300 | 63 | 21.0 | 16.5 | 26.1 |
| Vomiting | All | 900 | 136 | 15.1 | 12.8 | 17.6 | 300 | 55 | 18.3 | 14.1 | 23.2 |
| | Grade 3 | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 11 | 3.7 | 1.8 | 6.5 |
| | Related | 900 | 127 | 14.1 | 11.9 | 16.6 | 300 | 51 | 17.0 | 12.9 | 21.7 |
| | | | | Dose 2 | | | | | | | |
| Cough/runny nose | All | 898 | 291 | 32.4 | 29.4 | 35.6 | 299 | 109 | 36.5 | 31.0 | 42.2 |
| | Grade 3 | 898 | 8 | 0.9 | 0.4 | 1.7 | 299 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 898 | 242 | 26.9 | 24.1 | 30.0 | 299 | 89 | 29.8 | 24.6 | 35.3 |
| Diarrhoea | All | 898 | 22 | 2.4 | 1.5 | 3.7 | 299 | 8 | 2.7 | 1.2 | 5.2 |
| | Grade 3 | 898 | 5 | 0.6 | 0.2 | 1.3 | 299 | 3 | 1.0 | 0.2 | 2.9 |
| | Related | 898 | 22 | 2.4 | 1.5 | 3.7 | 299 | 8 | 2.7 | 1.2 | 5.2 |
| Fever(°C) | All | 898 | 253 | 28.2 | 25.3 | 31.2 | 299 | 74 | 24.7 | 20.0 | 30.0 |
| | Grade 3 | 898 | 4 | 0.4 | 0.1 | 1.1 | 299 | 3 | 1.0 | 0.2 | 2.9 |
| | Related | 898 | 246 | 27.4 | 24.5 | 30.4 | 299 | 71 | 23.7 | 19.0 | 29.0 |
| Irritability | All | 898 | 627 | 69.8 | 66.7 | 72.8 | 299 | 200 | 66.9 | 61.2 | 72.2 |
| | Grade 3 | 898 | 43 | 4.8 | 3.5 | 6.4 | 299 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 898 | 615 | 68.5 | 65.3 | 71.5 | 299 | 196 | 65.6 | 59.9 | 70.9 |
| Loss of appetite | All | 898 | 202 | 22.5 | 19.8 | 25.4 | 299 | 62 | 20.7 | 16.3 | 25.8 |
| | Grade 3 | 898 | 1 | 0.1 | 0.0 | 0.6 | 299 | 0 | 0.0 | 0.0 | 1.2 |
| | Related | 898 | 194 | 21.6 | 19.0 | 24.4 | 299 | 60 | 20.1 | 15.7 | 25.1 |
| Vomiting | All | 898 | 116 | 12.9 | 10.8 | 15.3 | 299 | 41 | 13.7 | 10.0 | 18.1 |
| | Grade 3 | 898 | 23 | 2.6 | 1.6 | 3.8 | 299 | 11 | 3.7 | 1.9 | 6.5 |
| | Related | 898 | 112 | 12.5 | 10.4 | 14.8 | 299 | 40 | 13.4 | 9.7 | 17.8 |

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects having received the considered dose

n/% = number/percentage of subjects reporting the specified symptom for the considered dose

All = any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination Grade 3 = any occurrence of the specified symptom rated as grade 3

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

Template 21 Percentage of doses and subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, after each dose of the HRV lyophilised and HRV PCV-free HRV liquid vaccine for all groups. - Exposed Set

| | | LIQ_ | A | | | | LIQ | В | | | | LIQ | С | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 % | CI | | | | 95 % | CI | | | | 95 % | CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | | • | • | | ( | Overal | l/dos | е | • | | • | • | • | • | | • |
| Cough/runny nose | All | 595 | 164 | 27.6 | 24.0 | 31.3 | 603 | 194 | 32.2 | 28.5 | 36.1 | 600 | 166 | 27.7 | 24.1 | 31.4 |
| | Grade 3 | 595 | 3 | 0.5 | 0.1 | 1.5 | 603 | 2 | 0.3 | 0.0 | 1.2 | 600 | 5 | 0.8 | 0.3 | 1.9 |
| | Related | 595 | | 23.7 | 20.3 | 27.3 | | | 26.5 | 23.0 | 30.3 | 600 | | 21.3 | 18.1 | 24.8 |
| Diarrhoea | All | 595 | 11 | 1.8 | 0.9 | 3.3 | 603 | | 2.7 | 1.5 | 4.3 | 600 | 20 | 3.3 | 2.0 | 5.1 |
| | Grade 3 | 595 | 4 | 0.7 | 0.2 | 1.7 | 603 | | 0.7 | 0.2 | 1.7 | 600 | 4 | 0.7 | 0.2 | 1.7 |
| | Related | 595 | 11 | 1.8 | 0.9 | 3.3 | 603 | | 2.7 | 1.5 | 4.3 | 600 | 20 | 3.3 | 2.0 | 5.1 |
| Fever(°C) | All | 595 | | 24.0 | 20.7 | 27.7 | | | 22.9 | 19.6 | 26.4 | 600 | | 25.2 | 21.7 | 28.8 |
| | Grade 3 | 595 | 3 | 0.5 | 0.1 | 1.5 | 603 | | 0.2 | 0.0 | 0.9 | 600 | 2 | 0.3 | 0.0 | 1.2 |
| | Related | 595 | | 23.5 | 20.2 | 27.1 | | | 22.2 | 19.0 | 25.8 | 600 | | 24.3 | 21.0 | 28.0 |
| Irritability | All | 595 | | 69.6 | 65.7 | 73.3 | | | 74.5 | 70.8 | 77.9 | 600 | | 65.5 | 61.5 | 69.3 |
| , | Grade 3 | 595 | 23 | 3.9 | 2.5 | 5.7 | 603 | | 5.8 | 4.1 | 8.0 | 600 | 23 | 3.8 | 2.4 | 5.7 |
| | Related | 595 | | 66.9 | 62.9 | 70.7 | | 440 | | 69.2 | 76.5 | 600 | | 64.0 | 60.0 | 67.8 |
| Loss of appetite | All | 595 | | 24.9 | 21.4 | 28.6 | | | 23.5 | 20.2 | 27.1 | 600 | | 23.8 | 20.5 | 27.4 |
| | Grade 3 | 595 | 1 | 0.2 | 0.0 | 0.9 | 603 | | 0.0 | 0.0 | 0.6 | 600 | 1 | 0.2 | 0.0 | 0.9 |
| | Related | 595 | 142 | 23.9 | 20.5 | 27.5 | 603 | | | 19.4 | 26.3 | 600 | 135 | 22.5 | 19.2 | 26.1 |
| Vomiting | All | 595 | 90 | 15.1 | 12.3 | 18.3 | 603 | | 14.1 | 11.4 | 17.1 | 600 | 77 | 12.8 | 10.3 | 15.8 |
| | Grade 3 | 595 | 18 | 3.0 | 1.8 | 4.7 | 603 | | 2.5 | 1.4 | 4.1 | 600 | 15 | 2.5 | 1.4 | 4.1 |
| | Related | 595 | 85 | 14.3 | 11.6 | 17.4 | 603 | | 13.8 | 11.1 | 16.8 | 600 | 71 | 11.8 | 9.4 | 14.7 |
| | | | | | | verall/ | | | | | | | -1 | | 1 | |
| Cough/runny nose | All | 298 | 134 | 45.0 | 39.2 | 50.8 | | | 48.7 | 42.9 | 54.5 | 300 | 132 | 44.0 | 38.3 | 49.8 |
| | Grade 3 | 298 | 3 | 1.0 | 0.2 | 2.9 | 302 | 2 | 0.7 | 0.1 | 2.4 | 300 | 5 | 1.7 | 0.5 | 3.8 |
| | Related | 298 | 118 | 39.6 | 34.0 | 45.4 | | 125 | 41.4 | 35.8 | 47.2 | 300 | 108 | 36.0 | 30.6 | 41.7 |
| Diarrhoea | All | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | 15 | 5.0 | 2.8 | 8.1 | 300 | 19 | 6.3 | 3.9 | 9.7 |
| | Grade 3 | 298 | 4 | 1.3 | 0.4 | 3.4 | 302 | 4 | 1.3 | 0.4 | 3.4 | 300 | 3 | 1.0 | 0.2 | 2.9 |
| | Related | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | | 5.0 | 2.8 | 8.1 | 300 | 19 | 6.3 | 3.9 | 9.7 |
| Fever(°C) | All | 298 | 111 | 37.2 | 31.7 | 43.0 | 302 | 104 | 34.4 | 29.1 | 40.1 | 300 | 122 | 40.7 | 35.1 | 46.5 |
| ` , | Grade 3 | 298 | 3 | 1.0 | 0.2 | 2.9 | 302 | 1 | 0.3 | 0.0 | 1.8 | 300 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 298 | 109 | 36.6 | 31.1 | 42.3 | 302 | 100 | 33.1 | 27.8 | 38.7 | 300 | 118 | 39.3 | 33.8 | 45.1 |
| Irritability | All | 298 | 254 | 85.2 | 80.7 | 89.1 | 302 | 267 | 88.4 | 84.3 | 91.8 | 300 | 240 | 0.08 | 75.0 | 84.4 |
| - | Grade 3 | 298 | 20 | 6.7 | 4.1 | 10.2 | 302 | 31 | 10.3 | 7.1 | 14.3 | 300 | 21 | 7.0 | 4.4 | 10.5 |
| | Related | 298 | 252 | 84.6 | 80.0 | 88.5 | 302 | 265 | 87.7 | 83.5 | 91.2 | 300 | 238 | 79.3 | 74.3 | 83.8 |
| Loss of appetite | All | 298 | | 37.2 | 31.7 | 43.0 | | | 37.4 | 31.9 | 43.1 | 300 | | 37.0 | 31.5 | 42.7 |
| • • | Grade 3 | 298 | 1 | 0.3 | 0.0 | 1.9 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 106 | 35.6 | 30.1 | 41.3 | 302 | 108 | 35.8 | 30.4 | 41.5 | 300 | 109 | 36.3 | 30.9 | 42.1 |
| Vomiting | All | 298 | 70 | 23.5 | 18.8 | 28.7 | 302 | | 19.5 | 15.2 | 24.5 | 300 | 61 | 20.3 | 15.9 | 25.3 |
| | Grade 3 | 298 | 18 | 6.0 | 3.6 | 9.4 | 302 | | 4.0 | 2.1 | 6.8 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 298 | 69 | 23.2 | 18.5 | 28.4 | 302 | 58 | 19.2 | 14.9 | 24.1 | 300 | 58 | 19.3 | 15.0 | 24.3 |

115461 (ROTA-081) Statistical Analysis Plan Final

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses followed by the specified symptom

For overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once the specified symptom

All = any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination

Grade 3 = any occurrence of the specified symptom rated as grade 3

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

Template 22 Percentage of subjects with unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination in each HRV PCV-free vaccine liquid group - Exposed Set

| | | | | )_A<br>298 | | | | Q_B<br>302 | | | | Q_C<br>300 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 6 CI | | | | % CI | | | | % CI |
| Primary System Organ<br>Class (CODE) | Preferred<br>Term (CODE) | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | , | 24 | 8.1 | 5.2 | 11.7 | 26 | 8.6 | 5.7 | 12.4 | 33 | 11.0 | 7.7 | 15.1 |
| Ear and labyrinth | Ear pain | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| disorders (10013993) | (10014020) | | | | | | | | | | | | |
| Eye disorders (10015919) | Conjunctivitis<br>(10010741) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| Gastrointestinal disorders (10017947) | Diarrhoea<br>(10012735) | 0 | 0.0 | 0.0 | 1.2 | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 |
| | Flatulence<br>(10016766) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| General disorders and administration site conditions (10018065) | Injection site<br>erythema<br>(10022061) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Injection site pain (10022086) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Injection site<br>swelling<br>(10053425) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Irritability<br>(10022998) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| | Pyrexia<br>(10037660) | 4 | 1.3 | 0.4 | 3.4 | 3 | 1.0 | 0.2 | 2.9 | 4 | 1.3 | 0.4 | 3.4 |
| Immune system disorders (10021428) | Hypersensitivit y (10020751) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| Infections and infestations (10021881) | Bronchitis<br>(10006451) | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Ear infection (10014011) | 1 | 0.3 | 0.0 | 1.9 | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 |
| | Exanthema subitum (10015586) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Eye infection (10015929) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Gastroenteritis (10017888) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Impetigo<br>(10021531) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Influenza<br>(10022000) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Laryngitis<br>(10023874) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Otitis media<br>(10033078) | 5 | 1.7 | 0.5 | 3.9 | 6 | 2.0 | 0.7 | 4.3 | 11 | 3.7 | 1.8 | 6.5 |
| | Perianal<br>abscess<br>(10034447) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |

| | | | LIC | Q_A | | | LIC | )_B | usuca | /\li | | Q_C | 11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 298 | | | | 302 | | | | 300 | |
| | | | | | 6 CI | | | | % CI | | | | % CI |
| Primary System Organ<br>Class (CODE) | Preferred<br>Term (CODE) | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| Oldos (OODL) | Pneumonia<br>(10035664) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Respiratory<br>tract infection<br>(10062352) | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 |
| | Respiratory<br>tract infection<br>viral<br>(10062106) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Rhinitis<br>(10039083) | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 | 3 | 1.0 | 0.2 | 2.9 |
| | Upper<br>respiratory tract<br>infection<br>(10046306) | 2 | 0.7 | 0.1 | 2.4 | 5 | 1.7 | 0.5 | 3.8 | 7 | 2.3 | 0.9 | 4.7 |
| | Varicella<br>(10046980) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| Psychiatric disorders (10037175) | Crying (10011469) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| Respiratory, thoracic and mediastinal disorders (10038738) | Cough<br>(10011224) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 6 | 2.0 | 0.7 | 4.3 |
| | Nasal<br>congestion<br>(10028735) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Rales<br>(10037833) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| Skin and subcutaneous tissue disorders (10040785) | Dermatitis<br>allergic<br>(10012434) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Eczema<br>(10014184) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Rash<br>(10037844) | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once a specified unsolicited symptom

At least one symptom = number of subjects reporting at least one unsolicited symptom, whatever the MedDRA PT

<sup>95%</sup> CI = exact 95% Confidence Interval, LL = Lower Limit, UL = Upper Limit

Template 23 Percentage of doses with unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after vaccination in each HRV PCV-free liquid vaccine group - Exposed Set

| | | | | )_A<br>595 | | | | Q_B<br>= 603 | | | | Q_C<br>600 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <del>,</del> | | | | 6 CI | | | | % CI | | | 959 | % CI |
| Primary System Organ<br>Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | | 25 | 4.2 | 2.7 | 6.1 | 30 | 5.0 | 3.4 | 7.0 | 38 | 6.3 | 4.5 | 8.6 |
| Ear and labyrinth disorders (10013993) | Ear pain (10014020) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| Eye disorders<br>(10015919) | Conjunctivitis (10010741) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | 0 | 0.0 | 0.0 | 0.6 | 2 | 0.3 | 0.0 | 1.2 | 1 | 0.2 | 0.0 | 0.9 |
| , | Flatulence (10016766) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 2 | 0.3 | 0.0 | 1.2 |
| General disorders and administration site conditions (10018065) | Injection site erythema (10022061) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Injection site pain (10022086) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Injection site swelling (10053425) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Irritability (10022998) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | | 0.9 | 1 | 0.2 | 0.0 | 0.9 |
| | Pyrexia (10037660) | 4 | 0.7 | 0.2 | 1.7 | 3 | 0.5 | 0.1 | 1.4 | 4 | 0.7 | 0.2 | 1.7 |
| Immune system disorders (10021428) | Hypersensitivity (10020751) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| Infections and infestations (10021881) | Bronchitis (10006451) | 2 | 0.3 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| , | Ear infection (10014011) | 1 | 0.2 | 0.0 | 0.9 | 3 | 0.5 | 0.1 | 1.4 | 2 | 0.3 | 0.0 | 1.2 |
| | Exanthema subitum (10015586) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Eye infection (10015929) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Gastroenteritis (10017888) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Impetigo (10021531) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Influenza (10022000) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Laryngitis (10023874) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Otitis media (10033078) | 6 | 1.0 | 0.4 | 2.2 | 7 | 1.2 | 0.5 | 2.4 | 12 | 2.0 | 1.0 | 3.5 |
| | Perianal abscess<br>(10034447) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Pneumonia (10035664) | 0 | 0.0 | 0.0 | 0.6 | 1 | | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Respiratory tract infection (10062352) | 3 | 0.5 | 0.1 | 1.5 | 2 | | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 0.6 |
| | Respiratory tract infection viral (10062106) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Rhinitis (10039083) | 2 | 0.3 | 0.0 | 1.2 | 1 | | 0.0 | 0.9 | 3 | 0.5 | 0.1 | 1.5 |
| | Upper respiratory tract infection (10046306) | 2 | 0.3 | 0.0 | 1.2 | 6 | | 0.4 | 2.2 | 8 | 1.3 | 0.6 | 2.6 |
| <b>D</b> 11 (1 11 1 | Varicella (10046980) | 0 | 0.0 | 0.0 | 0.6 | 1 | | 0.0 | 0.9 | 2 | 0.3 | 0.0 | 1.2 |
| Psychiatric disorders (10037175) | Crying (10011469) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| Respiratory, thoracic and mediastinal disorders | Cough (10011224) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 6 | 1.0 | 0.4 | 2.2 |

115461 (ROTA-081) Statistical Analysis Plan Final

| | | | LIC<br>N = | )_A<br>595 | | | | Q_B<br>= 603 | | | | Q_C<br>600 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | 959 | % CI | | | 959 | % CI |
| Primary System Organ<br>Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| (10038738) | Nasal congestion (10028735) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Rales (10037833) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| Skin and subcutaneous tissue disorders | Dermatitis allergic<br>(10012434) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| (10040785) | Eczema (10014184) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Rash (10037844) | 2 | 0.3 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |

LIQ\_A = HRV vaccine liquid formulation Lot A

n/% = number/percentage of doses followed by at least one report of the specified unsolicited symptom
At least one symptom = number of doses followed by at least one report of an unsolicited symptom whatever the

MedDRA PT

95% CI = Exact 95% Confidence Interval; LL = Lower Limit, UL = Upper Limit

Template 24 Percentage of subjects reporting any GE episodes from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set

| Group | Ве | twee | - | se 1 and<br>ose 2 | before | Betv | veen | Dose | 2 and | Visit 3 | В | etwe | en Dos | se 1 and V | isit 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | Cl | | | | 95% | 6 CI | | | | 95% | 6 CI |
| | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| LIQ_A | 298 | 16 | 5.4 | 3.1 | 8.6 | 297 | 10 | 3.4 | 1.6 | 6.1 | 298 | 25 | 8.4 | 5.5 | 12.1 |
| LIQ_B | 302 | 17 | 5.6 | 3.3 | 8.9 | 301 | 15 | 5.0 | 2.8 | 8.1 | 302 | 29 | 9.6 | 6.5 | 13.5 |
| LIQ_C | 300 | 17 | 5.7 | 3.3 | 8.9 | 300 | 18 | 6.0 | 3.6 | 9.3 | 300 | 33 | 11.0 | 7.7 | 15.1 |
| LIQPOOL | 900 | 50 | 5.6 | 4.2 | 7.3 | 898 | 43 | 4.8 | 3.5 | 6.4 | 900 | 87 | 9.7 | 7.8 | 11.8 |
| LY0 | 300 | 8 | 2.7 | 1.2 | 5.2 | 299 | 15 | 5.0 | 2.8 | 8.1 | 300 | 22 | 7.3 | 4.7 | 10.9 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

Between Dose 1 and before Dose 2: N = number of subjects having received the first dose

Between Dose 2 and Visit 3: N = number of subjects having received the second dose

Between Dose 1 and Visit 3: N = number of subjects having received at least one dose

n/% = number/percentage of subjects reporting at least one gastroenteritis episode during the specified period

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = Total number of doses administered

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

# Template 25 Percentage of subjects reporting RV (vaccine strain or wild type RV) GE episodes from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set

| Group | Ве | twe | - | se 1 and<br>ose 2 | before | Ве | etwe | en Do | ose 2 and | Visit 3 | Be | twee | n Do | se 1 and | Visit 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | | 95% | 6 CI | | | | 95% | CI |
| | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| LIQ_A | 298 | 0 | 0.0 | 0.0 | 1.2 | 297 | 0 | 0.0 | 0.0 | 1.2 | 298 | 0 | 0.0 | 0.0 | 1.2 |
| LIQ_B | 302 | 1 | 0.3 | 0.0 | 1.8 | 301 | 0 | 0.0 | 0.0 | 1.2 | 302 | 1 | 0.3 | 0.0 | 1.8 |
| LIQ_C | 300 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| LIQPOOL | 900 | 1 | 0.1 | 0.0 | 0.6 | 898 | 1 | 0.1 | 0.0 | 0.6 | 900 | 2 | 0.2 | 0.0 | 0.8 |
| LYO | 300 | 0 | 0.0 | 0.0 | 1.2 | 299 | 0 | 0.0 | 0.0 | 1.2 | 300 | 0 | 0.0 | 0.0 | 1.2 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

Between Dose 1 and before Dose 2: N = number of subjects having received the first dose

Between Dose 2 and Visit 3: N = number of subjects having received the second dose

Between Dose 1 and Visit 3: N = number of subjects having received at least one dose

n/% = number/percentage of subjects reporting at least one RV GE episode during the specified period

# Template 26 Summary of RV GE episodes reported from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set

| Subject no | Onset of episode | Isolated RV type |
|------------|------------------|----------------------|
| PP | Day 3 of Dose 1 | G1/P8 vaccine strain |
| PΡ | Day 23 of Dose 2 | G1/P8 vaccine strain |

Template 27 Number and percentage of doses and of subjects who took at least one concomitant medication from Day 0 to Day 7 after vaccination by type in each HRV PCV-free vaccine liquid group - Exposed Set

| | | | LIQ_A | ١ | | | | LIQ_ | В | | | | LIQ_ | С | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | | 95% | 6 CI | | | | 959 | % CI |
| | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | | | • | Do | se 1 | | • | | | | | | |
| Any | 298 | 173 | 58.1 | 52.2 | 63.7 | 302 | 175 | 57.9 | 52.2 | 63.6 | 300 | 157 | 52.3 | 46.5 | 58.1 |
| Any antipyretic | 298 | 97 | 32.6 | 27.3 | 38.2 | 302 | 94 | 31.1 | 25.9 | 36.7 | 300 | 71 | 23.7 | 19.0 | 28.9 |
| Prophylactic | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 6 | 2.0 | 0.7 | 4.3 | 300 | 9 | 3.0 | 1.4 | 5.6 |
| antipyretic | | | | | | | | | | | | | | | |
| Any antibiotic | 298 | 6 | 2.0 | 0.7 | 4.3 | 302 | 5 | 1.7 | 0.5 | 3.8 | 300 | 5 | 1.7 | 0.5 | 3.8 |
| | | | | | | | se 2 | | | | | | | | |
| Any | 297 | 105 | 35.4 | 29.9 | 41.1 | 301 | 117 | 38.9 | 33.3 | 44.6 | 300 | 89 | 29.7 | 24.6 | 35.2 |
| Any antipyretic | 297 | 98 | 33.0 | 27.7 | 38.7 | 301 | 109 | 36.2 | 30.8 | 41.9 | 300 | 86 | 28.7 | 23.6 | 34.1 |
| Prophylactic | 297 | 7 | 2.4 | 1.0 | 4.8 | 301 | 8 | 2.7 | 1.2 | 5.2 | 300 | 6 | 2.0 | 0.7 | 4.3 |
| antipyretic | | | | | | | | | | | | | | | |
| Any antibiotic | 297 | 4 | 1.3 | 0.4 | 3.4 | 301 | 8 | 2.7 | 1.2 | 5.2 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | | | | | ( | Overa | ıll/do | se | | | | | | | |
| Any | 595 | 278 | 46.7 | 42.7 | 50.8 | 603 | 292 | 48.4 | 44.4 | 52.5 | 600 | 246 | 41.0 | 37.0 | 45.1 |
| Any antipyretic | 595 | 195 | 32.8 | 29.0 | 36.7 | 603 | 203 | 33.7 | 29.9 | 37.6 | 600 | 157 | 26.2 | 22.7 | 29.9 |
| Prophylactic | 595 | 15 | 2.5 | 1.4 | 4.1 | 603 | 14 | 2.3 | 1.3 | 3.9 | 600 | 15 | 2.5 | 1.4 | 4.1 |
| antipyretic | | | | | | | | | | | | | | | |
| Any antibiotic | 595 | 10 | 1.7 | 8.0 | 3.1 | 603 | 13 | 2.2 | 1.2 | 3.7 | 600 | 9 | 1.5 | 0.7 | 2.8 |
| | | | | | | veral | l/sub | ject | | | | | | | |
| Any | 298 | 194 | 65.1 | 59.4 | 70.5 | 302 | 205 | 67.9 | 62.3 | 73.1 | 300 | 182 | 60.7 | 54.9 | 66.2 |
| Any antipyretic | 298 | 130 | 43.6 | 37.9 | 49.5 | 302 | 141 | 46.7 | 41.0 | 52.5 | 300 | 111 | 37.0 | 31.5 | 42.7 |
| Prophylactic | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | 12 | 4.0 | 2.1 | 6.8 | 300 | 13 | 4.3 | 2.3 | 7.3 |
| antipyretic | | | | | | | | | | | | | | | |
| Any antibiotic | 298 | 10 | 3.4 | 1.6 | 6.1 | 302 | 13 | 4.3 | 2.3 | 7.2 | 300 | 9 | 3.0 | 1.4 | 5.6 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

For each dose and overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects who started to take the specified concomitant medication at least once during the mentioned period

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses after which the specified concomitant medication was started at least once during the mentioned period

Template 28 Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each documented dose in each HRV PCV-free liquid group - Exposed Set

| İ | | | | LIQ | _A | | | | LIQ | В | | | | LIQ | _C | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 9 | % CI | | | | 95 | % CI | | | | 95 | % CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| 1 | | | | | | Do | se 1 | | | | | | | | | |
| Cough/runny nose | All | 298 | | 24.2 | 19.4 | 29.4 | 302 | 90 | 29.8 | 24.7 | 35.3 | 300 | | 23.7 | 19.0 | 28.9 |
| l | Grade 3 | 298 | | 0.3 | 0.0 | 1.9 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | | 0.3 | 0.0 | 1.8 |
| l | Related | 298 | 62 | 20.8 | 16.3 | 25.9 | 302 | 76 | 25.2 | 20.4 | 30.5 | 300 | 49 | 16.3 | 12.3 | 21.0 |
| Diarrhoea | All | 298 | | 2.7 | 1.2 | 5.2 | 302 | | 3.0 | 1.4 | 5.6 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| l | Grade 3 | 298 | 3 | 1.0 | 0.2 | 2.9 | 302 | 2 | 0.7 | 0.1 | 2.4 | 300 | 2 | 0.7 | 0.1 | 2.4 |
| l | Related | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 9 | 3.0 | 1.4 | 5.6 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| Fever(°C) | All | 298 | 63 | 21.1 | 16.6 | 26.2 | 302 | 59 | 19.5 | 15.2 | 24.5 | 300 | 57 | 19.0 | 14.7 | 23.9 |
| <br>I | Grade 3 | 298 | 1 | 0.3 | 0.0 | 1.9 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| l | Related | 298 | 61 | 20.5 | 16.0 | 25.5 | 302 | 58 | 19.2 | 14.9 | 24.1 | 300 | 55 | 18.3 | 14.1 | 23.2 |
| Irritability | All | 298 | 213 | 71.5 | 66.0 | 76.5 | 302 | 225 | 74.5 | 69.2 | 79.3 | 300 | 191 | 63.7 | 57.9 | 69.1 |
| -<br>I | Grade 3 | 298 | 12 | 4.0 | 2.1 | 6.9 | 302 | 17 | 5.6 | 3.3 | 8.9 | 300 | 9 | 3.0 | 1.4 | 5.6 |
| l | Related | 298 | 203 | 68.1 | 62.5 | 73.4 | 302 | 220 | 72.8 | 67.5 | 77.8 | 300 | 184 | 61.3 | 55.6 | 66.9 |
| Loss of appetite | All | 298 | 79 | 26.5 | 21.6 | 31.9 | 302 | 79 | 26.2 | 21.3 | 31.5 | 300 | 73 | 24.3 | 19.6 | 29.6 |
| · · · | Grade 3 | 298 | 0 | 0.0 | 0.0 | 1.2 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| l | Related | 298 | | 25.2 | 20.3 | 30.5 | 302 | 78 | 25.8 | 21.0 | 31.2 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| Vomiting | All | 298 | 47 | 15.8 | 11.8 | 20.4 | 302 | 45 | 14.9 | 11.1 | 19.4 | 300 | 44 | 14.7 | 10.9 | 19.2 |
| | Grade 3 | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | 7 | 2.3 | 0.9 | 4.7 | 300 | 7 | 2.3 | 0.9 | 4.7 |
| l | Related | 298 | | 15.1 | 11.2 | 19.7 | 302 | 43 | 14.2 | 10.5 | 18.7 | 300 | 39 | 13.0 | 9.4 | 17.3 |
| | | | | ļ. | | Do | se 2 | | | | | | | | | - |
| Cough/runny nose | All | 296 | 92 | 31.1 | 25.9 | 36.7 | 301 | 104 | 34.6 | 29.2 | 40.2 | 299 | 95 | 31.8 | 26.5 | 37.4 |
| | Grade 3 | 296 | 2 | 0.7 | 0.1 | 2.4 | 301 | 2 | 0.7 | 0.1 | 2.4 | 299 | 4 | 1.3 | 0.4 | 3.4 |
| l | Related | 296 | 79 | 26.7 | 21.7 | 32.1 | 301 | 84 | 27.9 | 22.9 | 33.3 | 299 | 79 | 26.4 | 21.5 | 31.8 |
| Diarrhoea | All | 296 | 3 | 1.0 | 0.2 | 2.9 | 301 | 7 | 2.3 | 0.9 | 4.7 | 299 | 12 | 4.0 | 2.1 | 6.9 |
| l | Grade 3 | 296 | 1 | 0.3 | 0.0 | 1.9 | 301 | 2 | 0.7 | 0.1 | 2.4 | 299 | 2 | 0.7 | 0.1 | 2.4 |
| l | Related | 296 | 3 | 1.0 | 0.2 | 2.9 | 301 | 7 | 2.3 | 0.9 | 4.7 | 299 | 12 | 4.0 | 2.1 | 6.9 |
| Fever(°C) | All | 296 | 80 | 27.0 | 22.1 | 32.5 | 301 | 79 | 26.2 | 21.4 | 31.6 | 299 | 94 | 31.4 | 26.2 | 37.0 |
| , <i>,</i> | Grade 3 | 296 | 2 | 0.7 | 0.1 | 2.4 | 301 | 1 | 0.3 | 0.0 | 1.8 | 299 | 1 | 0.3 | 0.0 | 1.8 |
| l | Related | | | 26.7 | 21.7 | 32.1 | 301 | 76 | 25.2 | 20.4 | 30.6 | 299 | | 30.4 | 25.3 | 36.0 |
| Irritability | All | 296 | 201 | 67.9 | 62.3 | 73.2 | 301 | | 74.4 | 69.1 | 79.3 | 299 | 202 | 67.6 | 61.9 | 72.8 |
| | Grade 3 | 296 | 11 | 3.7 | 1.9 | 6.6 | 301 | 18 | 6.0 | 3.6 | 9.3 | 299 | 14 | 4.7 | 2.6 | 7.7 |
| 1 | Related | | | 65.9 | 60.2 | 71.3 | 301 | 220 | 73.1 | 67.7 | 78.0 | | 200 | 66.9 | 61.2 | 72.2 |
| Loss of appetite | All | 296 | | 23.3 | 18.6 | 28.6 | 301 | | 20.9 | 16.5 | 26.0 | | | 23.4 | 18.7 | 28.6 |
| 11 - | Grade 3 | | | 0.3 | 0.0 | 1.9 | 301 | | 0.0 | 0.0 | 1.2 | 299 | | 0.0 | 0.0 | 1.2 |
| 1 | Related | 296 | | 22.6 | 18.0 | 27.8 | | 59 | 19.6 | 15.3 | 24.5 | 299 | | 22.7 | 18.1 | 27.9 |
| Vomiting | All | 296 | | 14.5 | 10.7 | 19.1 | 301 | | 13.3 | 9.7 | 17.7 | 299 | | 11.0 | 7.7 | 15.1 |
| - <b>J</b> | Grade 3 | | | 2.4 | 1.0 | 4.8 | | 8 | 2.7 | 1.2 | 5.2 | 299 | | 2.7 | 1.2 | 5.2 |
| ì | Related | | | 13.5 | 9.8 | 17.9 | | 40 | 13.3 | 9.7 | 17.7 | 299 | | 10.7 | 7.4 | 14.8 |

LIQ\_A = HRV vaccine liquid formulation Lot A

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = number of subjects with the considered documented dose

n/% = number/percentage of subjects reporting the specified symptom for the considered dose

<sup>95%</sup> CI = Exact 95% Confidence Interval; LL = Lower Limit, UL = Upper Limit

Grade 3 = any occurrence of the specified symptom rated as grade 3

# Template 29 Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort)

| Study-<br>Subject<br>No. | Country | Gender | AE Description | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|
| PP<br>D | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |
| PP<br>D | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |

# Template 30 Subjects with Serious Adverse Events reported up to Visit 3 - Exposed Set

| Sub | Countr | • | | Verbatim | Preferred | - | | | | | Causalit | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | у | onset<br>(Week | X | | term | Organ<br>Class | typ<br>e | е | of | n | у | |
| | | `) | | | | | | | onse | | | |
| Р | US | Р | М | Kawasaki' | Kawasaki' | Infections | НО | 1 | τ<br>12 | 29 | N | Recovered/resolve |
| Р | | P | | | s disease | and infestation | | | | | | d |
| | | | | | | S | | | | | | |

MA = medical attention

HO = hospitalisation

Dose = dose given prior to the start of the SAE

Day of onset = number of days since last study vaccine dose

Template 31 Number (%) of subjects with serious adverse events from Dose 1 up to study end, including number of events reported (Exposed Set)

| | | | | Gr<br>N = | - | | Gr.<br>N | _ |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System Organ<br>Class | Preferred Term<br>(CODE) | n* | n | % | n* | n | % |
| SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

Gr 1 = Group 1 description

Gr 2 = Group 2 description

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

Template 32 Solicited and unsolicited symptoms experienced by at least 5 % of subjects classified by MedDRA Primary System Organ Class and Preferred Term within 31-day (Days 0-30) post-vaccination period after any dose of HRV PCV-free liquid vaccine - SAE excluded (Exposed Set)

| | | HPV_2D<br>N = | | | MMR_DTPa<br>N = | | |
|---|---|---|---|---|---|---|---|
| <b>Primary System Organ Class (CODE)</b> | Preferred Term (CODE) | n* | n | % | n* | n | % |
| At least one symptom | | | | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

# Template 33 Number of subjects by country

| | ACWY-TT<br>N = 259 | ACWYHPV<br>N = 259 | HPV<br>N = 261 | Co-ad<br>N = 260 | Tdap<br>N = 261 | Total<br>N = 1300 |
|---|---|---|---|---|---|---|
| Country | n | n | N | n | n | n |
| Dominican Republic | 86 | 87 | 88 | 87 | 87 | 435 |
| Estonia | 87 | 86 | 87 | 87 | 88 | 435 |
| Thailand | 86 | 86 | 86 | 86 | 86 | 430 |

ACWY-TT = Subjects who received MenACWY-TT at Month 0 and Cervarix at Month 1, 2 and 7

ACWYHPV = Subjects who received MenACWY-TT and Cervarix at Month 0 and Cervarix at Month 1 and 6

HPV = Subjects who received Cervarix at Month 0, 1 and 6

Co-ad = Subjects who received MenACWY-TT, Cervarix and Boostrix at Month 0 and Cervarix at Month 1 and 6 Tdap = Subjects who received Boostrix and Cervarix at Month 0 and Cervarix at Month 1 and 6

N = number of subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories

115461 (ROTA-081) Statistical Analysis Plan Final

# Template 34 Number of enrolled subjects by age category (Exposed Set)

| | | Gr 1<br>N = | Gr 2<br>N = | Gr 3<br>N = | Total<br>N = |
|---|---|---|---|---|---|
| Characteristics | Categories | n | n | n | n |
| Age category | In utero | | | | |
| | Preterm newborn infants | | | | |
| | (gestational age < 37 wks) | | | | |
| | Newborns (0-27 days) | | | | |
| | Infants and toddlers (28 days- | | | | |
| | 23 months) | | | | |
| | Children (2-11 years) | | | | |
| | Adolescents (12-17 years) | | | | |
| | Adults (18-64 years) | | | | |
| | From 65-84 years | | | | |
| | 85 years and over | | | | |
| | Missing | | | | |

Gr 1 = Group 1 description

Gr 2 = Group 2 description

Gr 3 = Group 3 description

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = <describe missing>

# Template 35 Study population (Exposed Set)

| Number of subjects | [each group] | Total |
|---|---|---|
| Planned, N | | |
| Randomised, N ( <total cohort="" vaccinated="">)</total> | | |
| Completed, n (%) | | |
| Demographics | | |
| N ( <total cohort="" vaccinated="">)</total> | | |
| Females:Males | | |
| Mean Age, <years> (SD)</years> | | |
| Median Age, <years> (minimum, maximum)</years> | | |
| <most category="" frequent="" of="" race="">, n (%)</most> | | |
| Second most frequent category of race>, n (%) | | |
| <third category="" frequent="" most="" of="" race="">, n (%)</third> | | |

[each group]:

Short group label= long group label

# 115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

| | | Statistical Analysis Plan Amendment 1 Final |
|---|---|---|
| <b>gsk</b> GlaxoSmithKline | | Statistical Analysis Plan |
| Detailed Title: | A phase IIIA, randomised, observer-blind, multi-centre study to evaluate the clinical consistency of three production lots of the Porcine circovirus (PCV)-free liquid formulation of GlaxoSmithKline (GSK) Biologicals' oral live attenuated human rotavirus (HRV) vaccine and to evaluate the PCV-free liquid formulation of GSK Biologicals' HRV vaccine as compared to the currently licensed lyophilised formulation of the HRV vaccine in terms of immunogenicity, reactogenicity and safety when administered as a two-dose vaccination in healthy infants starting at age 6-12 weeks. | |
| eTrack study number and Abbreviated Title | 115461 (R | ROTA-081) |
| Scope: | All data pertaining to the above study. Note that this analysis plan does not cover analyses devoted to iDMC. A separate SAP is available for the iDMC analyses. | |
| Date of Statistical Analysis<br>Plan | | ent 1 Final: 05-Feb-2018 |
| Co-ordinating authors: | manager) | (study statistician); PPD (Stat |
| Reviewed by: | PPD PPD Lead) PPD PPD PPD PPD | (Clinical and Epidemiology Project Lead) (Clinical Research and Development (Lead statistician) (peer reviewer statistician), (Lead statistical analyst) (Lead Scientific writer) |
| Approved by: | PPD<br>PPD<br>PPD<br>PPD | (Regulatory Affair) (Clinical Safety representative) (Public Disclosure) (Clinical and Epidemiology Project Lead) |
| rippioved by. | PPD Lead) PPD PPD PPD | (Clinical and Epidemiology Project Lead) (Clinical Research and Development (Lead statistician) (Lead statistical analyst) (Scientific writer) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | ABBREVIATIONS | 9 |
| 1. | DOCU | JMENT HISTORY | 10 |
| 2. | STUD | Y DESIGN | 10 |
| 3. | OBJE | CTIVES | 14 |
| ٠. | 3.1. | Co-Primary | |
| | 3.2. | | |
| 4. | ENDF | POINTS | 15 |
| | 4.1. | Primary | 15 |
| | 4.2. | Secondary | |
| 5. | ANAL | YSIS SETS | 16 |
| | 5.1. | Definitions | |
| | | 5.1.1. Exposed Set | 16 |
| | | 5.1.2. Per-Protocol analysis Set of immunogenicity (PPS) | 16 |
| | 5.2. | Criteria for eliminating data from analyses sets | |
| | | 5.2.1. Elimination from Exposed set (ES) | |
| | | 5.2.2. Elimination from Per-Protocol analysis Set (PPS) | |
| | | 5.2.3. Right censored Data | |
| | | 5.2.4. Visit-specific censored Data | 18 |
| | 5.3. | Important protocol deviation not leading to elimination from per-<br>protocol analysis set | 19 |
| 6. | СТДТ | ISTICAL ANALYSES | 10 |
| 0. | 6.1. | Demography | |
| | 0.1. | 6.1.1. Analysis of demographics/baseline characteristics planned | |
| | | in the protocol | |
| | 6.2. | | |
| | 0.2. | Exposure | |
| | | 6.2.2. Additional considerations | |
| | 6.3. | Immunogenicity | |
| | 0.0. | 6.3.1. Analysis of immunogenicity planned in the protocol | |
| | | 6.3.1.1. Within groups assessment | |
| | | 6.3.1.2. Between groups assessment | |
| | | 6.3.1.3. Statistical Methods | |
| | | 6.3.2. Additional considerations | |
| | 6.4. | Analysis of safety | |
| | | 6.4.1. Analysis of safety planned in the protocol | |
| | | 6.4.2. Additional considerations | |
| 7. | ANAL | YSIS INTERPRETATION | 24 |
| 8. | СОИГ | DUCT OF ANALYSES | 25 |
| ٥. | 8 1 | Sequence of analyses | 25 |

| | | | | 15461 (ROTA-081) |
|---|---|---|---|---|
| | | | Statistical Analysis Plan | Amendment 1 Final |
| | | 8.1.1. | Final analysis up to Visit 3: | 25 |
| | 8.2. | Final ana | ılysis | |
| | 8.3. | | l considerations for interim analyses | |
| 9. | CHAN | GES FRO | M PLANNED ANALYSES | 26 |
| 10. | LIST C | F FINAL | REPORT TABLES, LISTINGS AND FIGURES | 26 |
| 11. | ANNE)<br>METH | | DARD DATA DERIVATION RULE AND STATISTI | |
| | 11 1 | | I Method References | 26 |
| | | | Date derivation | |
| | | 11.1.2. | Dose number | |
| | | 11.1.3. | Demography | |
| | | 11.1.4. | Immunogenicity | |
| | | 11.1.5. | Safety | |
| | | 11.1.6. | Management of missing data | |
| | | 11.1.7. | Data presentation description | |
| 12. | ANNE | X 2: SUMI | MARY ON ELIMINATION CODES | 30 |
| 13. | ANNE | X 3: STUE | DY SPECIFIC MOCK TFL | 31 |

# 115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

# **LIST OF TABLES**

| | | PAGE |
|---------|---------------------------------------------------|------|
| Table 1 | Study groups and epoch foreseen in the study | 11 |
| Table 2 | Study groups and treatments foreseen in the study | 11 |
| Table 3 | Blinding of study epoch | 12 |

115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

# **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Sequence for evaluating the study objectives in order to control | |
| | the overall type I error below 2.5% | <mark>24</mark> |

115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

# **LIST OF TEMPLATES**

| | | PAGE |
|---|---|---|
| Template 1 | Minimum and maximum activity dates (Exposed Set) | 31 |
| Template 2 | Number of subjects enrolled by center - Exposed Set | 31 |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal entire study period- Exposed Set | 32 |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Exposed Set) | 33 |
| Template 5 | Number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses with reasons for exclusion | 34 |
| Template 6 | Summary of demographic characteristics (Per Protocol Analysis Set of Immunogenicity) | 35 |
| Template 7 | Deviations from specifications for age and intervals between study visits - Exposed Set | 36 |
| Template 8 | Summary of co-administered vaccination by dose - Exposed Set | 37 |
| Template 9 | Summary of vaccinations other than HRV vaccine administered from birth until Visit 3, excluding vaccination given on the day of HRV doses - Exposed Set | 37 |
| Template 10 | Anti-rotavirus IgA antibody GMC and seroconversion rates – Per Protocol Analysis Set of Immunogenicity | 38 |
| Template 11 | Anti-rotavirus IgA antibody GMC calculated on subjects seropositive for anti-rotavirus IgA antibodies – Per Protocol Analysis Set of Immunogenicity | 38 |
| Template 12 | Ratio of anti-rotavirus IgA antibody GMCs 1-2 months after Dose 2 of the HRV vaccine between each pair of the three lots of the HRV PCV-free liquid vaccine — Per Protocol Analysis Set of Immunogenicity | 39 |
| Template 13 | Difference between groups in the percentage of subjects who seroconverted for anti-rotavirus IgA antibody 1-2 months after Dose 2 of the HRV vaccine – Per Protocol Analysis Set of Immunogenicity | 39 |
| Template 14 | Ratio of anti-rotavirus IgA antibody GMCs 1-2 months after Dose 2 of the HRV vaccine between the HRV lyophilised vaccine group and the pooled HRV PCV-free liquid vaccine — Per Protocol Analysis Set of Immunogenicity | 39 |

115461 (ROTA-081)

| | Statistical Analysis Plan Amendment 1 | Final |
|---|---|---|
| Template 15 | Reverse cumulative distribution curve for anti-rotavirus IgA antibody concentrations at Visit 3 - Per Protocol Analysis Set of Immunogenicity | 40 |
| Template 16 | Number and percentage of subjects who received study vaccine doses - Exposed Set | 40 |
| Template 17 | Compliance in returning symptom sheets - Exposed Set | 41 |
| Template 18 | Percentage of doses and of subjects reporting symptoms (solicited or unsolicited) reported during the 8-day (Day 0 to Day 7) follow-up period - Exposed Set | 42 |
| Template 19 | Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, after each dose of the HRV lyophilised and HRV PCV-free liquid vaccine for all groups Exposed Set | 43 |
| Template 20 | Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each dose in the pooled HRV PCV-free liquid vaccine group and the HRV vaccine lyophilised formulation group - Exposed Set | 45 |
| Template 21 | Percentage of doses and subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, after each dose of the HRV lyophilised and HRV PCV-free HRV liquid vaccine for all groups. - Exposed Set | 46 |
| Template 22 | Percentage of subjects with unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination in each HRV PCV-free vaccine liquid group - Exposed Set | 48 |
| Template 23 | Percentage of doses with unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after vaccination in each HRV PCV-free liquid vaccine group - Exposed Set | <b>5</b> 0 |
| Template 24 | Percentage of subjects reporting any GE episodes from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set | 51 |
| Template 25 | Percentage of subjects reporting RV (vaccine strain or wild type RV) GE episodes from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set | 52 |
| Template 26 | Summary of RV GE episodes reported from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set | 52 |

| 115461 | (ROTA-081 |
|--------|-----------|
|--------|-----------|

| | Statistical Analysis Plan Amendment 1 | , |
|---|---|---|
| Template 27 | Number and percentage of doses and of subjects who took at least one concomitant medication from Day 0 to Day 7 after vaccination by type in each HRV PCV-free vaccine liquid group - Exposed Set | |
| Template 28 | Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each documented dose in each HRV PCV-free liquid group - Exposed Set | 54 |
| Template 29 | Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort) | 55 |
| Template 30 | Subjects with Serious Adverse Events reported up to Visit 3 - Exposed Set | 55 |
| Template 31 | Number (%) of subjects with serious adverse events from Dose 1 up to study end, including number of events reported (Exposed Set) | <b>5</b> 5 |
| Template 32 | Solicited and unsolicited symptoms experienced by at least 5 % of subjects classified by MedDRA Primary System Organ Class and Preferred Term within 31-day (Days 0-30) post-vaccination period after any dose of HRV PCV-free liquid vaccine - SAE excluded (Exposed Set) | 56 |
| Template 33 | Number of subjects by country | 56 |
| Template 34 | Number of enrolled subjects by age category (Exposed Set) | 57 |
| Template 35 | Study population (Exposed Set) | 57 |

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

#### LIST OF ABBREVIATIONS

AE Adverse event

ANOVA Analysis of Variance

cDISCI Clinical Data Interchange Standards Consortium

CI Confidence Interval
CRF Case Report Form

CTRS Clinical Trial Registry Summary

EL.U/ml ELISA unit per milliliter

Eli Type Internal GSK database code for type of elimination code

ELISA Enzyme-linked immunosorbent assay

ES Exposed Set
GE Gastroenteritis
GSK GlaxoSmithKline

iDMC Independent Data Monitoring Committee

IU/ml International units per milliliter

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not Applicable

PD Protocol Deviation

PPS Per Protocol Set

RV RotaVirus

SAE Serious adverse event SAP Statistical Analysis Plan

SAS Statistical Analysis Software

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 30 May 2017 | first version | Amendment 1 (09March |
| | | 2017) |
| 05 Feb 2018 | Amendment 1: the derivation of gastroenteritis | Amendment 1 (09March |
| | was added in section 6.4.2. | 2017) |

#### 2. STUDY DESIGN



N: Number of subjects planned to be enrolled, n = number of subjects in each group

Review of the safety data for the first 800 enrolled subjects (50% of total enrolment) will be conducted as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available for 800 subjects.

Protocol waivers or exemptions are not allowed with the exception of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the outline of study procedures (Section 5.5 of protocol), are essential and required for study conduct.

<sup>\*</sup> Contact (by telephone call or any other convenient procedure) for the safety follow-up will take place 6 months after the last dose of HRV vaccine.

<sup>\*\*</sup> Two oral doses of the study vaccines will be administered at an approximate 1-month or 2-months interval to subjects, according to the immunisation schedule for RV vaccine administration in participating countries.

<sup>#</sup>Blood samples will be taken before the first dose and 1 to 2 months after the second dose.

<sup>\$</sup> An IDMC will review the safety data for the first 80 enrolled subjects (5% of total enrolment) and first 160 enrolled subjects (10% of total enrolment) as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available. Enrolment will be paused when first 10% of the subjects are enrolled for the purpose of the IDMC review of the safety data and will only resume if the outcome of the IDMC review is positive.

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

- Experimental design: Phase IIIA, observer-blind, randomised (1:1:1:1), controlled, multi-centric, with four parallel groups and a staggered enrolment (Part A and Part B).
- Duration of the study: The intended duration of the study, per subject, will be approximately 7-8 months including the 6 months of extended safety follow-up period after the last dose of HRV vaccine.
  - Epoch 001: Primary starting at Visit 1 (Day 0) and ending at the safety follow-up contact (Month 7-8).
- Primary completion Date (PCD): Visit 3 (Month 2-4).

Refer to protocol glossary for the definition of PCD.

• End of Study (EoS): Last testing results released of samples collected at Visit 3 or Last Subject Last Visit (LSLV) (Follow up contact at month 7-8).

Refer to protocol glossary for the definition of EoS.

• Study groups: The study groups and epoch foreseen in the study are provided in Table 1.

Table 1 Study groups and epoch foreseen in the study

| Study Groups | Number of subjects | Age at Dose 1 (Min-Max) | Epoch<br>Epoch 001 |
|---|---|---|---|
| Liq_A | 400 | 6 weeks-12 weeks | • |
| Liq_B | 400 | 6 weeks-12 weeks | • |
| Liq_C | 400 | 6 weeks-12 weeks | • |
| Lyo | 400 | 6 weeks-12 weeks | • |

The study groups and treatments foreseen in the study are given in Table 2.

Table 2 Study groups and treatments foreseen in the study

| | Vaccina nama | | | Study Groups | |
|-----------------|----------------|-------|-------|--------------|-----|
| Treatment name | Vaccine name | Liq_A | Liq_B | Liq_C | Lyo |
| HRV Liquid | HRV PCV-free ‡ | Х | Х | Х | |
| HRV Lyophilised | HRV * | | | | Х |

<sup>‡</sup>PCV-free HRV liquid vaccine

- PCV-free HRV liquid formulation lot A (also referred to as Liq A group)
- PCV-free HRV liquid formulation lot B (also referred to as Liq B group)
- PCV-free HRV liquid formulation lot C (also referred to as Liq C group)
- GSK Biologicals' currently licensed lyophilised HRV formulation (also referred to as Lyo group)

<sup>\*</sup> Licensed formulation of HRV lyophilised vaccine

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

- Control: active control-GSK Biologicals' currently licensed lyophilised HRV vaccine.
- Vaccination schedule: Two doses of HRV vaccine to be administered according to a
  0, 1-2 month schedule according to the immunisation schedule for RV vaccine
  administration in participating countries.
  - Concomitant administration of routine childhood vaccines will be allowed according to local immunisation practices in each participating country.
- Treatment allocation: Randomised 1:1:1:1 using GSK Biologicals' central randomisation system on Internet (SBIR).
- Blinding: observer-blind

The blinding in the study is given in Table 3.

Table 3 Blinding of study epoch

| Study Epoch | Blinding* |
|-------------|----------------|
| Epoch 001 | Double-blind |
| Epoch 001 | Observer-blind |

<sup>\*</sup>Double blind for the three lots of PCV-free HRV liquid vaccine and observer-blind for the liquid formulation versus the lyophilised formulation.

- Sampling schedule: Blood samples will be collected from all subjects at Visit 1 and Visit 3 to measure serum anti-RV IgA antibody concentrations using Enzyme Linked Immunosorbent Assay (ELISA).
- Recording of GE episodes: Any GE episodes occurring from Dose 1 of HRV vaccine up to Visit 3 will be recorded for all subjects in the diary card. Parents/Legally Acceptable Representative(s) (LARs) will be instructed to collect stool sample(s) if the subject develops GE during the period from Dose 1 of HRV vaccine up to Visit 3. A stool sample should be collected as soon as possible after illness begins and preferably not later than 7 days after the start of GE symptoms. Two occurrences of diarrhoea will be classified as separate episodes if there will be five or more diarrhoea-free days between the episodes. Refer to the protocol glossary for definitions of GE and diarrhoea.
- Recording of Solicited AEs: Solicited AEs (fever, fussiness/irritability, loss of appetite, cough/runny nose, diarrhoea and vomiting) occurring between the day of each HRV vaccine dose and the following 7 days (Day 0-Day 7) will be recorded daily using diary cards for all subjects.
- Recording of Unsolicited AEs: Unsolicited AEs occurring within 31 days (Day 0-Day 30) after each dose of HRV vaccine will be recorded using diary cards for all subjects.
- Recording of SAEs: SAEs will be recorded from Visit 1 (Day 0) up to 6 months after Dose 2 of HRV vaccine.
- Type of study: self-contained
- Data collection: Electronic Case Report Form (eCRF)
115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

• Safety monitoring: An IDMC comprising of clinical experts and a biostatistician, will review the safety data accrued during the study and the details of the review will be described in an IDMC charter. The IDMC review will happen after enrolment of 5%, 10% and 50% of subjects. The IDMC review will happen at the following stages:

Review of all safety data for the first 80 enrolled subjects (5% of total enrolment) as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available for 80 subjects.

- any available data beyond 8 days post Dose 2 will also be reviewed.
- during this IDMC review, enrolment of subjects will continue.

Review of all safety data for the first 160 enrolled subjects (10% of total enrolment) as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available for 160 subjects.

- any available data beyond 8 days post Dose 2 will also be reviewed.
- until this IDMC review, enrolment of subjects will pause. Enrolment will resume only if no safety concerns are raised by IDMC.

Review of all safety data for the first 800 enrolled subjects (50% of total enrolment) as soon as data until 8 days post Dose 2 (Day 0-Day 7) are available for 800 subjects.

- any available data beyond 8 days post Dose 2 will also be reviewed.
- during this IDMC review, enrolment of subjects will continue.

Statistical Analysis Plan Amendment 1 Final

### 3. OBJECTIVES

# 3.1. Co-Primary

• To demonstrate the lot-to-lot consistency of the PCV-free liquid HRV vaccine in terms of immunogenicity as measured by serum anti-RV IgA antibody concentrations 1-2 months after Dose 2.

Consistency will be demonstrated if, for all pairs of lots, the two-sided 95% confidence intervals (CIs) for the ratio of anti-RV IgA antibody GMCs 1-2 months after Dose 2 are within the [0.5; 2] clinical limit interval.

• To demonstrate the immunological non-inferiority of PCV-free liquid HRV vaccine as compared to the currently licensed lyophilised HRV vaccine in terms of seroconversion rates 1-2 months after Dose 2.

Non-inferiority will be demonstrated if the lower limit of the two-sided asymptotic standardized 95% CI for the difference in seroconversion rate between the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and licensed lyophilised HRV vaccine is greater than or equal to -10%.

• To demonstrate the non-inferiority of the PCV-free liquid HRV vaccine to that of the currently licensed lyophilised HRV vaccine in terms of serum anti-RV IgA antibody concentrations 1-2 months after Dose 2.

Non-inferiority will be demonstrated if the lower limit of the two-sided 95% CI for the ratio of anti-RV IgA antibody GMCs 1-2 months after Dose 2 between the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and the lyophilised HRV vaccine is greater than or equal to 0.67.

### 3.2. Secondary

### Reactogenicity and safety

- To evaluate the reactogenicity of the liquid HRV vaccine and currently licensed lyophilised HRV vaccine in terms of solicited AEs during the 8 days (Day 0-Day 7) follow-up period after each vaccination.
- To assess the safety of the study vaccines in terms of unsolicited AEs during the 31 days (Day 0-Day 30) follow-up period after each vaccination and Serious Adverse Events (SAEs) during the entire study period.

### **Immunogenicity**

• To assess the immunogenicity of the PCV-free liquid HRV vaccine and the currently licensed lyophilised HRV vaccine, in terms of percentage of subjects with anti-RV IgA antibody concentrations ≥ 90 U/mL 1-2 months after Dose 2.

### 4. ENDPOINTS

## 4.1. Primary

- Evaluation of immunogenicity in terms of anti-RV antibody concentrations
  - Serum anti-RV IgA antibody concentrations expressed as GMCs 1-2 months after Dose 2 in each of the HRV liquid formulation groups (Liq\_A, Liq\_B and Liq\_C).
  - Anti-RV IgA antibody seroconversion rate\* 1-2 months after Dose 2 in the lyophilised and pooled liquid groups.
  - Serum anti-RV IgA antibody concentrations expressed as GMCs 1-2 months after Dose 2 in the lyophilised and pooled liquid groups.

## 4.2. Secondary

- Solicited adverse events
  - Occurrence of each general solicited symptom within the 8 days (Day 0-Day 7) follow-up period after each dose of the lyophilised and PCV-free HRV liquid vaccine
- Unsolicited adverse events.
  - Occurrence of unsolicited AEs within 31 days (Day 0-Day 30) after any dose of HRV vaccine, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification.
- Serious adverse events
  - Occurrence of serious adverse events from Dose 1 up to study end.
- Evaluation of immunogenicity in terms of anti-RV antibody concentrations.
  - Serum anti-RV IgA antibody concentrations ≥ 90 U/mL 1-2 months after Dose 2 in the lyophilised and pooled liquid groups.

<sup>\*</sup>Seroconversion rate is defined as the percentage of subjects who were initially seronegative (i.e., with anti-RV IgA antibody concentration < 20 U/mL prior the first dose of HRV vaccine) and developed anti-RV IgA antibody concentration  $\ge 20$  U/mL at Visit 3.

### 5. ANALYSIS SETS

### 5.1. Definitions

### 5.1.1. Exposed Set

The ES will include all subjects with at least one study vaccine administration documented:

- a safety analysis based on the ES will include all vaccinated subjects,
- an immunogenicity analysis based on the ES will include all vaccinated subjects for whom immunogenicity data are available.

The ES analysis will be performed per treatment actually administered at dose 1.

### 5.1.2. Per-Protocol analysis Set of immunogenicity (PPS)

The PPS for immunogenicity will include all subjects from the ES:

- who have received all doses of study vaccine,
- for whom the HRV vaccine liquid or lyophilised formulation was administered according to protocol and subjects did not regurgitate after vaccination,
- who have not received a vaccine prohibited by the protocol up to Visit 3,
- for whom the randomisation code has not been broken
- who were seronegative for serum anti-RV IgA antibodies on the day of Dose 1
- who have not received medication prohibited by the protocol up to Visit 3 as listed in Section 6.7.2 of the study protocol,
- whose underlying medical condition was not prohibited by the protocol up to Visit 3 as listed in Section 6.8 of the study protocol,
- who comply with the vaccination schedule (Table 5 of the study protocol),
- who comply with blood sampling schedule (Table 5 of the study protocol),
- for whom immunogenicity data are available at the post-vaccination sampling time point,
- who have no RV other than vaccine strain in Gastroenteritis (GE) stool samples collected up to Visit 3,
- who have no concomitant infection unrelated to the vaccine up to Visit 3, which may influence the immune response.

## 5.2. Criteria for eliminating data from analyses sets

## 5.2.1. Elimination from Exposed set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES.

# 5.2.2. Elimination from Per-Protocol analysis Set (PPS)

A subject will be excluded from the PPS analysis under the following conditions

| Code | Decode => Condition under which the code is used |
|---|---|
| 900 | Questionable subject => subjects with invalid informed consent or fraudulent data Study vaccine dose not administrated but subject number allocated => subjects enrolled but not vaccinated |
| 1040 | Administration of vaccine(s) forbidden in the protocol => Administration of a vaccine not foreseen by the study protocol and administered during the period starting from 30 days before the first vaccination and ending at Visit 3, with the exception of the inactivated influenza vaccine, which is allowed at any time during the study, and other licensed routine childhood vaccinations. |
| 1060 | Randomisation code broken at the investigator site => Subjects unblinded in SBIR or unblinding reported as protocol deviation |
| 1070 | <ul> <li>Study vaccine dose not administered according to protocol =&gt;</li> <li>Subjects vaccinated with the correct vaccine but who regurgitated for one of the 2 doses;</li> </ul> |
| | • subjects for whom the second administered dose is not aligned with the first dose (e.g. lyo as second dose after a first dose with liquid from lot A; or liquid from lot B as second dose after a first dose with liquid from lot A) |
| | • Subject who did not receive the second dose and return to visit 3 blood sample |
| | Subject who was given multiple doses at one visit |
| | Route of vaccination which is not oral |
| 1080 | Vaccine temperature deviation => Subjects who have received a vaccine which had a temperature deviation qualified as inappropriate for use by Quality Assurance. |
| 1090 | Expired vaccine administered => Subjects who received an expired vaccine |

# 115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

| | Statistical Analysis Flatt Amendment 11 mai |
|---|---|
| Code | Decode => Condition under which the code is used |
| 2010 | Protocol violation (inclusion/exclusion criteria) => Ineligible subjects who was vaccinated (i.e. Age at dose 1 is not between 42-90 days, gestational age is < 37 weeks 0 day or > 41 weeks 6 days or other eligibility criteria – see section 4.2 and 4.3 of the protocol) |
| 2020 | Initially seropositive or initially unknown antibody status = > Anti-HRV concentration ≥ 20 U/mL or unknown at pre-dose 1 blood sample |
| 2040 | Administration of any medication forbidden by the protocol => administration of |
| | <ul> <li>Any investigational or non-registered product (drug or vaccine) other than the study vaccines used between Visit 1 and Visit 3 during the study period.</li> <li>Immunosuppressants or other immune-modifying drugs administered chronically (i.e., more than 14 days) during the study period between Visit 1 to Visit 3. For corticosteroids, this will mean prednisone (0.5 mg/kg/day, or equivalent). Inhaled and topical steroids are allowed.</li> <li>Immunoglobulins and/or any blood products administered during the study period between Visit 1 to Visit 3.</li> <li>Long-acting immune-modifying drugs administered at any time during the</li> </ul> |
| | study period (e.g., infliximab). |
| 2060 | Concomitant infection related to the vaccine which may influence immune response => Subjects with non-vaccine type RV detected in GE stool samples that may impact immunogenicity at Visit 3. |
| 2070 | Concomitant infection not related to the vaccine which may influence immune response = > Condition that has the capability of altering their immune response at visit 3 such autoimmune disease. |
| 2080 | Non-compliance with vaccination schedule (including wrong and unknown dates ) => Subjects who did not comply with the interval for dose 2 (Dose 2 should be between 28-83 days after Dose 1). |
| 2090 | Non-compliance with blood sampling schedule (including wrong and unknown dates => Subjects who did not comply with the blood sample interval (blood sample post dose 2 should be between 28-83 days after Dose 2); subjects with a blood sample at visit 3 and without a second HRV vaccine administered |
| 2100 | Essential serological data missing => Anti-HRV results not available post-vaccination |
| 2120 | Obvious incoherence or abnormality or error in data => subjects without blood sample at visit 3 for whom a sample post-vaccination is found. |

#### 5.2.3. **Right censored Data**

Not applicable

#### 5.2.4. Visit-specific censored Data

Not applicable

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

- Forced randomization: In case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event.
- Manual randomization: In case the randomization system is unavailable, the investigator has the option to perform randomization by selecting supplies available at the site according to a pre-defined rule. In case the randomization system is available, a vaccine different from the randomized treatment may have been administered at dose 1.
- Short follow-up: subjects with a safety follow-up period after the last dose of HRV vaccine that is less than 180 days.
- Vaccinated subjects without documentation of solicited symptoms i.e. for a vaccine dose administered, at least one solicited symptom is not documented as being present or absent.

### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in Annex 1 and will not be repeated below. All Confidence Interval (CI) will be two-sided 95% CI.

# 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The following calculations will be performed for each group and for the pooled liquid vaccine group:

- The distribution of subjects enrolled among the study centres and countries will be tabulated as a whole and for each group.
- The numbers of subjects who withdraw from the study will be tabulated by group according to the reason for drop-out.
- The deviations from specifications for age and intervals between study visits will be tabulated by group.
- The median, mean, range and standard deviation of age (in weeks) at each HRV vaccine dose and of the gestational age will be computed by group. The median, mean and standard deviation of height (in centimetres) and weight (in kilograms) at

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

Visit 1 will be computed by group. The racial and sex composition will be presented. These calculations will also be performed by country.

• Summary of co-administered vaccinations (i.e., vaccinations given on the day of each HRV vaccine dose) and intercurrent vaccinations (i.e., vaccinations from birth up to Visit 3, excluding vaccination given on the day of HRV vaccine doses) will be summarized by group for the ES.

### 6.1.2. Additional considerations

All demography summaries will be generated for the ES. The summary of age, height, weight, race and sex will also be provided for the PPS. Number and reason for elimination from PPS will be tabulated by group. Summary of important protocol deviations not leading to elimination will be provided by groups for the PPS.

### 6.2. Exposure

### 6.2.1. Analysis of exposure planned in the protocol

Not applicable

### 6.2.2. Additional considerations

The number of doses administered will be tabulated for each group.

# 6.3. Immunogenicity

### 6.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the PPS for analysis of immunogenicity. If, in any vaccine group, the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is 5% or more, a second analysis based on the ES will be performed to complement the PPS analysis.

### 6.3.1.1. Within groups assessment

The following calculations will be performed for each group and for the pooled liquid vaccine group.

- For each group, at each time point that anti-rotavirus IgA is measured,
  - Seropositivity/seroconversion rates and their exact 95% CI will be computed,
  - Percentage of subjects with anti-RV IgA antibody concentrations ≥ 90 U/mL and their exact 95% CI will be computed.
  - GMCs and their 95% CIs will be computed.
- The above mentioned descriptive analyses will also be performed by country.

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

• The distribution of anti-RV IgA antibody concentrations at Visit 3 will be displayed using Reverse Cumulative Curves (RCCs).

### 6.3.1.2. Between groups assessment

- The 95% CI for the ratio of anti-RV IgA antibody GMCs at Visit 3 between any pair of the three lots of the HRV liquid vaccine will be computed (first co-primary objective).
- The asymptotic standardized 95% CI for the difference in seroconversion rate at Visit 3 between the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and lyophilised HRV vaccine will be computed (second co-primary objective).
- The 95% CI for the ratio of anti-RV IgA antibody GMCs at Visit 3 between the PCV-free liquid HRV vaccine (pooled HRV liquid groups) and lyophilised HRV vaccine will be computed (third co-primary objective).

### 6.3.1.3. Statistical Methods

- The exact CIs for a proportion within a group will be calculated using SAS [see section 11.1].
- The standardized asymptotic CI for the group difference in proportion will be calculated using SAS [see section 11.1].
- The CI for GMCs will be obtained within each group separately. The CI for the mean of log-transformed concentration will be first obtained assuming that log-transformed values were normally distributed with unknown variance. The CI for the GMCs will then be obtained by exponential-transformation of the CI for the mean of log-transformed concentration.
- The GMC group ratio will be obtained using an ANOVA model on the logarithm-transformed concentrations. The ANOVA model will include the vaccine group and the country as fixed effects. The GMC ratio and their 95% CI will be derived by exponential-transformation of the corresponding group contrast in the model.

### 6.3.2. Additional considerations

The ANOVA model for the lot-to-lot GMC ratio will include the data from the 3 HRV liquid groups only.

The country effect for the ANOVA model will be accounted by country indicator variables that will be treated as continuous variable in order to obtain adjusted GMCs that reflect the distribution of subjects between countries.

Summaries planned per countries will be limited to the PPS. These summaries will also be generated by frequent race and by gender. Note that a race category is considered if it includes more than 40 subjects. Infrequent race categories will be combined together and summarized if it includes more than 40 subjects.

Statistical Analysis Plan Amendment 1 Final

### 6.4. Analysis of safety

### 6.4.1. Analysis of safety planned in the protocol

The ES will be used for the analysis of safety.

The following calculations will be performed for each group and for the pooled liquid vaccine group:

The percentage of doses and of subjects reporting at least one symptom (solicited or unsolicited) during the 8 days (Day 0-Day 7) solicited follow-up period post vaccination will be computed, along with exact 95% CI. The same calculations will be done for symptoms (solicited or unsolicited) rated as grade 3 in intensity and for symptoms (solicited or unsolicited) assessed as causally related to vaccination.

The percentage of doses and of subjects reporting each individual solicited general symptom will be computed, over the 8 days (Day 0-Day 7) solicited follow-up period post vaccination, along with exact 95% CI. The same calculations will be done for each individual general solicited symptom rated as grade 3 in intensity, for each individual solicited general symptom assessed as causally related to vaccination and those that resulted in a medically attended visit.

The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to MedDRA. Every verbatim term will be matched with the appropriate Preferred Term. The percentage of subjects with unsolicited AEs occurring within 31 days (Day 0-Day 30) follow-up period after any dose with its exact 95% CI will be tabulated by group, and by preferred term. Similar tabulation will be done for unsolicited AEs rated as grade 3, for unsolicited AEs with causal relationship to vaccination and those that resulted in a medically attended visit.

The percentage of subjects reporting GE episodes from Dose 1 of HRV vaccine up to Visit 3 will be tabulated by group.

The percentage of subjects with presence of RV in GE stool samples collected from Dose 1 of HRV vaccine up to Visit 3 will be tabulated by group.

The percentage of GE episodes with no available stool results from Dose 1 of HRV vaccine up to Visit 3 will be tabulated.

The percentage of subjects who started taking at least one concomitant medication from HRV vaccination to Day 7 after vaccinations will be tabulated with exact 95% CI. The percentages of subjects who started taking at least one concomitant medication during the study period will be tabulated with exact 95% CI.

SAEs reported during the study period will be described in detail.

Statistical Analysis Plan Amendment 1 Final

### 6.4.2. Additional considerations

As indicated in section 10.5 of the protocol and in line with the project history, analysis of safety will be primarily performed per dose administered and subjects who missed reporting symptoms (solicited/unsolicited or concomitant medications) will be treated as subjects without symptoms (solicited/unsolicited or concomitant medications, respectively). A sensitivity analysis will be performed on documented doses i.e. accounting only for doses where solicited symptoms are indicated as being absent/present in case more than 5% of the doses are not documented.

Summary of temperature will be provided by  $0.5^{\circ}$  increment (i.e.  $\geq 38.0^{\circ}$ C, >38.5; >39, >39.5, >40).

Gastroenteritis is assumed to take place when either:

- a stool collection is reported
- three or more than 3 loose stools are reported as solicited diarrhoea symptom.
- an unsolicited symptom, which has an onset date more than 7 days after vaccination (i.e. with onset day > 8), is associated with the high lever MedDRA terms hereunder but excluding Diarrhoea as primary preferred term (10012735): 'Gastric and gastroenteric infections' (10017887), 'Gastrointestinal infections, site unspecified' (10017968), 'Intestinal infections (10022678)', 'Faecal, abnormalities NEC' (10016097), 'Diarrhoea (excl infective)' (10012736).

Summary of solicited symptoms will also be provided by country, gender and frequent race(s) while summary of unsolicited symptoms within 31 days post-vaccination will be provided by country – see section 6.3.2 for the definition of frequent race.

Summary of solicited symptoms will also be provided for each individual general solicited symptom causally related to vaccination and rated as grade 3 in intensity. Likewise the percentage of subjects and of doses with grade 3 causally related unsolicited AEs occurring within 31 days (Day 0-Day 30) follow-up period after any dose with its exact 95% CI will be tabulated by group, and by preferred term. These summaries will not be provided by country, gender or frequent race(s).

Note that the study will be converted in cDISC. Accordingly Day 0-Day 7 and Day 0-Day 30 will be replaced by Day 1-Day 8 and Day 1-Day 31 for the statistical analysis.

### 7. ANALYSIS INTERPRETATION

Except for analyses addressing criteria specified in the co-primary objectives referred as confirmatory analyses, all the analyses will be descriptive/exploratory in nature. The use of these descriptive/exploratory analyses should be limited to support the confirmatory analyses or to generate hypothesis.

To control the overall type I error below 2.5%, the confirmatory objectives will be evaluated using a hierarchical procedure as shown in Figure 1. A confirmatory objective will be reached if the associated criteria are met and the previous objectives have been met.

Figure 1 Sequence for evaluating the study objectives in order to control the overall type I error below 2.5%



### 8. CONDUCT OF ANALYSES

# 8.1. Sequence of analyses

Safety data that is as clean as possible will be analysed for IDMC review. Details of the review are described in an IDMC charter.

### 8.1.1. Final analysis up to Visit 3:

An analysis will be conducted once all the study data up to Visit 3 are available and cleaned and Rota-IgA ELISA testing at 1-2 month post-dose 2 has been fully completed. The Clinical Study Report (CSR) with data up to Visit 3 will be used for the registration of PCV-free liquid vaccine in European Union (EU) and 'rest of world' countries.

The study report will include the following:

- All analysis of the serum anti-RV IgA antibody concentrations, 1-2 months after Dose 2 in the lyophilised and pooled liquid groups.
- All analyses of safety up to visit 3 and analysis of SAEs and AEs leading to drop out based on the database lock for the analysis.

# 8.2. Final analysis

If the previous analysis does not cover all study data, the study report will be amended when all data will be available. The study report amendment will include the additional safety information

The following table provides the plan for analyses excluding analyses dedicated to IDMC

| Description | Analysis<br>ID | Disclosure Purpose (IN=internal, CTRS=public posting, SR=study report and public posting) | Dry run<br>review<br>needed (Y/N) | Study Headline<br>Summary<br>(SHS)requiring<br>expedited<br>communication<br>to upper<br>management<br>(Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final analysis up to Visit 3 | E1_05 | SR | Yes | Yes | TFL TOC first<br>version – All TFLs<br>as per database<br>lock date |
| Final | E1_01 | SR | No | Yes | TFL TOC first version - All TFLs |

# 8.3. Statistical considerations for interim analyses

All confirmatory analyses will be conducted for the Final analysis up to Visit 3 and therefore no statistical adjustment for interim analyses is required.

### 9. CHANGES FROM PLANNED ANALYSES

Not applicable

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS,...). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The mock tables referred under column named 'layout' can be found in Annex 3 of this SAP.

The following group names will be used in the TFLs, to be in line with the T-domains:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | Liq_A | PCV-free HRV liquid vaccine - lot A |
| 2 | Liq_B | PCV-free HRV liquid vaccine - lot B |
| 3 | Liq_C | PCV-free HRV liquid vaccine - lot C |
| 4 | Liq pooled | PCV-free HRV liquid vaccine - Pooled Lot |
| 5 | Lyo | HRV Lyophilised vaccine |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

### 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413.

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper: Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890. The standardised asymptotic method used is the method six.

#### 11.1.1. **Date derivation**

- SAS date derived from a character date: in case day is missing, pp is used. In case day & month are missing, pp is used.
- Onset day for an event (ae, medication, vaccination, ...): the onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 1 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.

#### 11.1.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered and an event occurs after the subsequent study dose (e.g. 2<sup>nd</sup> study dose), the relative dose of the event will be study dose associated to the subsequent study dose (e.g. dose 2).
- The number of doses for a product is the number of time the product was administered to a subject.
- The incidence per dose is the number of vaccination visits at which an event was reported among all vaccination visits.

#### 11.1.3. Demography

Age: Age at the reference activity, computed as the number of complete weeks between the date of birth and the reference activity.

Conversion of weight to kg: the following conversion rule is used:

Weight in Kilogram= weight in Pounds / 2.2

Weight in Kilogram = weight in ounces / 35.2

The result is rounded to 2 decimals.

Conversion of height to cm: the following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48

Height in Centimetres = Height in Inch \* 2.54

The result is rounded to the unit (i.e. no decimal).

Statistical Analysis Plan Amendment 1 Final

Conversion of temperature to °C: the following conversion rule is used:

Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9 The result is rounded to 1 decimal.

### 11.1.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced.
- The Geometric Mean Concentrations (GMCs) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in Section 5.7.3 of the protocol.
- A seronegative subject is a subject whose antibody concentration is below the cut-off value of the assay. A seropositive subject is a subject whose antibody concentration is greater than or equal to the cut-off value of the assay.
- The assay cut-off is the value under which there is no quantifiable result available. For an assay with a specific 'cut\_off', numerical immuno result is derived from a character field (rawres):
  - If rawres is 'NEG' or '-' or '(-)', numeric result= cut off/2,
  - if rawres is 'POS' or '+' or '(+)', numeric result = cut off,
  - if rawres is '< value' and value<=cut off, numeric result =cut off/2,
  - if rawres is '< value' and value>cut off, numeric result =value,
  - if rawres is '> value' and value<cut off, numeric result =cut off/2,
  - if rawres is '> value' and value>=cut off, numeric result =value,
  - if rawres is '<= value' or '>= value' and value<cut\_off, numeric result =cut\_off/2,</p>
  - if rawres is '<= value' or '>= value' and value>=cut off, numeric result =value,
  - if rawres is a value < cut off, numeric result = cut off/2,
  - if rawres is a value >= cut off, numeric result = rawres,
  - if rawres is a value >= cut off, numeric result = rawres,
  - else numeric result is left blank

### 11.1.5. Safety

- For analysis of solicited, unsolicited adverse events (such as serious adverse events or adverse events by primary MedDRA term) and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report the event or the concomitant medication will be considered as subjects without the event or the concomitant medication respectively.
- In case there will be more than 5% of subjects without documented dose for solicited symptoms (i.e., symptom screen not completed), sensitivity analysis will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed).

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

- The following rules will be used for the analysis of solicited symptoms:
  - Subject who didn't document the presence or absence of a solicited symptom
    after one dose will be considered not having that symptom after that dose in the
    analysis done on "administrated dose"
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
  - Subjects who documented the presence of a solicited symptom and fully or
    partially recorded daily measurement over the solicited period will be included in
    the summaries at that dose and classified according to their maximum observed
    daily recording over the solicited period.
  - Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be considered as having that symptom after that dose).
- For the analysis, temperatures will be coded as follows for oral, axillary or tympanic route:

| Grade | Temperature |
|-------|---------------------|
| 0 | < 38.0°C |
| 1 | ≥ 38.0°C - ≤ 38.5°C |
| 2 | > 38.5°C - ≤ 39.5°C |
| 3 | > 39.5°C |

• Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for<br>Vaccination phase | N used for deriving % per dose for<br>Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited general symptom | Primary analysis: all subjects with study vaccine administered Sensitivity analysis as applicable (see section 6.4.2): all subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) | Primary analysis: all study visits with study vaccine administered Sensitivity analysis: all study visits with study vaccine administered and with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

Statistical Analysis Plan Amendment 1 Final

For summaries by MedDRA primary preferred term combining solicited and unsolicited adverse events, solicited adverse events will be coded as per the following MedDRA codes

| Solicited symptom | Lower level term code | Corresponding |
|------------------------|-----------------------|------------------|
| | | Lower level term |
| | | decode |
| Fever | 10016558 | Fever |
| Irritability/Fussiness | 10022998 | Irritability |
| Diarrhoea | 10012727 | Diarrhoea |
| Vomiting | 10047700 | Vomiting |
| Loss of appetite | 10003028 | Appetite lost |
| Cough/runny nose | 10011224 | Cough |

### 11.1.6. Management of missing data

### **Demography:**

• For a given subject and a given demographic variable, missing measurements will not be replaced.

### **Immunogenicity:**

• For a given subject and a given immunogenicity measurement time point, missing or non-evaluable measurements will not be replaced.

### Reactogenicity and safety:

• Subjects who missed reporting symptoms (solicited/unsolicited or concomitant medications) will be treated as subjects without symptoms (solicited/unsolicited or concomitant medications, respectively).

### 11.1.7. Data presentation description

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| All summaries | % of count, including LL & UL of CI | 1 |
| Demographic characteristics | Mean, median, SD | 1 |
| Immunogenicity | % of difference, including LL & UL of CI | 2 |
| Immunogenicity | GMC group ratio, including LL & UL of CI | 2 |
| Immunogenicity | Anti-RV IgA GMC | 1 |

### 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to Section 5.2.

### 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following draft study specific mock TFLs will be used.

The data display, title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

These templates were copied from ROTA-061 and additional tables required for public disclosure were added. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

Note that all tables will include the pooled lot group for HRV liquid as shown in Template 2.

Template 1 Minimum and maximum activity dates (Exposed Set)

| Visit | Minimum date | Maximum date |
|-------|--------------|--------------|
| 1 | 19JUN2007 | 29DEC2007 |
| 2 | 24JUL2007 | 08FEB2008 |
| 3 | 24AUG2007 | 18MAR2008 |
| 4 | 25MAR2008 | 22NOV2008 |
| 5 | 24MAR2009 | 31MAR2009* |

<sup>\*</sup>Database Lock Date = 31MAR2009

Template 2 Number of subjects enrolled by center - Exposed Set

| | | LIQ_A | LIQ_B | LIQ_C | LIQ_pool | LYO | Total | |
|---------|--------|-------|-------|-------|----------|-----|-------|------|
| Country | Center | r n | n | n | n | n | n | % |
| XXXX | PPD | 38 | 38 | 38 | | 37 | 151 | 12.6 |
| | PPD | 20 | 20 | 20 | | 20 | 80 | 6.7 |
| | PPD | 30 | 30 | 29 | | 29 | 118 | 9.8 |
| | PPD | 19 | 19 | 20 | | 20 | 78 | 6.5 |
| | All | | | | | | | |
| YYYYY | PPD | 15 | 15 | 15 | | 15 | 60 | 5.0 |
| | PPD | 22 | 22 | 23 | | 22 | 89 | 7.4 |
| | PPD | 35 | 36 | 36 | | 35 | 142 | 11.8 |
| | PPD | 28 | 28 | 28 | | 28 | 112 | 9.3 |
| | PPD | 20 | 21 | 20 | | 21 | 82 | 6.8 |
| | PPD | 22 | 23 | 22 | | 23 | 90 | 7.5 |
| | PPD | 22 | 23 | 22 | | 23 | 90 | 7.5 |
| | PPD | 27 | 27 | 27 | | 27 | 108 | 9.0 |
| | All | | | | | | | |
| All | All | 298 | 302 | 300 | | 300 | 1200 | 100 |

<sup>&</sup>lt;group description >

n = number of subjects included in each group or in total for a given center or for all centers All = sum of all subjects in each group or in total (sum of all groups)

 $<sup>% =</sup> n/AII \times 100$ 

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

Template 3 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal entire study period- Exposed Set

| | LIQ_A | LIQ_B | LIQ_C | LYO | Total |
|---|---|---|---|---|---|
| Number of subjects vaccinated | 298 | 302 | 300 | 300 | 1200 |
| Number of subjects completed | 297 | 301 | 298 | 297 | 1193 |
| Number of subjects withdrawn | 1 | 1 | 2 | 3 | 7 |
| Reasons for withdrawal : | | | | | |
| Serious Adverse Event | 0 | 0 | 0 | 1 | 1 |
| Non-serious adverse event | 0 | 0 | 0 | 0 | 0 |
| Protocol violation | 0 | 0 | 0 | 0 | 0 |
| Consent withdrawal (not due to an adverse event) | 1 | 0 | 1 | 2 | 4 |
| Migrated/moved from study area | 0 | 1 | 1 | 0 | 2 |
| Lost to follow-up (subjects with incomplete vaccination course) | 0 | 0 | 0 | 0 | 0 |
| Lost to follow-up (subjects with complete vaccination course) | 0 | 0 | 0 | 0 | 0 |
| Others | 0 | 0 | 0 | 0 | 0 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LYO = HRV vaccine lyophilised formulation

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed study visit 3

Withdrawn = number of subjects who did not come for study visit 3

115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

# Number of subjects at each visit and list of withdrawn subjects (Exposed Set) Template 4

| Group | VISIT | N | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| Liq_A | VISIT 1 | 508 | • | |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no PP | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 504 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | SERIOUS ADVERSE EXPERIENCE |
| | VISIT 3 | 501 | | |
| | | | no. P | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | VISIT 4 | 492 | | |
| Lyo | VISIT 1 | 257 | | |
| | | | no. PP | PROTOCOL VIOLATION |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 255 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 3 | 254 | | |
| | | | no.PPD | MIGRATION FROM STUDY AREA |
| | | | no. PP | LOST TO FOLLOW-UP |
| | | | no.PPD | LOST TO FOLLOW-UP |
| | | | no PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | LOST TO FOLLOW-UP |
| | | | no. PPD | ADVERSE EXPERIENCE |
| - | VISIT 4 | 247 | | |

Statistical Analysis Plan Amendment 1 Final

Template 5 Number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses with reasons for exclusion

| | | То | tal | | | _IQ_/ | A | | _IQ_I | 3 | | _IQ_( | 3 | - | _Y0 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Title | N | n | S | % | N | n | s | N | n | s | N | n | s | N | n | s |
| Total enrolled cohort | 1200 | | | | 298 | | | 302 | | | 300 | | | 300 | | |
| Exposed Set | 1200 | | | 100 | 298 | | | 302 | | | 300 | | | 300 | | |
| Administration of vaccine(s) | | 2 | 2 | | | 1 | 1 | | 1 | 1 | | 0 | 0 | | 0 | 0 |
| forbidden in the protocol (code 1040) | | | | | | | | | | | | | | | | |
| Study vaccine dose not | | 73 | 73 | | | 21 | 21 | | 13 | 13 | | 23 | 23 | | 16 | 16 |
| administered according to protocol (code 1070) | | | | | | | | | | | | | | | | |
| Initially seropositive or unknown | | 10 | 11 | | | 3 | 4 | | 3 | 3 | | 3 | 3 | | 1 | 1 |
| anti-rotavirus IgA antibody on<br>day of dose 1 (code 1500) | | | | | | | • | | | | | | | | • | |
| Protocol violation | | 1 | 1 | | | 0 | 0 | | 0 | 0 | | 1 | 1 | | 0 | 0 |
| (inclusion/exclusion criteria) | | • | • | | | | | | | | | ' | | | | |
| (code 2010) | | | | | | | | | | | | | | | | |
| Administration of any | | 1 | 1 | | | 0 | 0 | | 0 | 0 | | 0 | 0 | | 1 | 1 |
| medication forbidden by the | | - | - | | | | | | | | | | | | - | - |
| protocol (code 2040) | | | | | | | | | | | | | | | | |
| Underlying medical condition | | 1 | 1 | | | 1 | 1 | | 0 | 0 | | 0 | 0 | | 0 | 0 |
| forbidden by the protocol (code 2050) | | | | | | | | | | | | | | | | |
| Concomitant infection not | | 0 | 1 | | | 0 | 0 | | 0 | 0 | | 0 | 0 | | 0 | 1 |
| related to the vaccine which | | | | | | | | | | | | | | | | |
| may influence immune | | | | | | | | | | | | | | | | |
| response (code 2070) | | | | | | | | | | | | | | | | |
| Non-compliance with | | 14 | 16 | | | 5 | 5 | | 0 | 0 | | 6 | 7 | | 3 | 4 |
| vaccination schedule (including | | | | | | | | | | | | | | | | |
| wrong and unknown dates ) (code 2080) | | | | | | | | | | | | | | | | |
| Non-compliance with blood | | 12 | 16 | | | 2 | 3 | | 3 | 3 | | 3 | 5 | | 4 | 5 |
| sampling schedule (including | | | | | | | | | | | | | | | | |
| wrong and unknown dates) | | | | | | | | | | | | | | | | |
| (code 2090) | | | | | | | | | | | | | | | | |
| Essential serological data | | 87 | 95 | | | 23 | 25 | | 21 | 22 | | 20 | 22 | | 23 | 26 |
| missing (code 2100) | | | | | | | | | | | | | | | | |
| Subjects with incomplete study | | 1 | 1 | | | 0 | 0 | | 1 | 1 | | 0 | 0 | | 0 | 0 |
| vaccination schedule but with | | | | | | | | | | | | | | | | |
| post serological result (code 2500) | | | | | | | | | | | | | | | | |
| Per protocol set | 998 | | | 83.2 | 242 | | | 260 | | | 244 | | | 252 | | T |

LIQ\_A = HRV vaccine liquid formulation Lot A LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C LYO = HRV vaccine lyophilised formulation

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

<sup>% =</sup> percentage of subjects in the per protocol set (PPS) relative to the exposed set (ES)

115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

Template 6 Summary of demographic characteristics (Per Protocol Analysis Set of Immunogenicity)

| | | LIQ_A<br>N = 242 | | LIQ_B<br>N = 26 | | LIQ_C<br>N = 24 | | LYO<br>N = 25 | 52 | Total<br>N = 99 | 18 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Value | % | Value | | Value | | Value | | Value | - |
| Characteristics | Parameters or Categories | or n | /0 | or n | /0 | or n | /0 | or n | /0 | or n | /0 |
| Age at Dose 1 | Mean | 11.6 | _ | 11.5 | _ | 11.5 | _ | 11.6 | _ | 11.6 | _ |
| of HRV vaccine | SD | 1.32 | _ | 1.16 | _ | 1.19 | _ | 1.20 | _ | 1.22 | _ |
| (weeks) | Median | 11.0 | _ | 11.0 | _ | 11.0 | _ | 11.0 | _ | 11.0 | _ |
| () | Minimum | 10 | _ | 10 | _ | 10 | _ | 10 | _ | 10 | _ |
| | Maximum | 17 | _ | 15 | _ | 15 | _ | 16 | _ | 17 | _ |
| Age at Dose 2 | Mean | 16.6 | _ | 16.5 | _ | 16.5 | _ | 16.7 | _ | 16.6 | _ |
| of HRV vaccine | SD | 1.48 | _ | 1.40 | _ | 1.37 | _ | 1.34 | _ | 1.40 | _ |
| (weeks) | Median | 17.0 | _ | 16.0 | _ | 16.0 | _ | 17.0 | _ | 17.0 | _ |
| (Wooko) | Minimum | 14 | _ | 14 | _ | 14 | _ | 14 | _ | 14 | _ |
| | Maximum | 22 | _ | 20 | _ | 20 | _ | 21 | _ | 22 | _ |
| Gender | Female | 122 | 50.4 | 121 | 46.5 | 120 | 49.2 | 120 | 47.6 | 483 | 48.4 |
| | Male | 120 | 49.6 | 139 | 53.5 | 124 | 50.8 | 132 | 52.4 | 515 | 51.6 |
| Ethnicity | American Hispanic or Latino | 0 | 0.0 | 2 | 0.8 | 1 | 0.4 | 0 | 0.0 | 3 | 0.3 |
| Lumony | Not American Hispanic or Latino | 242 | 100.0 | | 99.2 | 243 | 99.6 | 252 | 100.0 | | 99.7 |
| Race | African heritage / African<br>American | 1 | 0.4 | 0 | 0.0 | 1 | 0.4 | 0 | 0.0 | 2 | 0.2 |
| | American Indian or Alaskan native | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - central/south Asian heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - east Asian heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - Japanese heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Asian - south east Asian heritage | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | Native Hawaiian or other pacific islander | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | White - Arabic / north African heritage | 0 | 0.0 | 0 | 0.0 | 2 | 8.0 | 0 | 0.0 | 2 | 0.2 |
| | White - Caucasian / European heritage | 239 | 98.8 | 258 | 99.2 | 240 | 98.4 | 247 | 98.0 | 984 | 98.6 |
| | Other | 2 | 8.0 | 2 | 8.0 | 1 | 0.4 | 5 | 2.0 | 10 | 1.0 |
| Height at Visit | Mean | 60.4 | - | 60.5 | - | 60.7 | - | 60.6 | - | 60.5 | - |
| 1 (cm) | SD | 2.35 | - | 2.37 | - | 2.32 | - | 2.22 | - | 2.32 | - |
| | Median | 61.0 | - | 60.0 | - | 61.0 | - | 61.0 | - | 61.0 | - |
| | Unknown | 0 | - | 1 | - | 2 | - | 0 | - | 3 | - |
| Weight at Visit | Mean | 6.0 | - | 6.1 | - | 6.2 | - | 6.1 | - | 6.1 | - |
| 1 (kg) | SD | 0.77 | - | 0.76 | - | 0.77 | - | 0.75 | - | 0.76 | - |
| | Median | 6.0 | - | 6.0 | <u> -</u> | 6.2 | - | 6.1 | - | 6.1 | <u> -</u> |
| BMI at Visit 1 | Mean | 16.5 | - | 16.6 | - | 16.7 | - | 16.7 | - | 16.6 | - |
| (kg/m²) | SD | 1.49 | - | 1.46 | - | 1.46 | - | 1.46 | - | 1.47 | - |
| | Median | 16.3 | - | 16.5 | - | 16.5 | - | 16.7 | - | 16.5 | - |
| | Unknown | 0 | - | 1 | _ | 2 | - | 0 | _ | 3 | - |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B LIQ\_C = HRV vaccine liquid formulation Lot C

Statistical Analysis Plan Amendment 1 Final

LYO = HRV vaccine lyophilised formulation
N = total number of subjects
n (%) = number / percentage of subjects in a given category
Value = value of the considered parameter
SD = standard deviation

Template 7 Deviations from specifications for age and intervals between study visits - Exposed Set

| | | Age | PRE-Dose:1 | Dose:1 | l-Dose:2 | Dose:2 | -PII(M2) |
|---|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Adapted | Protocol | Adapted |
| | | from 10 to 17 | from 0 to 0 days | from 30 to 48 | from 21 to 48 | from 30 to 48 | from 21 to 48 |
| | | weeks | | days | days | days | days |
| LIQ_A | N | 298 | 298 | 297 | 297 | 287 | 287 |
| | n | 0 | 2 | 8 | 7 | 1 | 1 |
| | % | 0.0 | 0.7 | 2.7 | 2.4 | 0.3 | 0.3 |
| | range | 10 to 17 | 0 to 4 | 29 to 76 | 29 to 76 | 30 to 55 | 30 to 55 |
| LIQ_B | N | 302 | 302 | 301 | 301 | 294 | 294 |
| | n | 0 | 1 | 0 | 0 | 4 | 2 |
| | % | 0.0 | 0.3 | 0.0 | 0.0 | 1.4 | 0.7 |
| | range | 10 to 15 | 0 to 3 | 30 to 48 | 30 to 48 | 24 to 56 | 24 to 56 |
| LIQ_C | N | 300 | 300 | 300 | 300 | 291 | 291 |
| | n | 1 | 1 | 8 | 7 | 4 | 4 |
| | % | 0.3 | 0.3 | 2.7 | 2.3 | 1.4 | 1.4 |
| | range | 9 to 17 | 0 to 9 | 27 to 76 | 27 to 76 | 30 to 56 | 30 to 56 |
| LY0 | N | 300 | 300 | 299 | 299 | 289 | 289 |
| | n | 0 | 2 | 4 | 4 | 5 | 3 |
| | % | 0.0 | 0.7 | 1.3 | 1.3 | 1.7 | 1.0 |
| | range | 10 to 16 | 0 to 3 | 30 to 61 | 30 to 61 | 28 to 61 | 28 to 61 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LYO = HRV vaccine lyophilised formulation

PRE = pre-vaccination

PII (M2) = blood sample taken one month after Dose 2 of the HRV vaccine (Visit 3)

Adapted = interval used for defining the ATP cohorts for immunogenicity

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

Statistical Analysis Plan Amendment 1 Final

Template 8 Summary of co-administered vaccination by dose - Exposed Set

| Dose1 | LIQ_A<br>N = 298 | } | LIQ_B<br>N = 302 | ! | LIQ_C<br>N = 300 | ) | LYO<br>N = 300 | 1 | Total<br>N = 12 | 00 |
|---|---|---|---|---|---|---|---|---|---|---|
| | Value | % | Value | % | Value | % | Value | % | Value | % |
| Characteristics | or n | | or n | | or n | | or n | | or n | |
| Any | 298 | 100 | 302 | 100 | 299 | 99.7 | 300 | 100 | 1199 | 99.9 |
| Infanrix hexa | 298 | 100 | 302 | 100 | 299 | 99.7 | 300 | 100 | 1199 | 99.9 |
| Dose 2 | LIQ_A<br>N = 297 | , | LIQ_B<br>N = 301 | | LIQ_C<br>N = 300 | ) | LYO<br>N = 299 | ١ | Total<br>N = 11 | 97 |
| | Value | % | Value | % | Value | % | Value | % | Value | % |
| Characteristics | or n | | or n | | or n | | or n | | or n | |
| Any | 297 | 100 | 301 | 100 | 298 | 99.3 | 299 | 100 | 1195 | 99.8 |
| Infanrix hexa | 297 | 100 | 301 | 100 | 298 | 99.3 | 299 | 100 | 1195 | 99.8 |

LIQ A = HRV vaccine liquid formulation Lot A

LIQ B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LYO = HRV vaccine lyophilised formulation

N = total number of subjects having received the considered dose of HRV

n/% = number/percentage of subjects who received the specified vaccination on the same day as the considered dose of HRV vaccine

Template 9 Summary of vaccinations other than HRV vaccine administered from birth until Visit 3, excluding vaccination given on the day of HRV doses - Exposed Set

| Before Dose 1 | | LIQ | Α | | LIQ_ | В | | LIQ_ | C | | LYC | ) | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N = 2 | 98 | | N = 30 | )2 | | N = 3 | 00 | | N = 3 | 00 | | N = 120 | 00 |
| | # | n | % | # | n | % | # | n | % | # | n | % | # | n | % |
| Characteristics | | | | | | | | | | | | | | | |
| Any | 18 | 18 | 6.0 | 11 | 11 | 3.6 | 13 | 13 | 4.3 | 25 | 25 | 8.3 | 67 | 67 | 5.6 |
| BCG | 18 | 18 | 6.0 | 11 | 11 | 3.6 | 12 | 12 | 4.0 | 25 | 25 | 8.3 | 66 | 66 | 5.5 |
| Infanrix hexa™ | 0 | 0 | 0.0 | 0 | 0 | 0.0 | 1 | 1 | 0.3 | 0 | 0 | 0.0 | 1 | 1 | 0.1 |
| Between Dose 1 and | | LIQ | Α | | LIQ_ | В | | LIQ | С | | LYC | ) | | Total | • |
| Dose 2§ | | N = 2 | 298 | | N = 30 | )2 | | N = 3 | 00 | | N = 3 | 00 | | N = 120 | 00 |
| - | # | n | % | # | n | % | # | n | % | # | n | % | # | n | % |
| Characteristics | | | | | | | | | | | | | | | |
| Any | 0 | 0 | 0.0 | 2 | 1 | 0.3 | 0 | 0 | 0.0 | 0 | 0 | 0.0 | 2 | 1 | 0.1 |
| Infanrix hexa™ | 0 | 0 | 0.0 | 2 | 1 | 0.3 | 0 | 0 | 0.0 | 0 | 0 | 0.0 | 2 | 1 | 0.1 |
| Between Dose 2 and | | LIQ | Α | | LIQ_ | В | | LIQ | С | | LYC | ) | | Total | |
| Visit 3* | | N = 2 | 97 | | N = 30 | )1 | | N = 3 | 00 | | N = 2 | 99 | | N = 119 | 97 |
| | # | n | % | # | n | % | # | n | % | # | n | % | # | n | % |
| Characteristics | | | | | | | | | | | | | | | |
| Any | 291 | 291 | 98.0 | 295 | 295 | 98.0 | 287 | 286 | 95.3 | 290 | 290 | 97.0 | 1163 | 1162 | 97.1 |
| DTPa+IPV+Hib | 0 | 0 | 0.0 | 1 | 1 | 0.3 | 0 | 0 | 0.0 | 0 | 0 | 0.0 | 1 | 1 | 0.1 |
| Infanrix hexa™ | 291 | 291 | 98.0 | 294 | 294 | 97.7 | 287 | 286 | 95.3 | 290 | 290 | 97.0 | 1162 | 1161 | 97.0 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LYO = HRV vaccine lyophilised formulation

N = Before Dose 1 and between Dose 1 and Dose 2: total number of subjects having received dose 1 of HRV Between Dose 2 and visit 3: total number of subjects having received dose 2 of HRV

#= number of doses administered of the specified vaccination excluding vaccination given on the day of HRV doses n/% = number/percentage of subjects who received at least one specified vaccination between the considered visits excluding vaccination given on the day of HRV doses

§= up to last contact of conclusion at Visit 3 if dose 2 of HRV was not administered

<sup>\*=</sup> up to last contact of conclusion at Visit 3 if visit 3 was not done

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

Template 10 Anti-rotavirus IgA antibody GMC and seroconversion rates – Per Protocol Analysis Set of Immunogenicity

| | | | | ≥ 20 | J/ml | | | GMC (U/ml) | |
|---|---|---|---|---|---|---|---|---|---|
| | | | 95% CI | | | 95% | 6 CI | | |
| Group | Timing | N | n | % | LL | UL | value | LL | UL |
| LIQ_A | PRE | 242 | 0 | 0.0 | 0.0 | 1.5 | <20 | - | - |
| | PII(M2) | 242 | 220 | 90.9 | 86.6 | 94.2 | 384.4 | 309.1 | 478.2 |
| LIQ_B | PRE | 260 | 0 | 0.0 | 0.0 | 1.4 | <20 | - | - |
| | PII(M2) | 260 | 235 | 90.4 | 86.1 | 93.7 | 418.8 | 337.8 | 519.1 |
| LIQ_C | PRE | 244 | 0 | 0.0 | 0.0 | 1.5 | <20 | - | - |
| | PII(M2) | 244 | 206 | 84.4 | 79.3 | 88.7 | 324.4 | 253.4 | 415.3 |
| LIQPOOL | PRE | 746 | 0 | 0.0 | 0.0 | 0.5 | <20 | - | - |
| | PII(M2) | 746 | 661 | 88.6 | 86.1 | 90.8 | 374.7 | 328.8 | 426.9 |
| LYO | PRE | 252 | 0 | 0.0 | 0.0 | 1.5 | <20 | - | - |
| | PII(M2) | 252 | 228 | 90.5 | 86.2 | 93.8 | 331.8 | 265.0 | 415.4 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects with available results

n (%) = number/percentage of subjects with concentration above the cut-off

95% CI = 95% Confidence Interval; L.L =Lower limit; U.L = upper limit

Pre = pre-vaccination

PII (M2) = blood sample taken one month after Dose 2 of HRV vaccine (Visit 3)

Template 11 Anti-rotavirus IgA antibody GMC calculated on subjects seropositive for anti-rotavirus IgA antibodies – Per Protocol Analysis Set of Immunogenicity

| | | | | GMC | |
|---------|---------|-----|-------|-------|-------|
| | | | | 95% | 6 CI |
| Group | Timing | N | value | LL | UL |
| LIQ_A | PII(M2) | 220 | 553.8 | 463.4 | 661.7 |
| LIQ_B | PII(M2) | 235 | 623.0 | 525.0 | 739.4 |
| LIQ_C | PII(M2) | 206 | 616.4 | 510.4 | 744.4 |
| LIQPOOL | PII(M2) | 661 | 597.1 | 538.7 | 661.8 |
| LYO | PII(M2) | 228 | 479.7 | 395.4 | 582.0 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects who were seropositive for anti-rotavirus IgA antibodies

95% CI = 95% Confidence Interval; LL = Lower Limit; UL = Upper Limit

PII(M2) = blood sample taken one month after Dose 2 of HRV vaccine (Visit 3)

Statistical Analysis Plan Amendment 1 Final

Template 12 Ratio of anti-rotavirus IgA antibody GMCs 1-2 months after Dose 2 of the HRV vaccine between each pair of the three lots of the HRV PCV-free liquid vaccine – Per Protocol Analysis Set of Immunogenicity

| | | | | | | | GMC rati | 0 | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 95% | 6 CI |
| Group | N | GMC | Group | N | GMC | Ratio order | Value | LL | UL |
| LIQ_A | 242 | 384.4 | LIQ_B | 260 | 418.8 | LIQ_A /LIQ_B | 0.92 | 0.67* | 1.26* |
| LIQ_A | 242 | 384.4 | LIQ_C | 244 | 324.4 | LIQ_A /LIQ_C | 1.19 | 0.86* | 1.64* |
| LIQ_B | 260 | 418.8 | LIQ_C | 244 | 324.4 | LIQ_B/LIQ_C | 1.29 | 0.94* | 1.77* |

LIQ\_A = HRV vaccine liquid formulation Lot A LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = number of subjects with available results

95% CI = 95% Confidence Interval (one-way ANOVA model with pooled variance from the four groups)

L.L. = Lower Limit, U.L. = Upper Limit

\*The two-sided 95% CIs are within [0.5, 2] (the pre-defined clinical limit interval for consistency)

Template 13 Difference between groups in the percentage of subjects who seroconverted for anti-rotavirus IgA antibody 1-2 months after Dose 2 of the HRV vaccine – Per Protocol Analysis Set of Immunogenicity

| | | | | | | Difference in | serocon | version r | ate |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | <b>95</b> % | 6 CI |
| Group | N | % | Group | N | % | Difference | % | LL | UL |
| LIQPOOL | 746 | 88.6 | LYO | 252 | 90.5 | LYO - LIQPOOL | 1.87 | -2.85 | 5.83* |

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects with available results

% = percentage of subjects who seroconverted at visit 3

95% CI = asymptotic standardised 95% Confidence Interval; LL = Lower Limit; UL = Upper Limit

\*Lower limit of the 95% CI ≥-10% (the pre-defined clinical limit for non-inferiority)

Template 14 Ratio of anti-rotavirus IgA antibody GMCs 1-2 months after Dose 2 of the HRV vaccine between the HRV lyophilised vaccine group and the pooled HRV PCV-free liquid vaccine – Per Protocol Analysis Set of Immunogenicity

| | | | | | | G | MC ratio | ) | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 95 | 5% CI |
| Group | N | GMC | Group | N | GMC | Ratio order | Value | LL | UL |
| LIQPOOL | 746 | 373.8† | LYO | 252 | 331.8 | LYO /LIQPOOL | 0.89 | 0.68 | 1.15* |

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects with available results

†geometric mean of the 3 GMC from the HRV liquid formulation groups

95% CI = 95% Confidence Interval (one-way ANOVA model using the group contrast between the HRV lyophilised formulation group and average of the HRV liquid formulation groups)

L.L. = Lower Limit, U.L. = Upper Limit

\*Lower limit of the 95% CI ≥ 0.67 (the pre-defined clinical limit for non-inferiority)

Statistical Analysis Plan Amendment 1 Final

Template 15 Reverse cumulative distribution curve for anti-rotavirus IgA antibody concentrations at Visit 3 - Per Protocol Analysis Set of Immunogenicity



Template 16 Number and percentage of subjects who received study vaccine doses - Exposed Set

| | LIQ_A<br>N = 298 | | N = 298 N = 302 | | LIQ_C<br>N = 300 | | LYO<br>N = 300 | | Total<br>N = 1200 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Total number of doses received | n | % | n | % | n | % | n | % | n | % |
| 1 | 1 | 0.3 | 1 | 0.3 | 0 | 0.0 | 1 | 0.3 | 3 | 0.3 |
| 2 | 297 | 99.7 | 301 | 99.7 | 300 | 100 | 299 | 99.7 | 1197 | 99.8 |
| Anv | 298 | 100 | 302 | 100 | 300 | 100 | 300 | 100 | 1200 | 100 |

LIQ\_A = HRV vaccine Liquid formulation lot A LIQ\_B = HRV vaccine Liquid formulation lot B

LIQ\_C = HRV vaccine Liquid formulation lot C LYO = HRV vaccine lyophilised formulation

N = number of subjects in each group or in total included in the considered cohort

n (%) = number/percentage of subjects receiving the specified total number of doses

Any = number and percentage of subjects receiving at least one dose

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

### Template 17 Compliance in returning symptom sheets - Exposed Set

| Dose | GROUP | Number | Doses | Number | Compliance |
|---|---|---|---|---|---|
| | | of doses | NOT according to protocol | of general SS | % general SS |
| 1 | LIQ_A | 298 | 10 | 298 | 100 |
| | LIQ_B | 302 | 7 | 302 | 100 |
| | LIQ_C | 300 | 6 | 300 | 100 |
| | LIQPOOL | 900 | 23 | 900 | 100 |
| | LYO | 300 | 6 | 299 | 99.7 |
| 2 | LIQ_A | 297 | 12 | 296 | 99.7 |
| | LIQ_B | 301 | 6 | 301 | 100 |
| | LIQ_C | 300 | 13 | 299 | 99.7 |
| | LIQPOOL | 898 | 31 | 896 | 99.8 |
| | LYO | 299 | 9 | 297 | 99.3 |
| Total | LIQ_A | 595 | 22 | 594 | 99.8 |
| | LIQ_B | 603 | 13 | 603 | 100 |
| | LIQ_C | 600 | 19 | 599 | 99.8 |
| | LIQPOOL | 1798 | 54 | 1796 | 99.9 |
| | LYO | 599 | 15 | 596 | 99.5 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

SS = Symptom sheets used for the collection of solicited AEs

Compliance % = (number of doses with symptom sheet return / number of administered doses) X 100

Doses not according to protocol = number of doses with regurgitation or vomiting

Statistical Analysis Plan Amendment 1 Final

Template 18 Percentage of doses and of subjects reporting symptoms (solicited or unsolicited) reported during the 8-day (Day 0 to Day 7) follow-up period - Exposed Set

| | | | Any | symptom | | |
|-----------------|---------|------|------|---------|------|------|
| | | | | | 959 | % CI |
| | Group | N | n | % | LL | UL |
| Dose 1 | LIQ_A | 298 | 251 | 84.2 | 79.6 | 88.2 |
| | LIQ_B | 302 | 267 | 88.4 | 84.3 | 91.8 |
| | LIQ_C | 300 | 247 | 82.3 | 77.5 | 86.5 |
| | LIQPOOL | 900 | 765 | 85.0 | 82.5 | 87.3 |
| | LYO | 300 | 249 | 83.0 | 78.3 | 87.1 |
| Dose 2 | LIQ_A | 297 | 247 | 83.2 | 78.4 | 87.2 |
| | LIQ_B | 301 | 260 | 86.4 | 82.0 | 90.0 |
| | LIQ_C | 300 | 236 | 78.7 | 73.6 | 83.2 |
| | LIQPOOL | 898 | 743 | 82.7 | 80.1 | 85.2 |
| | LYO | 299 | 247 | 82.6 | 77.8 | 86.7 |
| Overall/dose | LIQ_A | 595 | 498 | 83.7 | 80.5 | 86.6 |
| | LIQ_B | 603 | 527 | 87.4 | 84.5 | 89.9 |
| | LIQ_C | 600 | 483 | 80.5 | 77.1 | 83.6 |
| | LIQPOOL | 1798 | 1508 | 83.9 | 82.1 | 85.5 |
| | LYO | 599 | 496 | 82.8 | 79.5 | 85.7 |
| Overall/subject | LIQ_A | 298 | 283 | 95.0 | 91.8 | 97.2 |
| | LIQ_B | 302 | 287 | 95.0 | 91.9 | 97.2 |
| | LIQ_C | 300 | 275 | 91.7 | 87.9 | 94.5 |
| | LIQPOOL | 900 | 845 | 93.9 | 92.1 | 95.4 |
| | LYO | 300 | 279 | 93.0 | 89.5 | 95.6 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

For each dose:

N = number of subjects having received the considered dose

n/% = number/percentage of subjects reporting at least one symptom for the considered dose

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses followed by at least one symptom

For overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least one symptom

Statistical Analysis Plan Amendment 1 Final

Template 19 Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, after each dose of the HRV lyophilised and HRV PCV-free liquid vaccine for all groups. - Exposed Set

| | | | L | IQ_A | | | | | LIQ I | В | | | | LIQ | С | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 % | 6 CI | | | | 95 % | 6 CI | | | | | % CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| - / | 71. | | | | ļ. | Dos | se 1 | 1 | | | | ļ | | | | |
| Cough/runny | All | 298 | 72 | 24.2 | 19.4 | 29.4 | 302 | 90 | 29.8 | 24.7 | 35.3 | 300 | 71 | 23.7 | 19.0 | 28.9 |
| nose | Grade<br>3 | 298 | 1 | 0.3 | 0.0 | 1.9 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 62 | 20.8 | 16.3 | 25.9 | 302 | 76 | 25.2 | 20.4 | 30.5 | 300 | 49 | 16.3 | 12.3 | 21.0 |
| Diarrhoea | All | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 9 | 3.0 | 1.4 | 5.6 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| | Grade<br>3 | 298 | 3 | 1.0 | 0.2 | 2.9 | 302 | 2 | 0.7 | 0.1 | 2.4 | 300 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 9 | 3.0 | 1.4 | 5.6 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| Fever(°C) | All | 298 | 63 | 21.1 | 16.6 | 26.2 | 302 | 59 | 19.5 | 15.2 | 24.5 | 300 | 57 | 19.0 | 14.7 | 23.9 |
| | Grade<br>3 | 298 | 1 | 0.3 | 0.0 | 1.9 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 61 | 20.5 | 16.0 | 25.5 | 302 | 58 | 19.2 | 14.9 | 24.1 | 300 | 55 | 18.3 | 14.1 | 23.2 |
| Irritability | All | 298 | 213 | 71.5 | 66.0 | 76.5 | 302 | 225 | 74.5 | 69.2 | 79.3 | 300 | | 63.7 | 57.9 | 69.1 |
| | Grade<br>3 | 298 | 12 | 4.0 | 2.1 | 6.9 | 302 | 17 | 5.6 | 3.3 | 8.9 | 300 | 9 | 3.0 | 1.4 | 5.6 |
| | Related | 298 | 203 | 68.1 | 62.5 | 73.4 | 302 | 220 | 72.8 | 67.5 | 77.8 | | 184 | | 55.6 | 66.9 |
| Loss of appetite | All | 298 | 79 | 26.5 | 21.6 | 31.9 | 302 | 79 | 26.2 | 21.3 | 31.5 | 300 | 73 | 24.3 | 19.6 | 29.6 |
| | Grade<br>3 | 298 | 0 | 0.0 | 0.0 | 1.2 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 75 | 25.2 | 20.3 | 30.5 | 302 | 78 | 25.8 | 21.0 | 31.2 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| Vomiting | All | 298 | 47 | 15.8 | 11.8 | 20.4 | 302 | 45 | 14.9 | 11.1 | 19.4 | 300 | 44 | 14.7 | 10.9 | 19.2 |
| | Grade<br>3 | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | 7 | 2.3 | 0.9 | 4.7 | 300 | 7 | 2.3 | 0.9 | 4.7 |
| | Related | 298 | 45 | 15.1 | 11.2 | 19.7 | 302 | 43 | 14.2 | 10.5 | 18.7 | 300 | 39 | 13.0 | 9.4 | 17.3 |
| | | | | | | Dos | se 2 | | | | | | | | | |
| Cough/runny | All | 297 | 92 | 31.0 | 25.8 | 36.6 | 301 | 104 | 34.6 | 29.2 | 40.2 | 300 | 95 | 31.7 | 26.4 | 37.3 |
| nose | Grade<br>3 | 297 | 2 | 0.7 | 0.1 | 2.4 | 301 | 2 | 0.7 | 0.1 | 2.4 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Related | 297 | 79 | 26.6 | 21.7 | 32.0 | 301 | 84 | 27.9 | 22.9 | 33.3 | 300 | 79 | 26.3 | 21.4 | 31.7 |
| Diarrhoea | All | 297 | 3 | 1.0 | 0.2 | 2.9 | 301 | 7 | 2.3 | 0.9 | 4.7 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| | Grade<br>3 | 297 | 1 | 0.3 | 0.0 | 1.9 | 301 | 2 | 0.7 | 0.1 | 2.4 | 300 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 297 | 3 | 1.0 | 0.2 | 2.9 | 301 | 7 | 2.3 | 0.9 | 4.7 | 300 | | 4.0 | 2.1 | 6.9 |
| Fever(°C) | All | 297 | 80 | 26.9 | 22.0 | 32.4 | 301 | 79 | 26.2 | 21.4 | 31.6 | | | 31.3 | 26.1 | 36.9 |
| | Grade<br>3 | 297 | 2 | 0.7 | 0.1 | 2.4 | 301 | 1 | 0.3 | 0.0 | 1.8 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 297 | 79 | 26.6 | 21.7 | 32.0 | 301 | 76 | 25.2 | 20.4 | 30.6 | | | 30.3 | 25.2 | 35.9 |
| Irritability | All | 297 | 201 | 67.7 | 62.0 | 73.0 | 301 | 224 | 74.4 | 69.1 | 79.3 | | | | 61.7 | 72.6 |
| | Grade<br>3 | 297 | 11 | 3.7 | 1.9 | 6.5 | 301 | 18 | 6.0 | 3.6 | 9.3 | 300 | | 4.7 | 2.6 | 7.7 |
| | Related | 297 | 195 | 65.7 | 60.0 | 71.0 | 301 | 220 | | 67.7 | 78.0 | | | | 61.0 | 72.0 |
| Loss of appetite | All | 297 | 69 | 23.2 | 18.5 | 28.5 | 301 | 63 | 20.9 | 16.5 | 26.0 | | | 23.3 | 18.7 | 28.5 |
| | Grade<br>3 | 297 | 1 | 0.3 | 0.0 | 1.9 | 301 | 0 | 0.0 | 0.0 | 1.2 | 300 | 0 | 0.0 | 0.0 | 1.2 |

### 115461 (ROTA-081)

### Statistical Analysis Plan Amendment 1 Final

| | | | L | IQ_A | | | | | LIQ_E | 3 | | | | LIQ_ | С | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 % | 6 CI | | | | 95 % | 6 CI | | | | 95 9 | % CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | Related | 297 | 67 | 22.6 | 17.9 | 27.7 | 301 | 59 | 19.6 | 15.3 | 24.5 | 300 | 68 | 22.7 | 18.1 | 27.8 |
| Vomiting | All | 297 | 43 | 14.5 | 10.7 | 19.0 | 301 | 40 | 13.3 | 9.7 | 17.7 | 300 | 33 | 11.0 | 7.7 | 15.1 |
| | Grade<br>3 | 297 | 7 | 2.4 | 1.0 | 4.8 | 301 | 8 | 2.7 | 1.2 | 5.2 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| | Related | 297 | 40 | 13.5 | 9.8 | 17.9 | 301 | 40 | 13.3 | 9.7 | 17.7 | 300 | 32 | 10.7 | 7.4 | 14.7 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = number of subjects having received the considered dose

n/% = number/percentage of subjects reporting the specified symptom for the considered dose

All = any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination

Grade 3 = any occurrence of the specified symptom rated as grade 3

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

Statistical Analysis Plan Amendment 1 Final

Template 20 Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each dose in the pooled HRV PCV-free liquid vaccine group and the HRV vaccine lyophilised formulation group - Exposed Set

| | | | | LIQPO | OL | | | | LYO | ) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 9 | % CI | | | | 95 | % CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL |
| | | • | | Dose 1 | | | | | | | |
| Cough/runny nose | All | 900 | 233 | 25.9 | 23.1 | 28.9 | 300 | 79 | 26.3 | 21.4 | 31.7 |
| | Grade 3 | 900 | 2 | 0.2 | 0.0 | 8.0 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Related | 900 | 187 | 20.8 | 18.2 | 23.6 | 300 | 64 | 21.3 | 16.8 | 26.4 |
| Diarrhoea | All | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | Grade 3 | 900 | 7 | 8.0 | 0.3 | 1.6 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 3 | 1.0 | 0.2 | 2.9 |
| Fever(°C) | All | 900 | 179 | 19.9 | 17.3 | 22.6 | 300 | 68 | 22.7 | 18.1 | 27.8 |
| | Grade 3 | 900 | 2 | 0.2 | 0.0 | 8.0 | 300 | 0 | 0.0 | 0.0 | 1.2 |
| | Related | 900 | 174 | 19.3 | 16.8 | 22.1 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| Irritability | All | 900 | 629 | 69.9 | 66.8 | 72.9 | 300 | 207 | 69.0 | 63.4 | 74.2 |
| | Grade 3 | 900 | 38 | 4.2 | 3.0 | 5.7 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 900 | 607 | 67.4 | 64.3 | 70.5 | 300 | 201 | 67.0 | 61.4 | 72.3 |
| Loss of appetite | All | 900 | 231 | 25.7 | 22.8 | 28.7 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| | Grade 3 | 900 | 1 | 0.1 | 0.0 | 0.6 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 900 | 220 | 24.4 | 21.7 | 27.4 | 300 | 63 | 21.0 | 16.5 | 26.1 |
| Vomiting | All | 900 | 136 | 15.1 | 12.8 | 17.6 | 300 | 55 | 18.3 | 14.1 | 23.2 |
| | Grade 3 | 900 | 25 | 2.8 | 1.8 | 4.1 | 300 | 11 | 3.7 | 1.8 | 6.5 |
| | Related | 900 | 127 | 14.1 | 11.9 | 16.6 | 300 | 51 | 17.0 | 12.9 | 21.7 |
| | | | | Dose 2 | | | | | | | |
| Cough/runny nose | All | 898 | 291 | 32.4 | 29.4 | 35.6 | 299 | 109 | 36.5 | 31.0 | 42.2 |
| | Grade 3 | 898 | 8 | 0.9 | 0.4 | 1.7 | 299 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 898 | 242 | 26.9 | 24.1 | 30.0 | 299 | 89 | 29.8 | 24.6 | 35.3 |
| Diarrhoea | All | 898 | 22 | 2.4 | 1.5 | 3.7 | 299 | 8 | 2.7 | 1.2 | 5.2 |
| | Grade 3 | 898 | 5 | 0.6 | 0.2 | 1.3 | 299 | 3 | 1.0 | 0.2 | 2.9 |
| | Related | 898 | 22 | 2.4 | 1.5 | 3.7 | 299 | 8 | 2.7 | 1.2 | 5.2 |
| Fever(°C) | All | 898 | 253 | 28.2 | 25.3 | 31.2 | 299 | 74 | 24.7 | 20.0 | 30.0 |
| | Grade 3 | 898 | 4 | 0.4 | 0.1 | 1.1 | 299 | 3 | 1.0 | 0.2 | 2.9 |
| | Related | 898 | 246 | 27.4 | 24.5 | 30.4 | 299 | 71 | 23.7 | 19.0 | 29.0 |
| Irritability | All | 898 | 627 | 69.8 | 66.7 | 72.8 | 299 | 200 | 66.9 | 61.2 | 72.2 |
| | Grade 3 | 898 | 43 | 4.8 | 3.5 | 6.4 | 299 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 898 | 615 | 68.5 | 65.3 | 71.5 | 299 | 196 | 65.6 | 59.9 | 70.9 |
| Loss of appetite | All | 898 | 202 | 22.5 | 19.8 | 25.4 | 299 | 62 | 20.7 | 16.3 | 25.8 |
| | Grade 3 | 898 | 1 | 0.1 | 0.0 | 0.6 | 299 | 0 | 0.0 | 0.0 | 1.2 |
| | Related | 898 | 194 | 21.6 | 19.0 | 24.4 | 299 | 60 | 20.1 | 15.7 | 25.1 |
| Vomiting | All | 898 | 116 | 12.9 | 10.8 | 15.3 | 299 | 41 | 13.7 | 10.0 | 18.1 |
| | Grade 3 | 898 | 23 | 2.6 | 1.6 | 3.8 | 299 | 11 | 3.7 | 1.9 | 6.5 |
| | Related | 898 | 112 | 12.5 | 10.4 | 14.8 | 299 | 40 | 13.4 | 9.7 | 17.8 |

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

N = number of subjects having received the considered dose

n/% = number/percentage of subjects reporting the specified symptom for the considered dose

All = any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination Grade 3 = any occurrence of the specified symptom rated as grade 3

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

Statistical Analysis Plan Amendment 1 Final

Template 21 Percentage of doses and subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, after each dose of the HRV lyophilised and HRV PCV-free HRV liquid vaccine for all groups. - Exposed Set

| | | LIQ_ | A | | | | LIQ | В | | | | LIQ | С | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 % | CI | | | | 95 % | CI | | - | | 95 % | CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| - | | | | | ( | Overal | l/dos | е | | | | | | | | |
| Cough/runny nose | All | 595 | 164 | 27.6 | 24.0 | 31.3 | 603 | 194 | 32.2 | 28.5 | 36.1 | 600 | 166 | 27.7 | 24.1 | 31.4 |
| 11036 | Grade 3 | 595 | 3 | 0.5 | 0.1 | 1.5 | 603 | | 0.3 | 0.0 | 1.2 | 600 | 5 | 0.8 | 0.3 | 1.9 |
| | Related | 595 | 141 | 23.7 | 20.3 | 27.3 | | | 26.5 | 23.0 | 30.3 | 600 | 128 | 21.3 | 18.1 | 24.8 |
| Diarrhoea | All | 595 | 11 | 1.8 | 0.9 | 3.3 | 603 | | 2.7 | 1.5 | 4.3 | 600 | 20 | 3.3 | 2.0 | 5.1 |
| | Grade 3 | 595 | 4 | 0.7 | 0.2 | 1.7 | 603 | | 0.7 | 0.2 | 1.7 | 600 | 4 | 0.7 | 0.2 | 1.7 |
| | Related | 595 | 11 | 1.8 | 0.9 | 3.3 | 603 | 16 | 2.7 | 1.5 | 4.3 | 600 | 20 | 3.3 | 2.0 | 5.1 |
| Fever(°C) | All | 595 | 143 | 24.0 | 20.7 | 27.7 | 603 | 138 | 22.9 | 19.6 | 26.4 | 600 | 151 | 25.2 | 21.7 | 28.8 |
| | Grade 3 | 595 | 3 | 0.5 | 0.1 | 1.5 | 603 | 1 | 0.2 | 0.0 | 0.9 | 600 | 2 | 0.3 | 0.0 | 1.2 |
| | Related | 595 | 140 | 23.5 | 20.2 | 27.1 | 603 | 134 | 22.2 | 19.0 | 25.8 | 600 | 146 | 24.3 | 21.0 | 28.0 |
| Irritability | All | 595 | 414 | 69.6 | 65.7 | 73.3 | 603 | 449 | 74.5 | 70.8 | 77.9 | 600 | 393 | 65.5 | 61.5 | 69.3 |
| | Grade 3 | 595 | 23 | 3.9 | 2.5 | 5.7 | 603 | 35 | 5.8 | 4.1 | 8.0 | 600 | 23 | 3.8 | 2.4 | 5.7 |
| | Related | 595 | 398 | 66.9 | 62.9 | 70.7 | 603 | 440 | 73.0 | 69.2 | 76.5 | 600 | 384 | 64.0 | 60.0 | 67.8 |
| Loss of appetite | All | 595 | 148 | 24.9 | 21.4 | 28.6 | 603 | 142 | 23.5 | 20.2 | 27.1 | 600 | 143 | 23.8 | 20.5 | 27.4 |
| | Grade 3 | 595 | 1 | 0.2 | 0.0 | 0.9 | 603 | 0 | 0.0 | 0.0 | 0.6 | 600 | 1 | 0.2 | 0.0 | 0.9 |
| | Related | 595 | 142 | 23.9 | 20.5 | 27.5 | 603 | 137 | 22.7 | 19.4 | 26.3 | 600 | 135 | 22.5 | 19.2 | 26.1 |
| Vomiting | All | 595 | 90 | 15.1 | 12.3 | 18.3 | 603 | 85 | 14.1 | 11.4 | 17.1 | 600 | 77 | 12.8 | 10.3 | 15.8 |
| | Grade 3 | 595 | 18 | 3.0 | 1.8 | 4.7 | 603 | 15 | 2.5 | 1.4 | 4.1 | 600 | 15 | 2.5 | 1.4 | 4.1 |
| | Related | 595 | 85 | 14.3 | 11.6 | 17.4 | 603 | 83 | 13.8 | 11.1 | 16.8 | 600 | 71 | 11.8 | 9.4 | 14.7 |
| | | | ļ. | | 0 | verall/ | subje | ect | | | | , | | | , | |
| Cough/runny nose | All | 298 | 134 | 45.0 | 39.2 | 50.8 | 302 | 147 | 48.7 | 42.9 | 54.5 | 300 | 132 | 44.0 | 38.3 | 49.8 |
| | Grade 3 | 298 | 3 | 1.0 | 0.2 | 2.9 | 302 | 2 | 0.7 | 0.1 | 2.4 | 300 | 5 | 1.7 | 0.5 | 3.8 |
| | Related | 298 | | 39.6 | 34.0 | 45.4 | | | | 35.8 | 47.2 | 300 | | 36.0 | 30.6 | 41.7 |
| Diarrhoea | All | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | | 5.0 | 2.8 | 8.1 | 300 | 19 | 6.3 | 3.9 | 9.7 |
| | Grade 3 | 298 | 4 | 1.3 | 0.4 | 3.4 | 302 | | 1.3 | 0.4 | 3.4 | 300 | 3 | 1.0 | 0.2 | 2.9 |
| | Related | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | | 5.0 | 2.8 | 8.1 | 300 | 19 | 6.3 | 3.9 | 9.7 |
| Fever(°C) | All | 298 | | 37.2 | 31.7 | 43.0 | | | 34.4 | 29.1 | 40.1 | 300 | | | 35.1 | 46.5 |
| , | Grade 3 | 298 | 3 | 1.0 | 0.2 | 2.9 | 302 | | 0.3 | 0.0 | 1.8 | 300 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 298 | | 36.6 | 31.1 | 42.3 | | | 33.1 | 27.8 | 38.7 | 300 | | 39.3 | 33.8 | 45.1 |
| Irritability | All | 298 | | 85.2 | 80.7 | 89.1 | | | | 84.3 | 91.8 | 300 | | 80.0 | 75.0 | 84.4 |
| | Grade 3 | 298 | 20 | 6.7 | 4.1 | 10.2 | 302 | | 10.3 | 7.1 | 14.3 | 300 | 21 | 7.0 | 4.4 | 10.5 |
| | Related | 298 | | 84.6 | 80.0 | 88.5 | | | 87.7 | 83.5 | 91.2 | 300 | | 79.3 | 74.3 | 83.8 |
| Loss of appetite | All | 298 | | 37.2 | 31.7 | 43.0 | | | 37.4 | 31.9 | 43.1 | 300 | | 37.0 | 31.5 | 42.7 |
| | Grade 3 | 298 | 1 | 0.3 | 0.0 | 1.9 | 302 | | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | | 35.6 | 30.1 | 41.3 | | | 35.8 | 30.4 | 41.5 | 300 | | 36.3 | 30.9 | 42.1 |
| Vomiting | All | 298 | 70 | 23.5 | 18.8 | 28.7 | 302 | | 19.5 | 15.2 | 24.5 | 300 | 61 | 20.3 | 15.9 | 25.3 |
| · omining | Grade 3 | 298 | 18 | 6.0 | 3.6 | 9.4 | 302 | | 4.0 | 2.1 | 6.8 | 300 | 12 | 4.0 | 2.1 | 6.9 |
| | Related | 298 | 69 | 23.2 | 18.5 | 28.4 | 302 | | 19.2 | 14.9 | 24.1 | 300 | 58 | 19.3 | 15.0 | 24.3 |
| I IO A = HRV vac | | | | | 10.0 | 20.7 | 002 | 50 | 10.2 | 17.5 | <u>∠</u> -7.1 | 000 | 00 | 10.0 | 10.0 | |

LIQ\_A = HRV vaccine liquid formulation Lot A

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses followed by the specified symptom

For overall/subject:

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once the specified symptom

All = any occurrence of the specified symptom, irrespective of intensity grade and relationship to vaccination

Grade 3 = any occurrence of the specified symptom rated as grade 3

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

Template 22 Percentage of subjects with unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after any vaccination in each HRV PCV-free vaccine liquid group - Exposed Set

| | | | LIC<br>N = | Q_A<br>298 | | | | Q_B<br>: 302 | | | | Q_C<br>300 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 6 CI | | | | % CI | | | | % CI |
| Primary System Organ | Preferred | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| Class (CODE) | Term (CODE) | | | | | | | | | | | | |
| At least one symptom | , | 24 | 8.1 | 5.2 | 11.7 | 26 | 8.6 | 5.7 | 12.4 | 33 | 11.0 | 7.7 | 15.1 |
| Ear and labyrinth | Ear pain | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| disorders (10013993) | (10014020) | | | | | | | | | | | | |
| Eye disorders (10015919) | Conjunctivitis (10010741) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| Gastrointestinal disorders (10017947) | Diarrhoea<br>(10012735) | 0 | 0.0 | 0.0 | 1.2 | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 |
| , , | Flatulence<br>(10016766) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| General disorders and administration site conditions (10018065) | Injection site erythema (10022061) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| , , | Injection site pain (10022086) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Injection site swelling (10053425) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Irritability<br>(10022998) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 1 | 0.3 | 0.0 | 1.8 |
| | Pyrexia (10037660) | 4 | 1.3 | 0.4 | 3.4 | 3 | 1.0 | 0.2 | 2.9 | 4 | 1.3 | 0.4 | 3.4 |
| Immune system disorders (10021428) | Hypersensitivit y (10020751) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| Infections and infestations (10021881) | Bronchitis<br>(10006451) | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Ear infection (10014011) | 1 | 0.3 | 0.0 | 1.9 | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 |
| | Exanthema subitum (10015586) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Eye infection (10015929) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Gastroenteritis (10017888) | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | Impetigo<br>(10021531) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Influenza<br>(10022000) | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | Laryngitis<br>(10023874) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | Otitis media<br>(10033078) | 5 | 1.7 | 0.5 | 3.9 | 6 | 2.0 | 0.7 | 4.3 | 11 | 3.7 | 1.8 | 6.5 |
| | Perianal<br>abscess<br>(10034447) | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |

### 115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

| | | | LIC | ١ ٨ | Otati | | | • | , i iai | / (111 | | | ГПІС |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | )_A<br>298 | | | | Q_B<br>302 | | | | Q_C<br>300 | |
| | | | N = | 298<br>95% | 4 CI | | IN - | | % CI | | IN - | | % CI |
| Primary System Organ | Preferred | n | % | LL | UL | n | % | LL | % CI<br>UL | n | % | LL | % CI<br>UL |
| Class (CODE) | Term (CODE) | " | /0 | LL | UL | " | /0 | LL | UL | " | /0 | LL | UL |
| Class (CODE) | Pneumonia | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| | (10035664) | U | 0.0 | 0.0 | 1.2 | ' | 0.5 | 0.0 | 1.0 | U | 0.0 | 0.0 | 1.2 |
| | Respiratory | 3 | 1.0 | 0.2 | 2.9 | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 |
| | tract infection | Ü | 1.0 | 0.2 | 2.0 | _ | 0.7 | 0.1 | ∠.⊤ | | 0.0 | 0.0 | 1.2 |
| | (10062352) | | | | | | | | | | | | |
| | Respiratory | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | tract infection | | | | | | | | | | | | |
| | viral | | | | | | | | | | | | |
| | (10062106) | | | | | | | | | | | | |
| | Rhinitis | 2 | 0.7 | 0.1 | 2.4 | 1 | 0.3 | 0.0 | 1.8 | 3 | 1.0 | 0.2 | 2.9 |
| | (10039083) | | | | | | | | | | | | |
| | Upper | 2 | 0.7 | 0.1 | 2.4 | 5 | 1.7 | 0.5 | 3.8 | 7 | 2.3 | 0.9 | 4.7 |
| | respiratory tract | | | | | | | | | | | | |
| | infection | | | | | | | | | | | | |
| | (10046306) | | | | | | | | | | | | |
| | Varicella | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 | 2 | 0.7 | 0.1 | 2.4 |
| B. I. C. P. I. | (10046980) | | 0.0 | 0.0 | 4.0 | _ | 0.0 | 0.0 | 4.0 | 4 | 0.0 | 0.0 | 4.0 |
| Psychiatric disorders | Crying | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| (10037175) | (10011469) | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 6 | 2.0 | 0.7 | 4.3 |
| Respiratory, thoracic and mediastinal disorders | Cough<br>(10011224) | ı | 0.3 | 0.0 | 1.9 | | 0.3 | 0.0 | 1.0 | О | 2.0 | 0.7 | 4.3 |
| (10038738) | (10011224) | | | | | | | | | | | | |
| (10030730) | Nasal | 1 | 0.3 | 0.0 | 1.9 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | congestion | ' | 0.5 | 0.0 | 1.5 | U | 0.0 | 0.0 | 1.2 | U | 0.0 | 0.0 | 1.2 |
| | (10028735) | | | | | | | | | | | | |
| | Rales | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | (10037833) | - | 3.0 | | | | | | | | 3.0 | | |
| Skin and subcutaneous | Dermatitis | 1 | 0.3 | 0.0 | 1.9 | 1 | 0.3 | 0.0 | 1.8 | 0 | 0.0 | 0.0 | 1.2 |
| tissue disorders | allergic | | | | | | | | | | | | |
| (10040785) | (10012434) | | | | | | | | | | | | |
| | Èczema | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 | 1 | 0.3 | 0.0 | 1.8 |
| | (10014184) | | | | | | | | | | | | |
| | Rash | 2 | 0.7 | 0.1 | 2.4 | 0 | 0.0 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 1.2 |
| | (10037844) | | | | | | | | | | | | |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting at least once a specified unsolicited symptom

At least one symptom = number of subjects reporting at least one unsolicited symptom, whatever the MedDRA PT

<sup>95%</sup> CI = exact 95% Confidence Interval, LL = Lower Limit, UL = Upper Limit

115461 (ROTA-081) Statistical Analysis Plan Amendment 1 Final

Template 23 Percentage of doses with unsolicited symptoms classified by MedDRA SOC and PT from Day 0 to Day 30 after vaccination in each HRV PCV-free liquid vaccine group - Exposed Set

| | | | | A<br>595 | | | | Q_B<br>= 603 | | | | Q_C<br>600 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | - 11 | 95% | 6 CI | | - ' ' | | % CI | | - ' ' | | % CI |
| Primary System Organ<br>Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | | 25 | 4.2 | 2.7 | 6.1 | 30 | 5.0 | 3.4 | 7.0 | 38 | 6.3 | 4.5 | 8.6 |
| Ear and labyrinth disorders (10013993) | Ear pain (10014020) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| Eye disorders (10015919) | Conjunctivitis (10010741) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | 0 | 0.0 | 0.0 | 0.6 | 2 | 0.3 | 0.0 | 1.2 | 1 | 0.2 | 0.0 | 0.9 |
| | Flatulence (10016766) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 2 | 0.3 | 0.0 | 1.2 |
| General disorders and administration site conditions (10018065) | Injection site erythema (10022061) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Injection site pain (10022086) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Injection site swelling (10053425) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Irritability (10022998) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 |
| | Pyrexia (10037660) | 4 | 0.7 | 0.2 | 1.7 | 3 | 0.5 | 0.1 | 1.4 | 4 | 0.7 | 0.2 | 1.7 |
| Immune system disorders (10021428) | Hypersensitivity (10020751) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| Infections and infestations (10021881) | Bronchitis (10006451) | 2 | 0.3 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Ear infection (10014011) | 1 | 0.2 | 0.0 | 0.9 | 3 | 0.5 | 0.1 | 1.4 | 2 | 0.3 | 0.0 | 1.2 |
| | Exanthema subitum (10015586) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Eye infection (10015929) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Gastroenteritis (10017888) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Impetigo (10021531) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Influenza (10022000) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Laryngitis (10023874) Otitis media (10033078) | 1<br>6 | 1.0 | 0.0 | 0.9 | 0 | 1.2 | 0.0 | 0.6<br>2.4 | 0<br>12 | 2.0 | 1.0 | 0.6<br>3.5 |
| | Perianal abscess (10034447) | 1 | 0.2 | 0.4 | 0.9 | 7 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Pneumonia (10035664) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| | Respiratory tract infection (10062352) | 3 | 0.5 | 0.1 | 1.5 | 2 | 0.3 | 0.0 | 1.2 | 0 | 0.0 | 0.0 | 0.6 |
| | Respiratory tract infection viral (10062106) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| | Rhinitis (10039083) | 2 | 0.3 | 0.0 | 1.2 | 1 | | 0.0 | 0.9 | 3 | 0.5 | 0.1 | 1.5 |
| | Upper respiratory tract infection (10046306) | 2 | 0.3 | 0.0 | 1.2 | 6 | | 0.4 | 2.2 | 8 | 1.3 | 0.6 | 2.6 |
| | Varicella (10046980) | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 | 2 | 0.3 | 0.0 | 1.2 |

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

| | | | LIC | ) A | | | 110 | QВ | | | 110 | ) C | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 595 | | | | <br>= 603 | | | | 600 | |
| | | | | 95% | 6 CI | | | 959 | % CI | | | 959 | % CI |
| Primary System Organ<br>Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL | n | % | LL | UL |
| Psychiatric disorders (10037175) | Crying (10011469) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| Respiratory, thoracic and mediastinal disorders | Cough (10011224) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 6 | 1.0 | 0.4 | 2.2 |
| (10038738) | Nasal congestion (10028735) | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 |
| | Rales (10037833) | 0 | 0.0 | 0.0 | 0.6 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |
| Skin and subcutaneous tissue disorders | Dermatitis allergic (10012434) | 1 | 0.2 | 0.0 | 0.9 | 1 | 0.2 | 0.0 | 0.9 | 0 | 0.0 | 0.0 | 0.6 |
| (10040785) | Eczema (10014184)<br>Rash (10037844) | 0 2 | 0.0 | 0.0 | 0.6<br>1.2 | 0 | 0.0 | 0.0 | 0.6 | 1 | 0.2 | 0.0 | 0.9 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = Total number of doses administered

n/% = number/percentage of doses followed by at least one report of the specified unsolicited symptom
At least one symptom = number of doses followed by at least one report of an unsolicited symptom whatever the
MedDRA PT

95% CI = Exact 95% Confidence Interval; LL = Lower Limit, UL = Upper Limit

Template 24 Percentage of subjects reporting any GE episodes from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set

| Group | Ве | twee | _ | se 1 and<br>ose 2 | before | Betv | veen | Dose | 2 and | Visit 3 | В | etwe | en Dos | e 1 and \ | isit 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | Cl | | | | 95% | 6 CI | | | | 95% | 6 CI |
| | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| LIQ_A | 298 | 16 | 5.4 | 3.1 | 8.6 | 297 | 10 | 3.4 | 1.6 | 6.1 | 298 | 25 | 8.4 | 5.5 | 12.1 |
| LIQ_B | 302 | 17 | 5.6 | 3.3 | 8.9 | 301 | 15 | 5.0 | 2.8 | 8.1 | 302 | 29 | 9.6 | 6.5 | 13.5 |
| LIQ_C | 300 | 17 | 5.7 | 3.3 | 8.9 | 300 | 18 | 6.0 | 3.6 | 9.3 | 300 | 33 | 11.0 | 7.7 | 15.1 |
| LIQPOOL | 900 | 50 | 5.6 | 4.2 | 7.3 | 898 | 43 | 4.8 | 3.5 | 6.4 | 900 | 87 | 9.7 | 7.8 | 11.8 |
| LYO | 300 | 8 | 2.7 | 1.2 | 5.2 | 299 | 15 | 5.0 | 2.8 | 8.1 | 300 | 22 | 7.3 | 4.7 | 10.9 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

Between Dose 1 and before Dose 2: N = number of subjects having received the first dose

Between Dose 2 and Visit 3: N = number of subjects having received the second dose

Between Dose 1 and Visit 3: N = number of subjects having received at least one dose

n/% = number/percentage of subjects reporting at least one gastroenteritis episode during the specified period

Statistical Analysis Plan Amendment 1 Final

# Template 25 Percentage of subjects reporting RV (vaccine strain or wild type RV) GE episodes from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set

| Group | Ве | twe | | se 1 and<br>ose 2 | before | В | etwe | en Do | ose 2 and | Visit 3 | Be | twee | n Do | se 1 and | Visit 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | | 95% | 6 CI | | | | 95% | CI |
| | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| LIQ_A | 298 | 0 | 0.0 | 0.0 | 1.2 | 297 | 0 | 0.0 | 0.0 | 1.2 | 298 | 0 | 0.0 | 0.0 | 1.2 |
| LIQ_B | 302 | 1 | 0.3 | 0.0 | 1.8 | 301 | 0 | 0.0 | 0.0 | 1.2 | 302 | 1 | 0.3 | 0.0 | 1.8 |
| LIQ_C | 300 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| LIQPOOL | 900 | 1 | 0.1 | 0.0 | 0.6 | 898 | 1 | 0.1 | 0.0 | 0.6 | 900 | 2 | 0.2 | 0.0 | 0.8 |
| LYO | 300 | 0 | 0.0 | 0.0 | 1.2 | 299 | 0 | 0.0 | 0.0 | 1.2 | 300 | 0 | 0.0 | 0.0 | 1.2 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

LIQPOOL = Pooled HRV vaccine liquid formulation

LYO = HRV vaccine lyophilised formulation

Between Dose 1 and before Dose 2: N = number of subjects having received the first dose

Between Dose 2 and Visit 3: N = number of subjects having received the second dose

Between Dose 1 and Visit 3: N = number of subjects having received at least one dose

n/% = number/percentage of subjects reporting at least one RV GE episode during the specified period

Template 26 Summary of RV GE episodes reported from Dose 1 of HRV vaccine up to Visit 3 - Exposed Set

| Subject no | Onset of episode | Isolated RV type |
|------------|------------------|----------------------|
| PP | Day 3 of Dose 1 | G1/P8 vaccine strain |
| PΡ | Day 23 of Dose 2 | G1/P8 vaccine strain |

Statistical Analysis Plan Amendment 1 Final

Template 27 Number and percentage of doses and of subjects who took at least one concomitant medication from Day 0 to Day 7 after vaccination by type in each HRV PCV-free vaccine liquid group - Exposed Set

| | | | LIQ_A | 4 | | | | LIQ_ | В | | LIQ_C | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | | 95% | 6 CI | | | | 959 | % CI |
| | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | | | | Do | se 1 | | | | | | | | |
| Any | 298 | 173 | 58.1 | 52.2 | 63.7 | 302 | 175 | 57.9 | 52.2 | 63.6 | 300 | 157 | 52.3 | 46.5 | 58.1 |
| Any antipyretic | 298 | 97 | 32.6 | 27.3 | 38.2 | 302 | 94 | 31.1 | 25.9 | 36.7 | 300 | 71 | 23.7 | 19.0 | 28.9 |
| Prophylactic antipyretic | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 6 | 2.0 | 0.7 | 4.3 | 300 | 9 | 3.0 | 1.4 | 5.6 |
| Any antibiotic | 298 | 6 | 2.0 | 0.7 | 4.3 | 302 | 5 | 1.7 | 0.5 | 3.8 | 300 | 5 | 1.7 | 0.5 | 3.8 |
| | | | | | | | se 2 | | | | | | | | |
| Any | 297 | 105 | 35.4 | 29.9 | 41.1 | 301 | 117 | 38.9 | 33.3 | 44.6 | 300 | 89 | 29.7 | 24.6 | 35.2 |
| Any antipyretic | 297 | 98 | 33.0 | 27.7 | 38.7 | 301 | 109 | 36.2 | 30.8 | 41.9 | 300 | 86 | 28.7 | 23.6 | 34.1 |
| Prophylactic antipyretic | 297 | 7 | 2.4 | 1.0 | 4.8 | 301 | 8 | 2.7 | 1.2 | 5.2 | 300 | 6 | 2.0 | 0.7 | 4.3 |
| Any antibiotic | 297 | 4 | 1.3 | 0.4 | 3.4 | 301 | 8 | 2.7 | 1.2 | 5.2 | 300 | 4 | 1.3 | 0.4 | 3.4 |
| | ļ. | | | | ( | Overa | II/do | se | | ļ. | | | | ļ. | |
| Any | 595 | 278 | 46.7 | 42.7 | 50.8 | 603 | 292 | 48.4 | 44.4 | 52.5 | 600 | 246 | 41.0 | 37.0 | 45.1 |
| Any antipyretic | 595 | 195 | 32.8 | 29.0 | 36.7 | 603 | 203 | 33.7 | 29.9 | 37.6 | 600 | 157 | 26.2 | 22.7 | 29.9 |
| Prophylactic antipyretic | 595 | 15 | 2.5 | 1.4 | 4.1 | 603 | 14 | 2.3 | 1.3 | 3.9 | 600 | 15 | 2.5 | 1.4 | 4.1 |
| Any antibiotic | 595 | 10 | 1.7 | 8.0 | 3.1 | 603 | 13 | 2.2 | 1.2 | 3.7 | 600 | 9 | 1.5 | 0.7 | 2.8 |
| | | | | | | veral | | ject | | | | | | | |
| Any | 298 | 194 | 65.1 | 59.4 | 70.5 | 302 | 205 | 67.9 | 62.3 | 73.1 | 300 | 182 | 60.7 | 54.9 | 66.2 |
| Any antipyretic | 298 | 130 | 43.6 | 37.9 | 49.5 | 302 | 141 | 46.7 | 41.0 | 52.5 | 300 | 111 | 37.0 | 31.5 | 42.7 |
| Prophylactic antipyretic | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | 12 | 4.0 | 2.1 | 6.8 | 300 | 13 | 4.3 | 2.3 | 7.3 |
| Any antibiotic | 298 | 10 | 3.4 | 1.6 | 6.1 | 302 | 13 | 4.3 | 2.3 | 7.2 | 300 | 9 | 3.0 | 1.4 | 5.6 |

LIQ\_A = HRV vaccine liquid formulation Lot A

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ C = HRV vaccine liquid formulation Lot C

For each dose and overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects who started to take the specified concomitant medication at least once during the mentioned period

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses after which the specified concomitant medication was started at least once during the mentioned period

Statistical Analysis Plan Amendment 1 Final

Template 28 Percentage of subjects reporting each solicited general symptom including those rated grade 3 in intensity and those assessed as related to vaccination during the 8-day (Day 0 to Day 7) follow-up period, for each documented dose in each HRV PCV-free liquid group - Exposed Set

| | | | | LIQ | | | | | LIQ | В | | | | LIQ | _C | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95 ( | % CI | | | | 95 | % CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| | | | | | | | se 1 | | | | | | | | | |
| Cough/runny nose | All | 298 | | 24.2 | 19.4 | 29.4 | 302 | | 29.8 | 24.7 | 35.3 | 300 | | 23.7 | 19.0 | 28.9 |
| | Grade 3 | | | 0.3 | 0.0 | 1.9 | 302 | | 0.0 | 0.0 | 1.2 | 300 | | 0.3 | 0.0 | 1.8 |
| | Related | | | 20.8 | 16.3 | 25.9 | 302 | | 25.2 | 20.4 | 30.5 | 300 | | 16.3 | 12.3 | 21.0 |
| Diarrhoea | All | 298 | | 2.7 | 1.2 | 5.2 | 302 | | 3.0 | 1.4 | 5.6 | 300 | | 2.7 | 1.2 | 5.2 |
| | Grade 3 | | | 1.0 | 0.2 | 2.9 | 302 | | 0.7 | 0.1 | 2.4 | 300 | | 0.7 | 0.1 | 2.4 |
| | Related | 298 | 8 | 2.7 | 1.2 | 5.2 | 302 | 9 | 3.0 | 1.4 | 5.6 | 300 | 8 | 2.7 | 1.2 | 5.2 |
| Fever(°C) | All | 298 | 63 | 21.1 | 16.6 | 26.2 | 302 | 59 | 19.5 | 15.2 | 24.5 | 300 | 57 | 19.0 | 14.7 | 23.9 |
| | Grade 3 | 298 | 1 | 0.3 | 0.0 | 1.9 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 61 | 20.5 | 16.0 | 25.5 | 302 | 58 | 19.2 | 14.9 | 24.1 | 300 | 55 | 18.3 | 14.1 | 23.2 |
| Irritability | All | 298 | 213 | 71.5 | 66.0 | 76.5 | 302 | 225 | 74.5 | 69.2 | 79.3 | 300 | 191 | 63.7 | 57.9 | 69.1 |
| • | Grade 3 | 298 | 12 | 4.0 | 2.1 | 6.9 | 302 | 17 | 5.6 | 3.3 | 8.9 | 300 | 9 | 3.0 | 1.4 | 5.6 |
| | Related | | 203 | 68.1 | 62.5 | 73.4 | 302 | 220 | 72.8 | 67.5 | 77.8 | 300 | 184 | 61.3 | 55.6 | 66.9 |
| Loss of appetite | All | 298 | 79 | 26.5 | 21.6 | 31.9 | 302 | 79 | 26.2 | 21.3 | 31.5 | 300 | 73 | 24.3 | 19.6 | 29.6 |
| | Grade 3 | 298 | 0 | 0.0 | 0.0 | 1.2 | 302 | 0 | 0.0 | 0.0 | 1.2 | 300 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 298 | 75 | 25.2 | 20.3 | 30.5 | 302 | 78 | 25.8 | 21.0 | 31.2 | 300 | 67 | 22.3 | 17.7 | 27.5 |
| Vomiting | All | 298 | 47 | 15.8 | 11.8 | 20.4 | 302 | 45 | 14.9 | 11.1 | 19.4 | 300 | 44 | 14.7 | 10.9 | 19.2 |
| | Grade 3 | 298 | 11 | 3.7 | 1.9 | 6.5 | 302 | 7 | 2.3 | 0.9 | 4.7 | 300 | 7 | 2.3 | 0.9 | 4.7 |
| | Related | 298 | 45 | 15.1 | 11.2 | 19.7 | 302 | 43 | 14.2 | 10.5 | 18.7 | 300 | 39 | 13.0 | 9.4 | 17.3 |
| | | | | ļ. | | Do | se 2 | | | | | | | | | |
| Cough/runny nose | All | 296 | 92 | 31.1 | 25.9 | 36.7 | 301 | 104 | 34.6 | 29.2 | 40.2 | 299 | 95 | 31.8 | 26.5 | 37.4 |
| | Grade 3 | 296 | 2 | 0.7 | 0.1 | 2.4 | 301 | 2 | 0.7 | 0.1 | 2.4 | 299 | 4 | 1.3 | 0.4 | 3.4 |
| | Related | 296 | 79 | 26.7 | 21.7 | 32.1 | 301 | 84 | 27.9 | 22.9 | 33.3 | 299 | 79 | 26.4 | 21.5 | 31.8 |
| Diarrhoea | All | 296 | 3 | 1.0 | 0.2 | 2.9 | 301 | 7 | 2.3 | 0.9 | 4.7 | 299 | 12 | 4.0 | 2.1 | 6.9 |
| | Grade 3 | 296 | 1 | 0.3 | 0.0 | 1.9 | 301 | 2 | 0.7 | 0.1 | 2.4 | 299 | 2 | 0.7 | 0.1 | 2.4 |
| | Related | 296 | 3 | 1.0 | 0.2 | 2.9 | 301 | 7 | 2.3 | 0.9 | 4.7 | 299 | 12 | 4.0 | 2.1 | 6.9 |
| Fever(°C) | All | 296 | 80 | 27.0 | 22.1 | 32.5 | 301 | 79 | 26.2 | 21.4 | 31.6 | 299 | 94 | 31.4 | 26.2 | 37.0 |
| , , | Grade 3 | 296 | 2 | 0.7 | 0.1 | 2.4 | 301 | 1 | 0.3 | 0.0 | 1.8 | 299 | 1 | 0.3 | 0.0 | 1.8 |
| | Related | 296 | 79 | 26.7 | 21.7 | 32.1 | 301 | 76 | 25.2 | 20.4 | 30.6 | 299 | 91 | 30.4 | 25.3 | 36.0 |
| Irritability | All | 296 | 201 | 67.9 | 62.3 | 73.2 | 301 | 224 | 74.4 | 69.1 | 79.3 | 299 | 202 | 67.6 | 61.9 | 72.8 |
| , | Grade 3 | | | 3.7 | 1.9 | 6.6 | 301 | 18 | 6.0 | 3.6 | 9.3 | 299 | | 4.7 | 2.6 | 7.7 |
| | Related | | | 65.9 | 60.2 | 71.3 | 301 | 220 | 73.1 | 67.7 | 78.0 | | 200 | | 61.2 | 72.2 |
| Loss of appetite | All | 296 | | 23.3 | 18.6 | 28.6 | 301 | | 20.9 | 16.5 | 26.0 | 299 | | 23.4 | 18.7 | 28.6 |
| 17 (7 - 7 - 7 | Grade 3 | | | 0.3 | 0.0 | 1.9 | 301 | 0 | 0.0 | 0.0 | 1.2 | 299 | | 0.0 | 0.0 | 1.2 |
| | Related | 296 | | 22.6 | 18.0 | 27.8 | 301 | 59 | 19.6 | 15.3 | 24.5 | 299 | | 22.7 | 18.1 | 27.9 |
| Vomiting | All | 296 | | 14.5 | 10.7 | 19.1 | 301 | | 13.3 | 9.7 | 17.7 | 299 | | 11.0 | 7.7 | 15.1 |
| 9 | Grade 3 | 296 | | 2.4 | 1.0 | 4.8 | | 8 | 2.7 | 1.2 | 5.2 | 299 | | 2.7 | 1.2 | 5.2 |
| | Related | | | 13.5 | 9.8 | 17.9 | 301 | | 13.3 | 9.7 | 17.7 | 299 | | 10.7 | 7.4 | 14.8 |
| LIO A = HRV vacci | | | | | | 11.3 | JU 1 | τU | 10.0 | 3.1 | 17.7 | 233 | υZ | 10.1 | / .→ | 17.0 |

LIQ\_A = HRV vaccine liquid formulation Lot A

Related = any occurrence of the specified symptom assessed as causally related to the vaccination

LIQ\_B = HRV vaccine liquid formulation Lot B

LIQ\_C = HRV vaccine liquid formulation Lot C

N = number of subjects with the considered documented dose

n/% = number/percentage of subjects reporting the specified symptom for the considered dose

<sup>95%</sup> CI = Exact 95% Confidence Interval; LL = Lower Limit, UL = Upper Limit

Grade 3 = any occurrence of the specified symptom rated as grade 3

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

# Template 29 Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort)

| Study-<br>Subject<br>No. | Country | Gender | AE Description | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|
| PP<br>D | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |
| PP | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |

# Template 30 Subjects with Serious Adverse Events reported up to Visit 3 - Exposed Set

| Sub | Countr | Age at | Se | Verbatim | Preferred | System | MA | Dos | Day | Duratio | Causalit | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N. | У | onset | | | term | Organ | typ | е | of | n | У | |
| No. | | (Week | | | | Class | е | | onse | | | |
| | | , | | | | | | | t | | | |
| P | US | P | M | | Kawasaki'<br>s disease | Infections<br>and<br>infestation | НО | 1 | 12 | 29 | N | Recovered/resolve d |

MA = medical attention

HO = hospitalisation

Dose = dose given prior to the start of the SAE

Day of onset = number of days since last study vaccine dose

Template 31 Number (%) of subjects with serious adverse events from Dose 1 up to study end, including number of events reported (Exposed Set)

| | | | | Gr<br>N = | - | | Gr2<br>N = | |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System Organ<br>Class | Preferred Term<br>(CODE) | n* | n | % | n* | n | % |
| SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

Gr 1 = Group 1 description

Gr 2 = Group 2 description

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

Template 32 Solicited and unsolicited symptoms experienced by at least 5 % of subjects classified by MedDRA Primary System Organ Class and Preferred Term within 31-day (Days 0-30) post-vaccination period after any dose of HRV PCV-free liquid vaccine - SAE excluded (Exposed Set)

| | HPV_2D<br>N = | | | MM | MMR_DTPa<br>N = | | |
|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | n* | n | % |
| At least one symptom | | | | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

### Template 33 Number of subjects by country

| | ACWY-TT<br>N = 259 | ACWYHPV<br>N = 259 | HPV<br>N = 261 | Co-ad<br>N = 260 | Tdap<br>N = 261 | Total<br>N = 1300 |
|---|---|---|---|---|---|---|
| Country | n | n | N | n | n | n |
| Dominican Republic | 86 | 87 | 88 | 87 | 87 | 435 |
| Estonia | 87 | 86 | 87 | 87 | 88 | 435 |
| Thailand | 86 | 86 | 86 | 86 | 86 | 430 |

ACWY-TT = Subjects who received MenACWY-TT at Month 0 and Cervarix at Month 1, 2 and 7

ACWYHPV = Subjects who received MenACWY-TT and Cervarix at Month 0 and Cervarix at Month 1 and 6

HPV = Subjects who received Cervarix at Month 0, 1 and 6

Co-ad = Subjects who received MenACWY-TT, Cervarix and Boostrix at Month 0 and Cervarix at Month 1 and 6 Tdap = Subjects who received Boostrix and Cervarix at Month 0 and Cervarix at Month 1 and 6

N = number of subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories

115461 (ROTA-081)

Statistical Analysis Plan Amendment 1 Final

## Template 34 Number of enrolled subjects by age category (Exposed Set)

| | | Gr 1<br>N = | Gr 2<br>N = | Gr 3<br>N = | Total<br>N = |
|---|---|---|---|---|---|
| Characteristics | Categories | n | n | n | n |
| Age category | In utero | | | | |
| | Preterm newborn infants | | | | |
| | (gestational age < 37 wks) | | | | |
| | Newborns (0-27 days) | | | | |
| | Infants and toddlers (28 days- | | | | |
| | 23 months) | | | | |
| | Children (2-11 years) | | | | |
| | Adolescents (12-17 years) | | | | |
| | Adults (18-64 years) | | | | |
| | From 65-84 years | | | | |
| | 85 years and over | | | | |
| | Missing | | | | |

Gr 1 = Group 1 description

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = <describe missing>

### **Template 35 Study population (Exposed Set)**

| Number of subjects | [each group] | Total |
|---|---|---|
| Planned, N | | |
| Randomised, N ( <total cohort="" vaccinated="">)</total> | | |
| Completed, n (%) | | |
| Demographics | | |
| N ( <total cohort="" vaccinated="">)</total> | | |
| Females:Males | | |
| Mean Age, <years> (SD)</years> | | |
| Median Age, < years> (minimum, maximum) | | |
| <most category="" frequent="" of="" race="">, n (%)</most> | | |
| <second category="" frequent="" most="" of="" race="">, n (%)</second> | | |
| <third category="" frequent="" most="" of="" race="">, n (%)</third> | | |

### [each group]:

Short group label= long group label

Gr 2 = Group 2 description

Gr 3 = Group 3 description

N = Number of enrolled subjects